



# NON-INTERVENTIONAL FINAL STUDY REPORT

# **Appendix 4: Statistical Analysis Plan**

| Title | Real-World Observational Study of Zavicefta® (ceftazidime-avibactam) to Characterize Use Patterns, Effectiveness and Safety – EZTEAM Study |
|---|---|
| Protocol number | C3591031 |
| Active substance | Ceftazidime-avibactam, ACT: J01DD52 |
| <b>Medicinal product</b> | Zavicefta® (ceftazidime-avibactam) |
| Study report | Version 1.0 |

# STATISTICAL ANALYSIS PLAN AND TABLES AND LISTING SHELLS

| Document name | Date | Page |
|---------------------------------------|-----------------|------|
| Statistical Analysis Plan version 1.0 | 21 July 2020 | 3 |
| Tables and Listings shells | 11 January 2022 | 51 |



# **Non-Interventional Study Protocol**

C3591031

Real-World Observational Study of Zavicefta® (ceftazidime-avibactam) to Characterize Use Patterns, Effectiveness and Safety
– EZTEAM Study

# Statistical Analysis Plan (SAP)

Version: 1.0

Author: PPD Pfizer Inc, PPD

PPD , IQVIA Real World Solutions

**Date**: 21 July 2020


Statistical Analysis Plan

# **TABLE OF CONTENTS**

| L | IST OF TABLES | 4 |
|---|---|---|
| L | IST OF FIGURES | 4 |
| L | IST OF ABBREVIATIONS | 5 |
| 1 | INTRODUCTION | |
| | 1.1 RATIONALE AND BACKGROUND | |
| | 1.2 STUDY DESIGN | |
| | 1.3 STUDY POPULATION | |
| | 1.3.1 Study Size in Europe | 8 |
| | 1.3.2 Study size in Latin America | |
| | 1.3.3 Potential COVID-19 Impact | |
| | 1.4 Data Source | |
| | 1.5 STUDY OBJECTIVES | 11 |
| 2 | DECISION RULES | 11 |
| 3 | ANALYSIS SETS/ POPULATIONS | 12 |
| | 3.1 ALL PATIENTS ENROLLED SET | 12 |
| | 3.2 FULL ANALYSIS SET | |
| | 3.2.1 Inclusion criteria | 12 |
| | 3.2.2 Exclusion criteria | 12 |
| | 3.3 Analysis set with at least 72 hours exposure to ceftazidime- | |
| | AVIBACTAM. | 13 |
| | 3.4 Analysis set with less than 72 hours exposure to ceftazidime- | 10 |
| | AVIBACTAM. | |
| | 3.5 ANALYSIS DATA SET FOR CLINICAL OUTCOMES | |
| 4 | OUTCOMES AND COVARIATES | 14 |
| | 4.1 SITE CHARACTERISTICS | 14 |
| | 4.2 BASELINE DEMOGRAPHIC CHARACTERISTICS FOR PATIENTS EXPOSED TO | |
| | Ceftazidime-avibactam for ≥72 hours | 15 |
| | 4.3 BASELINE CLINICAL CHARACTERISTICS FOR PATIENTS EXPOSED TO | |
| | CEFTAZIDIME-AVIBACTAM FOR ≥72 HOURS | 15 |
| | 4.4 PATTERN OF USE OF CEFTAZIDIME-AVIBACTAM FOR PATIENTS EXPOSED TO | 1.7 |
| | CEFTAZIDIME-AVIBACTAM FOR ≥72 HOURS | 16 |
| | 4.5 EFFECTIVENESS OUTCOMES FOR PATIENTS EXPOSED TO CEFTAZIDIME-<br>AVIBACTAM FOR ≥72 HOURS | 17 |
| | 4.5.1 Clinical outcomes. | |
| | 4.5.2 Microbiological outcomes | |
| | 4.5.3 Prevalence of hospital readmissions | |
| | 4.6 MORTALITY OUTCOMES | |


Statistical Analysis Plan

| | 4.7 HEALTHCARE UTILIZATION OUTCOMES FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM FOR ≥72 HOURS | 10 |
|---|---|---|
| | 4.8 SAFETY OUTCOMES FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM | |
| | ≥72 HOURS | |
| | 4.8.1 Adverse Events | |
| | 4.8.2 Serious Adverse Events | 20 |
| | 4.9 VARIABLES AND OUTCOMES FOR ANALYSIS AMONG PATIENTS EXPOSED TO | |
| | CEFTAZIDIME-AVIBACTAM <72 HOURS | |
| 5 | DEFINITIONS | |
| 6 | HANDLING OF MISSING VALUES | 26 |
| 7 | STATISTICAL METHODS | 26 |
| 8 | STATISTICAL ANALYSES | 27 |
| | 8.1 GENERAL CONSIDERATIONS | 27 |
| | 8.2 SITE CHARACTERISTICS | |
| | 8.3 PATIENT DISPOSITION | |
| | 8.4 BASELINE DEMOGRAPHIC CHARACTERISTICS | 28 |
| | 8.5 BASELINE CLINICAL CHARACTERISTICS | 28 |
| | 8.6 PATTERN OF USE OF CEFTAZIDIME-AVIBACTAM | |
| | 8.6.1 Source of infection | |
| | 8.6.2 Indication for ceftazidime-avibactam | |
| | 8.6.3 Antibiotics used for index infection before ceftazidime-avibactam initia | |
| | 8.6.4 Use of ceftazidime-avibactam | |
| | 8.6.5 Concomitant antibiotic therapy during index hospitalization | 30 |
| | 8.6.6 Antibiotic therapy after ceftazidime-avibactam during the index hospitalization: | 20 |
| | 8.7 Microbiological Evaluation | |
| | 8.8 EFFECTIVENESS | |
| | 8.8.1 Clinical outcomes. | |
| | 8.8.2 Microbiological outcomes | |
| | 8.8.3 Prevalence of hospital readmissions | |
| | 8.9 Mortality | |
| | 8.10 HEALTHCARE RESOURCE UTILIZATION | 33 |
| | 8.10.1 Hospital length of stay | 33 |
| | 8.10.2 Resource utilization | 34 |
| | 8.11 ADVERSE EVENTS | 35 |
| 9 | | |
| E | XPOSURE | 35 |
| | 9.1 DEMOGRAPHIC CHARACTESITICS | 35 |
| | 9.2 SOURCE OF INFECTION | 35 |
| | 9.3 Indication for ceftazidime-avibactam | 35 |
| | 9.4 USE OF CEFTAZIDIME-AVIBACTAM | 35 |
| _ | 9.5 IN-HOSPITAL MORTALITY | 36 |
| | Page 3 o | f 47 |

| NIS Pr | otocol | C3591 | 031 |
|--------|--------|-------|-----|
|--------|--------|-------|-----|

# Statistical Analysis Plan

| 10 | SAFETY | 36 |
|---|---|---|
| 11 | REFERENCES | 37 |
| 12 | LIST OF TABLE SHELLS | 38 |
| 13 | LIST OF LISTINGS | |
| 14 | APPENDIX | |
| 1 | 4.1 PARTIAL DATE CONVENTIONS | |
| | LIST OF TABLES | |
| | ble 1. Sample Size and Precision of the Estimate for Clinical Treatment Success | |
| | ble 2. Sample Size and Precision of the Estimate for Microbiological Treatment | |
| | ble 3. Deyo-Charlson Comorbidity Index | |
| Tal | ble 4. Decimal Placees for Table Shells | 27 |
| Tal | ble 5. Clinical Outcomes Missing Data Rules at 30 Days or at 60 Days Post-Disc | _ |
| Tal | ble 6. Algorithm for Treatment Emergence of Adverse Events | |
| | ST OF FIGURES | |
| Fig | ure 1. Study Flow Chart | 7 |
| | ure 2. Patient Flow Chart | |
| Fig | ure 3. Data Sets | 14 |


Statistical Analysis Plan

# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | Adverse Event |
| APACHE | Acute Physiology and Chronic Health Evaluation Score |
| BMI | Body Mass Index |
| BSI | Bloodstream Infection |
| CAI | Community-Acquired Infection |
| CI | Confidence Interval |
| cIAI | Complicated Intra-Abdominal Infection |
| CLABSI | Central Line Associated Blood Stream Infection |
| COD | Clinical Outcomes Dataset |
| CT | Computerized Tomography |
| cUTI | Complicated Urinary Tract Infection |
| DCCI | Deyo-Charlson Comorbidity Index |
| eCRF | Electronic Case Report Form |
| ENR | Enrolled Dataset |
| FAS | Full Analysis Set |
| FAS72+ | Analysis Set With At Least 72 Hours Exposure To Ceftazidime-Avibactam |
| FAS72- | Analysis Set With Less Than 72 Hours Exposure To Ceftazidime-Avibactam |
| HAI | Hospital-Acquired Infection |
| HAP | Hospital-Acquired Pneumonia |
| HCAI | Healthcare-Associated Infection |
| ICU | Intensive Care Unit |
| IV | Intravenous |
| LOS | Length of Stay |
| MDR | Multidrug-Resistant |
| MRI | Magnetic Resonance Imaging |
| NI | Non-Interventional |
| NIS | Non-Interventional Study |
| NP | Nosocomial Pneumonia |
| PT | Preferred Term |
| Q1 | First Quartile |
| Q3 | Third Quartile |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System (SAS Institute) |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| VAP | Ventilator-Associated Pneumonia |


Statistical Analysis Plan

#### 1 INTRODUCTION

Note: in this document any text taken directly from the non-interventional study (NIS) study protocol is *italicized*.

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of the general treatment patterns, effectiveness, and the safety of ceftazidime-avibactam. It describes the data to be summarized and analyzed, including full details of the planned statistical analyses. This is a NIS based on the review of patient medical records.

This SAP is based on Protocol number C3591031, Version 4.0, Amendment 3 dated 29th April 2020.

#### 1.1 RATIONALE AND BACKGROUND

Antimicrobial resistance and healthcare-associated infections (HCAIs) are well known public health threats. Gram-negative bacteria cause common hospital-acquired infections (HAIs) and infection with multidrug-resistant gram-negative organisms (MDRGNs), and have been associated with increased morbidity, mortality, and healthcare costs. Zavicefta® (ceftazidime-avibactam) is a unique combination of ceftazidime and avibactam developed to treat infections caused by gram-negative pathogens.

In the European Union, Russia and several Latin American countries, ceftazidime-avibactam is an approved treatment of complicated intra-abdominal infection (cIAI), complicated urinary tract infections (cUTIs), hospital-acquired pneumonia/ventilator-associated pneumonia (HAP/VAP), and infection due to aerobic gram-negative organisms with limited treatment options. Ceftazidime-avibactam has proven efficacious in non-inferiority Phase III trials but real-world evidence is needed about treatment characteristics, safety, and efficacy against Pseudomonas and multidrug-resistant (MDR) bacteria including carbapenem-resistant Enterobacteriaceae (CRE).

#### 1.2 STUDY DESIGN

This is a NI medical chart review study aiming to examine the treatment patterns, effectiveness, and safety of ceftazidime-avibactam in approximately 12 countries and 63 sites in Europe (including Russia) and Latin America.

Patients treated with at least one dose of ceftazidime-avibactam (for the indication that is approved as per country label) in routine clinical practice at a participating site since 01 January 2018 or the date of launch in the country if after 2018 can be enrolled.

As this is an observational study, patients are treated as per local label based on the standard of care at the discretion of their physician. No drugs are supplied for this study and patients receive treatment through standard local practice. Patients treated as part of a compassionate program of ceftazidime-avibactam are not eligible to participate in the study.


Statistical Analysis Plan

All data will be collected through the abstraction of hospital medical records. Collected study data will include but will not be limited to patient characteristics, clinical and microbiological characteristics of the infection, and treatment patterns, effectiveness, and safety of ceftazidime-avibactam. The study data collection and assessment schedule are described in Figure 1.

Figure 1. Study Flow Chart



<sup>&</sup>lt;sup>1</sup> Indicates outcome that will be examined for patients exposed to ceftazidime-avibactam for  $\geq 72$  hours.

Patients who were exposed to ceftazidime-avibactam for ≥72 hours will be eligible for effectiveness analyses, including evaluation of treatment success. To avoid a selection bias that could result from restricting to patients with extended exposure, a small set of data elements will be collected and analyzed among patients with <72 hours of exposure. These data include details about exposure, indication, and safety. Safety data will be analyzed for all patients enrolled.

Patients who meet all the inclusion and exclusion criteria will be followed through their medical records up to 60 days after hospital discharge, death, withdrawal from the study, or loss-to-follow-up, whichever occurs first.

Besides routine treatment, no clinic visits are required as part of participation in this study. All data is intended to be collected by referencing the medical record. For patients missing any of the requested information, data will be reported as missing. Eligibility in the study has been summarized below in Section 3.2. Patients participating in clinical


<sup>&</sup>lt;sup>2</sup> Microbiological cultures performed during hospitalization.

<sup>&</sup>lt;sup>3</sup> Information about hospital readmissions or death after hospital discharge not available via medical chart abstraction will be ascertained by contacting the patient or their legal representative by phone >60 days after hospital discharge

<sup>†</sup> Patients followed from ceftazidime-avibactam initiation until 60 days after hospital discharge or another censoring event (in-hospital death, withdrawal from the study, or loss-to-follow-up, whichever occurs first). Data will be abstracted from patient medical charts.

Statistical Analysis Plan

trials are excluded from this study because protocol driven activities may be outside of normal practice and could confound safety assessments.

The study patient flow chart of events is presented in Figure 2.

Figure 2. Patient Flow Chart



#### 1.3 STUDY POPULATION

Overall, 700 patients with a gram-negative infection who have received at least one dose of ceftazidime-avibactam will be enrolled in this study.

#### 1.3.1 Study Size in Europe

Sample size for this study was calculated with the goal of maximizing precision when estimating clinical and microbiological treatment success.

Clinical Treatment Success Assumptions (1-3):

- 25% of the enrolled patients discontinue ceftazidime-avibactam before 72 hours of exposure (e.g. due to adverse event (AE), microbiological results)
- 75% of patients are exposed to ceftazidime-avibactam for ≥72 hours and are assessable for clinical effectiveness. 70% of the assessable patients experience clinical treatment success, as defined in Section\_5.


Statistical Analysis Plan

Table 1. Sample Size and Precision of the Estimate for Clinical Treatment Success

| | | - | Pi | revalence of Clinica | ıl Treatment Succe | SS |
|---|---|---|---|---|---|---|
| | | 60% | 65% | 70% | 75% | 80% |
| | 200 | (52.9% -<br>66.8%) | (58.0% - 71.6%) | (63.1% - 76.3%) | (68.4% - 80.8%) | (73.8% - 85.3%) |
| | 300 | (54.2% -<br>65.6%) | (59.3% - 70.4%) | (64.5% - 75.1%) | (69.7% - 79.8%) | (75.0 % - 84.4%) |
| N | 400 | (55.0% -<br>64.8%) | (60.1% - 69.7%) | (65.2 % - 74.5%) | (70.5% - 79.2%) | (75.7% - 83.8%) |
| | 500 | (55.6% -<br>64.3%) | (60.6% - 69.2%) | (65.8% - 74.0%) | (71.0% - 78.7%) | (76.2% - 83.4%) |
| | 600 | (56.0% -<br>63.9%) | (61.0% - 68.8%) | (66.2% - 73.6%) | (71.3% - 78.4%) | (76.6% - 83.1%) |

Note: Displayed range is the 95% confidence interval around the estimate of treatment success

*Microbiological Treatment Success Assumption* (1-3):

- 25% of the enrolled patients discontinue ceftazidime-avibactam before 72 hours of exposure (e.g. due to AE, microbiological results),
- 75% of patients are exposed to ceftazidime-avibactam for  $\geq$ 72 hours,
- 10% of patients exposed ≥ 72 hours (across all indications) have no pathogen identification and are not assessable for microbiological success,
- 80% of the assessable patients experience microbiological treatment success as defined in Section 5.

**Table 2. Sample Size and Precision of the Estimate for Microbiological Treatment Success** 

| | | | Prevai | lence of Microbiolo | ogical Treatment S | uccess |
|---|---|---|---|---|---|---|
| | | 70% | 75% | 80% | 85% | 90% |
| | 200 | (63.1% - 76.3%) | (68.4% - 80.8%) | (73.8% - 85.3%) | (79.3% - 89.6%) | (85.0% - 93.8%) |
| | 300 | (64.5% -<br>75.1%) | (69.7% - 79.8%) | (75.0% - 84.4%) | (80.4% - 88.8%) | (86.0% - 93.2%) |
| N | 400 | (65.2% -<br>74.5%) | (70.5% - 79.2%) | (75.7% - 83.8%) | (81.1% - 88.4%) | (86.6% - 92.8%) |
| | 500 | (65.8% -<br>74.0%) | (71.0% - 78.7%) | (76.2% - 83.4%) | (81.6% - 88.0%) | (87.0% - 92.5%) |
| | 600 | (66.2% -<br>73.6%) | (71.3% - 78.4%) | (76.6% - 83.1%) | (81.9% - 87.8%) | (87.3% - 92.3%) |

Note: Displayed range is the 95% confidence interval around the estimate of treatment success

Table 1 and Table 2 display estimates of clinical and microbiological treatment success, respectively, and the asymptotic precision of each estimate (95% confidence interval (CI)), for sample sizes ranging from 300 to 600 evaluable patients.


Statistical Analysis Plan

To obtain a 95% CI for treatment success that is approximately 12.3 percentage points or less for both clinical and microbiological treatment success, 225 evaluable patients are required. Given the assumptions above for both treatment outcomes, a minimum of 300 patients should be enrolled to obtain 225 evaluable patients. Minor gains in precision can be achieved by enrolling a larger number of patients.

Enrolling 300 patients would lead to 225 patients with  $\geq$  72 hours exposure to ceftazidime-avibactam evaluable for clinical success, and 202 patients evaluable for microbiological success. It would yield an expected 95% CI of 70.0% (63.6% - 75.9%) of patients experiencing clinical treatment success and 80.0% (73.8% - 85.3%) of patients experiencing microbiological treatment success using a two-sided exact method.

Note: The precision estimates were calculated using the Clopper Pearson (exact) CIs using statistical analysis system (SAS)<sup>®</sup> software version 9.2 (4).

# 1.3.2 Study size in Latin America

Based on the same assumptions for treatment outcomes as in Europe, to obtain a 95% CI for treatment success that is approximately 10.0 percentage points for both clinical and microbiological treatment success, 400 patients will be included in Latin America to obtain 300 evaluable patients for clinical success, and 270 evaluable patients for microbiological success. Using a two-sided exact method, enrolling 400 patients would yield an expected 95% CI of 70.0% (64.5% - 75.1%) of patients experiencing clinical treatment success and 80.0% (74.7% - 84.6%) of patients experiencing microbiological treatment success.

#### 1.3.3 Potential COVID-19 Impact

Coronavirus disease (COVID-19) pandemic is likely to impact the final sample size in both Europe and LATAM. Many sites did not work during this period, e.g. in Europe and LATAM there were approximately 24 unresponsive sites during the April and May 2020, and around 12 unresponsive sites in June 2020. However, this should not impact the analyses, but the precision of the estimates may have to be revised.

#### 1.4 DATA SOURCE

Patients will be enrolled from approximately 62 sites in 12 countries in Europe and in Latin America. Sites will be qualified and then selected based on responses to a series of questions intended to determine their capability of conducting the study and ability to contribute to the target patient population.

The data source for this study will be patient medical records. Data will be abstracted from records between the date of hospital admission and up to 60 days after hospital discharge or a censoring event (death, withdrawal from the study, or lost-to-follow-up). Patients should be carefully tracked to identify censoring events.

Adverse Events (AEs) will be collected as part of standard practice. Information regarding the reporting of AEs is described in Section 4.8.1 of this SAP and Section 11 of the protocol.


Statistical Analysis Plan

#### 1.5 STUDY OBJECTIVES

The main objective of this NI medical chart review study is to describe the general treatment patterns, effectiveness, and safety of ceftazidime-avibactam in real-world settings.

The primary objective of this study is to describe the patterns of use of ceftazidime-avibactam in real-world practice.

- 1. Describe the indications and reasons for use of ceftazidime-avibactam; provide detailed information about its use for the treatment of infections due to aerobic gram-negative organisms with limited treatment options.
- 2. Describe the usage patterns of ceftazidime-avibactam, including treatment line, dose, frequency of dose, duration, and polytherapy regimens.
- 3. Describe the microbiological evidence available for patients treated with ceftazidime-avibactam.
- 4. Describe the source of infection for which ceftazidime-avibactam is prescribed including community-acquired infections (CAIs), HCAIs, and HAIs.

The secondary objective of this study is to determine the effectiveness and safety of ceftazidime-avibactam in real-world practice.

- 1. Describe the clinical outcomes of patients treated with ceftazidime-avibactam (i.e. treatment success, failure, or indeterminate) in hospital and up to 30- and 60-days post hospital discharge.
- 2. Describe the microbiological outcomes among patients treated with ceftazidimeavibactam during the 14 days after ceftazidime-avibactam initiation
- 3. Describe safety outcomes in patients receiving ceftazidime-avibactam between treatment initiation and hospital discharge.
- 4. Describe the in-hospital length of stay (LOS), LOS in intensive care unit (ICU) and healthcare resource utilization in patients with infections treated by ceftazidime-avibactam.
- 5. Determine the prevalence of hospital readmissions for recurrence of the same infection within 30 and 60 days of hospital discharge among patients treated with ceftazidime-avibactam.
- 6. Determine the in-hospital mortality and mortality up to 30 and 60 days after hospital discharge.

#### 2 DECISION RULES

For patients treated with ceftazidime-avibactam, the clinical and microbiological outcomes will be evaluated according to the definitions in Section 5. Handling missing data, in general, is discussed in Section 6. The evaluation rules for missing clinical outcomes are provided in Table 5.


Statistical Analysis Plan

#### 3 ANALYSIS SETS/ POPULATIONS

The data from the chart reviews will be anonymized patient-level data that will be pooled to create the analysis data sets described below. Each country and patient will be assigned a unique identifier.

#### 3.1 ALL PATIENTS ENROLLED SET

All the patients enrolled set (ENR) will contain all subjects who provide informed consent. This set will only be used to calculate the attrition table, i.e. the number of patients retained at each application of the study inclusion/exclusion criteria.

#### 3.2 FULL ANALYSIS SET

The full analysis set (FAS) will contain all enrolled patients meeting the study eligibility criteria set out below. This set will also be used for safety analysis.

#### 3.2.1 <u>Inclusion criteria</u>

Patients must meet all the following inclusion criteria to be eligible:

- 1. Hospitalized patient  $\geq 18$  years old or considered an adult in accordance with the age of majority in the participant's country of residence at the time of treatment with ceftazidime-avibactam.
- **2.** Patient received ≥1 dose of ceftazidime-avibactam in routine practice at participating site since the date of ceftazidime-avibactam launch in the country, or January 2018, or the date of launch in the country if after 2018.
- **3.** Patient underwent microbiological sampling ≤5 days before the initiation of ceftazidime-avibactam (irrespective of results and actual bacteriological identification).
- 4. Patient has all required essential data elements which include:
  - **a.** Start and stop dates of ceftazidime-avibactam,
  - **b.** Start and stop dates of prior antibiotic therapy used for the index infection,
  - **c.** Type of combined antibiotic therapy (if applicable) and start and stop dates of any antibiotic combined with ceftazidime-avibactam.
- **5.** Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study where required by local regulations.

# 3.2.2 Exclusion criteria

Patients must not meet any of the following exclusion criteria to be eligible:

- 1. The patient is enrolled in any clinical trial of an investigational product. Patients who are enrolled in non-interventional studies (e.g. registries) are eligible for inclusion.
- 2. The patient has received ceftazidime-avibactam in a compassionate care program setting.


Statistical Analysis Plan

3. The patient was exposed to ceftazidime-avibactam before use for the index infection.

The FAS will be divided into patients with at least 72 hours of exposure to ceftazidime-avibactam, and patients with <72 hours exposure.

# 3.3 ANALYSIS SET WITH AT LEAST 72 HOURS EXPOSURE TO CEFTAZIDIME-AVIBACTAM.

Analysis set at least 72 hours (FAS72+) will be a subset of the FAS patients with at least 72 hours of exposure to ceftazidime-avibactam.

# 3.4 ANALYSIS SET WITH LESS THAN 72 HOURS EXPOSURE TO CEFTAZIDIME-AVIBACTAM.

Analysis set less than 72 hours (FAS72-) will be a subset of the FAS patients with <72 hours exposure to ceftazidime-avibactam.

# 3.5 ANALYSIS DATA SET FOR CLINICAL OUTCOMES

The clinical outcomes dataset (COD) will consist of all patients with at least 72 hours exposure to ceftazidime-avibactam and at least one non-missing clinical outcome. COD will be a subset of FAS72+.

# 3.6 ANALYSIS DATA SET FOR MICROBIOLOGY OUTCOMES

The microbiological outcomes dataset (MOD) will consist of patients with at least 72 hours exposure to ceftazidime-avibactam, identification of one or more pathogens before the start of ceftazidime-avibactam treatment, and at least one non-missing microbiological outcome. MOD will be a subset of FAS72+.

Figure 3 shows how the patients for each analysis data set are derived.


Statistical Analysis Plan

Figure 3. Data Sets



#### 4 OUTCOMES AND COVARIATES

# 4.1 SITE CHARACTERISTICS

Site characteristics will be described as below, based on data from FAS.

- Physician specialty:
  - o Infectious disease
  - o Microbiology
  - o Surgery
  - o Internal medicine
  - o Intensive care
  - Anesthesiology
  - Other
- Hospital information:
  - o Care level
  - o Type
  - o Total number of beds
  - o Total number of ICU beds
- Local gram-negative resistance rates (between 01 Jan 2018 and 30 Jun 2019, or other duration) to:
  - o 3rd generation cephalosporins
  - Carbapenem


Statistical Analysis Plan

- o 3rd generation cephalosporins and carbapenems
- o Colistin

# 4.2 BASELINE DEMOGRAPHIC CHARACTERISTICS FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM FOR ≥72 HOURS

Baseline demographic characteristics of patients will be described as below, based on data from FAS72+.

- Exposure to ceftazidime-avibactam:
  - Exposed to ceftazidime-avibactam for a duration of  $\geq$  72 hours
  - Exposed to ceftazidime-avibactam for a duration of < 72 hours
- Age
- Gender
- Height and weight (Body mass index [BMI] will be derived)
- Employment status
- Additional risk factors:
  - o Travel to foreign country within the past 3 months;
    - Country
    - Duration of travel
    - Hospitalization
  - o Pregnancy (weeks of gestation since last menstrual period);
  - o Alcohol use (drinks per week);
  - o Smoker status (current/previous/never/unknown) and cigarettes per day.

# 4.3 BASELINE CLINICAL CHARACTERISTICS FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM FOR ≥72 HOURS

Baseline clinical characteristics of patients will be described as below, based on data from FAS72+.

- Comorbidities, individual comorbidities and Deyo-Charlson Comorbidity Index (DCCI), see Section 5 for detailed description.
- *Indwelling devices that the patient had at the time of the infection diagnosis.*
- Hospitalization within 90 days prior to index hospitalization:
  - o LOS of hospitalization
  - Primary diagnosis at discharge.
- *Type(s) of healthcare procedure within the 30 days before the index date.*
- *History of antibiotic exposure within 90 days prior to index hospitalization:* 
  - Antibiotic name(s)
  - o Duration(s)
  - o Reason for treatment
    - Therapeutic
    - Prophylactic
- Prior antibiotic exposure for the index infection:
  - Antibiotic name(s)
  - o Dose(s)
  - o Duration(s) of use


Statistical Analysis Plan

- Reason for treatment
  - Microbiology
  - No improvement or worsening on previous antibiotic
  - Other
- o Reason for discontinuation
  - Perceived clinical failure/disease no improvement or worsening
  - Isolation of a resistant pathogen
  - Preference for empiric coverage
  - Secondary infection requiring regimen change
  - *Switch to oral therapy*
  - De-escalation
  - Cure
  - Death
  - Other
- Pre-treatment disease severity Acute Physiology and Chronic Health Evaluation Score (APACHE II) or other prognostic assessment within 7 days prior to index date, for patients directly admitted to intensive care unit (ICU).
- Source of infection: HAI, HCAI, CAI.
- Indication for ceftazidime-avibactam:
  - o cIAI, cUTI, HAP/VAP, other (primary and secondary diagnosis)
  - o Initial site of infection (organ)
- Indication for ceftazidime-avibactam other:
  - Type of infection (e.g., SSI, Central line associated blood stream infection (CLABSI), primary Bloodstream infection (BSI), meningitis, other)
  - o Initial site of infection (organ)
- Pre-treatment microbiology sample
  - Microbiological culture(s) of current infection during the 5 days of ceftazidime-avibactam initiation (sample date(s), sample source(s)).
- Pre-treatment microbiology results
- Results from microbiological culture (method of testing, identified pathogen(s), susceptibility, MDR).

# 4.4 PATTERN OF USE OF CEFTAZIDIME-AVIBACTAM FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM FOR >72 HOURS

Patterns of use of ceftazidime-avibactam will be described as below, based on data from FAS.

- *Ceftazidime-avibactam treatment patterns:* 
  - o Dose(s), frequency, and duration
  - o Reason for initiating
  - Reason for discontinuation (if applicable) (e.g. AE, perceived clinical failure, isolation of a resistant pathogen, preference for empiric coverage, secondary infection requiring regimen change, switch to oral therapy, deescalation, cure, death).

Patterns of use of antibiotics will be as described below, based on data from FAS72+.


Statistical Analysis Plan

- Antibiotic(s) used for the index infection before ceftazidime-avibactam initiation.
  - o *Lines of treatments*
  - o Dose(s), frequency, duration and route of administration
  - Reason for initiating (microbiology, no improvement or worsening on previous antibiotic), reason for discontinuation (AE, perceived clinical failure, isolation of a resistant pathogen, preference for empiric coverage, secondary infection requiring regimen change, switch to oral therapy, deescalation).
- *Lines of antibiotic therapy(s)* 
  - Number of lines
  - Reason for change in line (e.g. AE, perceived clinical failure, isolation of a resistant pathogen, preference for empiric coverage, secondary infection requiring regimen change, switch to oral therapy, deescalation, cure, death).
- Concomitant antibiotic therapy
  - Antibiotic(s) used concurrently with ceftazidime-avibactam,
  - Dose(s), frequency, duration and route of administration,
  - Reason for initiating and reason for discontinuation (e.g. AE, perceived clinical failure, isolation of a resistant pathogen, preference for empiric coverage, secondary infection requiring regimen change, switch to oral therapy, de-escalation, cure, death) (if applicable).

# 4.5 EFFECTIVENESS OUTCOMES FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM FOR >72 HOURS

#### 4.5.1 Clinical outcomes

Each line of therapy that includes ceftazidime-avibactam will be evaluated for the clinical effectiveness outcomes and will be described according to the variables listed below, based on data from COD.

- Clinical symptoms improvement
  - Symptoms improvement or worsening within 48 and 72 hours of ceftazidime-avibactam initiation
- Resolution of all signs and symptoms of infection with no need for escalation of antimicrobials.
  - De-escalation of antibiotic therapy is considered a treatment success unless ceftazidime-avibactam was used in a regimen with one or more other antibiotics and is the only antibiotic de-escalated.
- Hospital readmission during the 30 and 60 days after initial discharge, by reason for readmission.
- Clinical treatment outcome:
  - o Success, failure, or indeterminate (see Section 5 for definitions).


Statistical Analysis Plan

# 4.5.2 Microbiological outcomes

Each line of therapy that includes ceftazidime-avibactam will be evaluated for the microbiological effectiveness outcomes, providing that a pathogen was identified. *Microbiological treatment outcome should be assessed at the end of each regimen containing ceftazidime-avibactam.* 

The microbiological effectiveness outcomes will be described according to the variables listed below, based on data from MOD.

- Post treatment initiation microbiology sample. Microbiological culture(s) during the 14 days after ceftazidime-avibactam initiation (sample date, sample site).
- Post treatment initiation microbiology results
  - Results from microbiological culture after treatment initiation (method of testing, identified pathogen(s), susceptibility, MDR).
- Microbiological treatment outcome
  - Success, failure, emergent infections and unevaluable. See Section 8.7 or details on microbiological treatment outcomes.

# 4.5.3 Prevalence of hospital readmissions

Prevalence of hospital readmissions for recurrence of the index infection within 30 and 60 days of hospital discharge among patients treated with ceftazidime-avibactam.

- o readmissions within 60 days
  - reason for readmission
- o readmissions within 30 days
  - reason for readmission
- Summary of the number of days readmitted
- Prevalence rates of readmission for index infection at 30 days and 60 days postdischarge.

Results will be presented overall, stratified by country, indication, and bacteria.

#### 4.6 MORTALITY OUTCOMES

Mortality outcomes will be described according to the variables listed below, based on data from FAS72+.

- In-hospital mortality occurring after treatment initiation but before hospital discharge
  - o Numbers of days after treatment initiation
  - o Cause of death.
- 30-day mortality mortality within 30 days after hospital discharge
  - Numbers of days after hospital discharge
  - o Cause of death.
- 60-day mortality mortality within 60 days after hospital discharge
  - o Numbers of days after hospital discharge
  - o Cause of death.
- Cumulative 30-day mortality mortality within 30 days after hospital discharge


Statistical Analysis Plan

(in-hospital + 30 days after discharge)

- o Numbers of days after treatment initiation
- o Cause of death.
- Cumulative 60-day mortality mortality within 60 days after hospital discharge (in-hospital + 60 days after discharge)
  - o Numbers of days after treatment initiation
  - o Cause of death.

# 4.7 HEALTHCARE UTILIZATION OUTCOMES FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM FOR ≥72 HOURS

The outcomes related to healthcare utilization will be described according to the variables listed below, based on data from the FAS72+.

- Hospital stay
  - o LOS
  - o Diagnosis at admission
  - o Hospital ward
    - All wards attended, ward of admission, ward of diagnosis (surgical, medical, onco-hematology, infectious disease, ICU, other)
- ICU stay
  - $\circ$  LOS
  - o diagnosis at admission
- Healthcare utilization
  - Detailed list of healthcare utilization (diagnosis at admission, departments admitted/discharged, discharge diagnosis, mechanical ventilation, dialysis, computerized tomography (CT)/magnetic resonance imaging(MRI) imaging, tracheostomy, surgical intervention, percutaneous procedures, other) and dates of service.

# 4.8 SAFETY OUTCOMES FOR PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM FOR ≥72 HOURS

The safety outcomes are defined as AEs and serious adverse events (SAEs) attributable to ceftazidime-avibactam as captured in the patients' medical charts. The safety outcomes will be described according to the variables listed below, based on data from the FAS72+.

- Safety
  - All serious and non-serious AEs with explicit attribution to ceftazidimeavibactam that appear in the reviewed information and scenarios involving drug exposure to ceftazidime-avibactam, including exposure during pregnancy, exposure during breastfeeding, medication error, overdose, misuse, extravasation, lack of efficacy and occupational exposure associated with the use of ceftazidime-avibactam.

# 4.8.1 Adverse Events

• Adverse Events (AEs) will be coded using MedDRA Version 21.0 or higher.


Statistical Analysis Plan

- See Section 6 for the handling of partial dates for AEs.
- An overall summary of numbers of patients within each of the categories described in the sub-section below, will be provided. If a patient reports an AE more than once within a System Organ Class (SOC)/Preferred Term (PT), then all AEs will be described. Number and percent of serious and non-serious AEs will be presented by SOC and PT and broken down further by maximum severity and relationship to study medication.

The protocol requires human review of patient-level unstructured data with reporting of AEs with explicit attribution to any Pfizer drug that appear in the reviewed information (defined per the patient population and study period). Explicit attribution is not inferred by a temporal relationship between drug administration and an AE but will be based on a definite statement of causality by a healthcare provider linking drug administration to the AE.

Pfizer Safety requirements include the following:

- All serious and non-serious AEs with explicit attribution to any Pfizer drug.
- Scenarios involving exposure to any Pfizer drug, including exposure during
  pregnancy, exposure during breast feeding, medication error, overdose, misuse,
  extravasation, lack of efficacy and occupational exposure associated with the use
  of a Pfizer product

For these safety events with an explicit attribution to or associated with use of, respectively, a Pfizer product, the data captured in the medical record will constitute all clinical information known regarding these AEs. No follow-up on related AEs will be conducted.

#### 4.8.2 <u>Serious Adverse Events</u>

SAEs are those events recorded as "Serious" on the AEs Form of the electronic case report form (eCRF). An SAE is defined as any untoward medical occurrence that at any dose:

- · Results in death
- Is life-threatening
- Requires hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly or birth defect
- Is an important medical event.

Number and percent of serious AEs will be presented by SOC and PT.

# 4.9 VARIABLES AND OUTCOMES FOR ANALYSIS AMONG PATIENTS EXPOSED TO CEFTAZIDIME-AVIBACTAM <72 HOURS

- Age
- Sex


Statistical Analysis Plan

- Source of infection: HAI, HCAI, CAI
- Indication for ceftazidime-avibactam
  - o cIAI, cUTI, HAP/VAP, other
  - o Initial site of infection (organ)
- Indication for ceftazidime-avibactam Other
  - o Type of infection (e.g., SSI, CLABSI, primary BSI, meningitis, other)
  - o Initial site of infection (organ).

Patterns of use of ceftazidime-avibactam will be described as below.

- Ceftazidime-avibactam treatment patterns:
  - o Dose(s), frequency, and duration
  - o Reason for initiating
  - Reason for discontinuation (if applicable) (e.g. AE, perceived clinical failure, isolation of a resistant pathogen, preference for empiric coverage, secondary infection requiring regimen change, switch to oral therapy, deescalation, cure, death).
- In-hospital mortality occurring after treatment initiation but before hospital discharge
  - o Numbers of days after treatment initiation
  - o Cause of death.
- Safety
  - All serious and non-serious AEs with explicit attribution to ceftazidimeavibactam that appear in the reviewed information and scenarios involving drug exposure to ceftazidime-avibactam, including exposure during pregnancy, exposure during breastfeeding, medication error, overdose, misuse, extravasation, lack of efficacy and occupational exposure

#### 5 DEFINITIONS

- 1. Indication for ceftazidime-avibactam prescription
  - cUTI
  - cIAI
  - HAP/VAP
  - Other infection with limited treatment options: any infection, based upon empiric or microbiological evidence, for which ceftazidime-avibactam is prescribed. Detailed information on the infection should be collected for analysis including type of infection (e.g. primary BSI, SSI, CLABSI, meningitis, HAP), and original source of infection (i.e. specific organ/locale).

### 2. Pathogen:

In this NIS, any microorganism(s) that the investigator has considered as a pathogen likely to cause the infection presented by the patient.

3. Multidrug-resistance:

The isolate is non-susceptible to at least one agent in  $\geq 3$  antimicrobial categories, excluding the therapeutic classes to which the bacteria is intrinsically resistant.


Statistical Analysis Plan

Categories include but are not limited to aminoglycosides, carbapenems, cephalosporins, cephamycins, fluoroquinolones, folate pathway inhibitors, glycylcyclines, penicillins, monobactams, phosphonic acids, polymyxins, tetracyclines.

# 4. Source of infection:

- HCAI
- HAI
- CAI

#### 5. Infection site:

This refers to the origin of the infection (e.g. appendix, bladder, kidney, large intestine, lungs, liver, gall bladder, pancreas, peritoneum small intestine, stomach, urethra, other).

### 6. Antibiotic regimens

An antibiotic regimen is a planned therapeutic intervention which may involve 1 or more drugs.

# 7. Lines of therapy:

Each regimen is a line of therapy.

# 8. A new line of therapy is defined by:

- 1. Where a treatment regimen is discontinued, and a different regimen is started, the new regimen is considered a new line of therapy.
- 2. A line of treatment is considered finished when at least one antibiotic given in combination is modified.
- 3. Escalation, increasing the dosage, the dose or the unplanned addition or substitution of  $\geq 1$  drug(s) in an existing regimen is considered a new line of therapy.

Escalation after 4 days of treatment (dose increase or addition of another antibiotic for gram negative), will be considered as a failure

4. De-escalation, or reducing the dosage or eliminating  $\geq 1$  drug(s) from an existing regimen, or switching to oral antibiotics, is not considered a new line of therapy.

Stream lining (stop an antibiotic) or conversion to oral therapy will be considered as a success

#### 9. Treatment line number:

A new line of therapy starts when the antibiotic therapy is modified because an antibiotic is discontinued, the dose increased, patient is switched to an oral antibiotic therapy/regimen or a new antibiotic is added. Up to 5 lines of therapy will be collected. Assessment of treatment line will be based on generic name (i.e. active ingredient) of the drug (i.e. change in trade name with the same active ingredient, dose and strength will not be classified as a treatment line change).

# 10. The Deyo-Charlson Comorbidity Index (DCCI)

Table 3. outlines the Deyo-Charlson Comorbidity Index. To quantify comorbidity, the Deyo-Charlson Comorbidity score is computed by adding the weights that are assigned to the specific diagnoses. A score of 1 is attributed to myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular


disease, dementia, chronic obstructive pulmonary disease, rheumatologic disease, peptic ulcer disease, mild liver disease, depression, use of warfarin, hypertension and diabetes mild to moderate. The following diseases are scored as 2: hemiplegia or paraplegia, moderate or severe renal disease, skin ulcers/cellulitis, diabetes and complications and malignancy including leukemia and lymphoma. Moderate or severe liver disease is scored 3. Finally, a score of 6 is assigned to metastatic solid tumor, AIDS, and any transplant (bone marrow or sold organ).

Table 3. Deyo-Charlson Comorbidity Index

| Comorbidity | Deyo-Charlson Weight |
|-----------------------------------------------|----------------------|
| Myocardial Infarction | 1 |
| Congestive Heart Failure | 1 |
| Peripheral Vascular Disease | 1 |
| Cerebrovascular Disease (except hemiplegia) | 1 |
| Dementia | 1 |
| Chronic Obstructive Pulmonary Disease | 1 |
| Rheumatologic Disease | 1 |
| Peptic Ulcer Disease | 1 |
| Depression | 1 |
| Use of Warfarin | 1 |
| Hypertension | 1 |
| Mild Liver Disease | 1 |
| Diabetes Mild to Moderate | 1 |
| Hemiplegia | 2 |
| Paraplegia | 2 |
| Moderate or Severe Renal Disease | 2 |
| Diabetes with Complications | 2 |
| Skin Ulcers/Cellulitis | 2 |
| Malignancy (solid, non-metastatic) | 2 |
| Hematological malignancy (leukemia, lymphoma) | 2 |
| Moderate to Severe Liver Disease | 3 |
| Metastatic Solid Tumor | 6 |
| AIDS | 6 |
| Any transplant (bone marrow, solid organ) | 6 |

# 11. Index date

Start date of ceftazidime-avibactam.

### 12. Index infection

Infection treated with ceftazidime-avibactam.

# 13. Index hospitalization:

*Current hospitalization at time of index date.* 

# 14. Baseline period:


Statistical Analysis Plan

The baseline period is defined as the 90 days period preceding the date (inclusive) of diagnosis date for the index infection.

# 15. Follow-up period:

Each patient (in FAS72+) will be followed from index date, through their medical records up to 60 days after hospital discharge, in-hospital death, withdrawal from the study, or loss-to-follow-up, whichever occurs first.

# 16. Clinical success (cure):

- Resolution of all signs and symptoms of infection with no need for escalation of antimicrobials for gram-negative coverage.
- If there is stream lining. i.e., stopping an antibiotic treatment.
- If there is a de-escalation of antibiotic therapy unless ceftazidime-avibactam was used in a regimen with one or more other antibiotics and is the only antibiotic de-escalated.
- A clinical treatment outcome of "success" before discharge can be invalidated as "failure" if readmitted for recurrence of the same infection.
- Secondary infection will be not considered as failure.

# 17. Clinical failure:

Inadequate response to ceftazidime-avibactam therapy or resistant, worsening, or new recurrent signs and symptoms at the end of ceftazidime-avibactam therapy. Includes any of the following:

- In case of escalation within 4 days (addition of another antibiotic for gramnegative).
- Antimicrobial escalation (with ceftazidime-avibactam or an additional antibiotic for gram-negative coverage within 4 days).
- Discontinuation of ceftazidime-avibactam without clinical cure (e.g. AE, insufficient effect).
- Readmission to a hospital with the same infection within 60 days of the initial hospital discharge date.
- cIAI patient who required an additional unplanned source control procedure after ceftazidime-avibactam initiation.

A clinical treatment "failure" at any time cannot be redeemed

Note: Source control procedure: additional procedure (surgical, percutaneous) to control the infection, e.g. abscess drainage. All patients with cIAI are expected to have at least one source control procedure before or at start of the antibiotics.

#### 18. Clinical indeterminate:

There is not enough information to conclude whether the antibiotic regimen containing ceftazidime-avibactam was a clinical failure or a success.

# 19. Microbiological success:

- Eradication: Absence of causative pathogen from appropriately obtained specimens at the site of infection.
- Presumed eradication: Repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure (clinical success).
- Colonization: Detection of a new pathogen from the site of infection during therapy without the need for antimicrobial treatment or superinfection with a


Statistical Analysis Plan

microbiological agent outside the treatment spectrum of ceftazidimeavibactam (Gram+/fungi).

# 20. Microbiological failure:

- Verified persistence: The failure to eradicate the original pathogen from the site of isolation after completion of therapy.
- Presumed persistence: Absence of appropriate material for culture or absence of results of control microbiological tests coupled with lack of clinical improvement after a pathogen was initially isolated.
- Persistence with increasing minimal inhibitory concentration: Continued presence of the causative organism in culture during or upon completion of treatment with intravenous (IV) study therapy that displays a ≥4-fold higher minimum inhibitory concentration (MIC) to IV study therapy after treatment with IV study therapy.

# 21. Emergent infections:

- Superinfection: Detection of a new pathogen from the site of infection during therapy with the need for antimicrobial treatment.
- New Infection:
  - o Detection of a new pathogen from the site of infection after therapy with the need for antimicrobial treatment.
  - o Detection of a new pathogen on a different site.

# 22. Multi-bacteria infections:

For patients with multi-bacterial infections, the list of bacteria that must be considered pathogens.

# 23. Microbiological unevaluable:

• Unevaluable: Patients without cultures or evident pathogens from the presumed site of infection.

# **24.** *Hospital LOS* will be calculated as:

- 1) the total number of consecutive days the patient was treated in the hospital from admission to discharge during their initial hospitalization;
- 2) the total number of hospital days between diagnosis of infection and discharge;
- 3) the total number of days the patient was treated in the hospital after ceftazidime-avibactam initiation up to hospital discharge, including the first day of treatment.

Hospital LOS is defined as: (Date of hospital discharge - Date of hospital admission) +1 day.

- 25. ICU LOS will be calculated as: 1) the total number of consecutive or nonconsecutive days the patient was treated in the ICU during their initial hospitalization; and 2) the total number of days the patient was treated in the ICU after ceftazidime-avibactam initiation, including the first day of treatment. ICU LOS is defined as: (Date of ICU discharge - Date of ICU admission) +1 day.

26. In-hospital mortality rate is defined as: (# of patients who died in-hospital from index infection) / (total # of patients who received treatment with ceftazidime-


Statistical Analysis Plan

avibactam).

- **27.** Cumulative mortality rate at 30 days post-discharge is defined as: (# patients who died in-hospital or within 30 days post-discharge for the index hospitalization.) / (total # of patients who received treatment with ceftazidime-avibactam).
- **28.** Cumulative mortality rate at 60 days post-discharge is defined as: (# patients who died in-hospital or within 60 days post-discharge for the index hospitalization.) / (total # of patients who received treatment with ceftazidime-avibactam).
- **29.** *Duration (days) of an event* = stop date of event start date of event + 1. Note: Duration =1 day, if stop date = start date.
- **30.** *Total cumulative dose* (in ml or mg) of ceftazidime-avibactam or other antibiotics is defined as the sum of all doses received over the follow-up period.

#### **6 HANDLING OF MISSING VALUES**

Missing data will not be imputed, and data will be analyzed and presented as they are recorded in the eCRF as they were entered in the study database following resolution of all queries from data management. The number of missing cases will be reported for each variable of interest in the analysis. Patients with completely missing data for a variable will be excluded from the denominator when calculating proportions involving observed data for that variable.

For partial dates, a missing day element will default to the 15th of the month. Any event date occurring prior to the index hospitalization will not be imputed. Any event date occurring during the index hospitalization period must not be imputed beyond patient discharge or death during hospitalization. Any event occurring after discharge cannot be

imputed on the left prior to discharge and on the right after the 60 days of follow-up. See <u>Appendix</u> for additional rules for partial dates.

All data, including missing data, will be used for analysis of clinical outcomes. In data listings, all partial dates will be reported with the same precision as they appear in the eCRF.

#### 7 STATISTICAL METHODS

Unless otherwise specified, continuous/quantitative variables will be summarized using descriptive statistics which will include the number of patients with data to be summarized (n), mean, standard deviation (SD), 95% confidence interval (CI), median, first quartile (Q1) and third quartile (Q3), minimum and maximum.

All categorical/qualitative data will be presented using frequency counts and percentage with exact 95% CIs. The total number of patients with non-missing data (N) will be used as the denominator for percentage calculations, unless otherwise specified. Percentages equal to 100 will be presented as 100% and the percentage will not be presented for zero frequencies.


Statistical Analysis Plan

Missing data will be described in all summaries. Summary statistics will be displayed with decimal places as per Table 4.

**Table 4. Decimal Placees for Table Shells** 

| Description | Characteristic | Number of decimal places |
|---|---|---|
| Count | N | 0 |
| Count corresponding to the | N | 0 |
| number of subject for a group | | |
| Percentage | % | 1* |
| Mean, Median, First quartile, | Mean, Median, Q1, Q3 | As in CRF + 1 |
| Third quartile | | |
| Standard deviation | SD | As in CRF + 2 |
| Confidence interval | CI (LL, UL) | 1 |
| Minimum, maximum | Min, Max | As in CRF |
| p-value | p-value | 4, e.g. 0.0001. If the p-value |
| | | is rounded to below 0.0001 |
| | | then write as p<0.0001 |

\*Number of decimal places maybe 2, if necessary; CI lower limit (LL), CI upper limit (UL), CRF=case report form, Min= minimum, Max= maximum, Q1= quartile 1, and Q3=quartile 3. If there is no observation, a hyphen '-' will be displayed with no other statistics. If there is only one observation, the SD will be displayed as a hyphen '-'.

All computations and generation of Tables, Listings and Data for figures will be performed using SAS® Version 9.4 or higher (SAS Institute, Cary, NC, USA).

# 8 STATISTICAL ANALYSES

All analyses will be carried out separately for Europe and Latin America regions. Finally, on completion of the separate regional analyses, a pooled analysis combining data from both regions will be carried out.

#### 8.1 GENERAL CONSIDERATIONS

A detailed flow diagram will be provided to describe the patient selection process.

Antibiotic regimens including ceftazidime-avibactam will be examined.

All analyses, unless stated otherwise, will be performed among patients with exposure to ceftazidime-avibactam ≥72 hours (i.e., using the dataset FAS72+). Results will be presented overall and stratified by indication. For each analysis, there will an overall table that includes all countries and separate tables per country. The indication are: cIAI, cUTI, HAP/VAP, and other (use the primary diagnosis).

The effectiveness outcomes (see Section 4.5) will also be stratified by bacteria (*Escherichia coli*, *Klebsiella* spp., *Enterobacter* spp., *Pseudomonas* spp., and others).


Statistical Analysis Plan

A subgroup of patients with <72 hours of ceftazidime-avibactam exposure will be analysed to examine patient, infection, treatment characteristics, safety, and mortality. These analyses will be based on data from FAS72-.

Descriptive statistics will be used to summarize the baseline characteristics (study entry), treatment patterns (e.g. dosage, indications, infection source), effectiveness (e.g. clinical and microbiological outcomes), and safety (e.g. mortality, AEs) of ceftazidime-avibactam and healthcare resource utilization by patients prescribed ceftazidime-avibactam.

AEs will be recorded and summarized as the proportion of patients with each safety event out of all treated patients. Hospital readmissions will be analyzed as the proportion of patients readmitted to the hospital for recurrent infection out of all patients discharged from the initial hospitalization.

The Tables, Listings and Figure shells will be provided in a separate document. For the list of Tables see Section 12, and for the list of Listings see Section 13.

#### 8.2 SITE CHARACTERISTICS

 Site characteristics wiil be summarized overall and by country (variables described Section 4.1).

#### 8.3 PATIENT DISPOSITION

Summary statistics including number and percentages for the enrolled population will be presented for the following variables:

- Patients who included in the study.
- Patients in FAS population.
- Patients' study completion status and primary reasons for not completing the study.

#### 8.4 BASELINE DEMOGRAPHIC CHARACTERISTICS

The baseline charecteristics will be summarized by patients overall, by country and by indication..

- The number of enrolled patients.
- Socio-demographics data and risk factors of enrolled patients.

Variables are described Section 4.2

#### 8.5 BASELINE CLINICAL CHARACTERISTICS

- Recent medical history, overall, stratified by country and indication:
  - o Prior hospitalizations (within 90 days of index hospitalization).
    - Primary diagnosis at discharge.
    - LOS (days) of prior hospitalization.
  - o Prior healthcare procedures (within 30 days of index hospitalization).


Statistical Analysis Plan

- Number of procedure by type.
- History of antibiotic exposure overall, stratified by country and indication:
  - Prior antibiotics by class and molecule (within 90 days of index hospitalization).
  - o Reasons for treatment (therapeutic or prophylactic).
  - Duration of use of these antibiotics.
- Pre-treatment disease severity (APACHE score if available).
- Comorbidities will be described according to the list of comorbidities presented in Table 3, and by a summary of the DCCI index.
- Indwelling devices that the patient had at the time of the infection diagnosis.

Variables are described in Section 4.3.

#### 8.6 PATTERN OF USE OF CEFTAZIDIME-AVIBACTAM

# 8.6.1 Source of infection

Results will be presented overall stratified by country, indication, and bacteria. Descriptive analysis of the source of infection (HAI, HCAI and CAI).

# 8.6.2 Indication for ceftazidime-avibactam

Results will be presented, overall, and stratified by country and bacteria. Indication for ceftazidime-avibactam prescription (will vary depending on country local label) Descriptive analysis of the indication for ceftazidime-avibactam:

- o cIAI, cUTI, HAP, VAP, other
- o Initial site of infection (organ).

Descriptive analysis of the Indication for ceftazidime-avibactam Other (this indication is not approved in all participating countries):

- o Type of infection (e.g., SSI, CLABSI, primary BSI, meningitis, other)
- o Initial site of infection (organ).

#### 8.6.3 Antibiotics used for index infection before ceftazidime-avibactam initiation

The outcome of each line of therapy used for gram-negative coverage will be determined. The addition, modification or discontinuation of any antibiotic for coverage of gram-positive microorganisms co-prescribed with ceftazidime avibactam will be described but will not affect the outcome of the antibiotic regimen targeted at gram-negative microorganisms.

Results will be presented overall and stratified by country and indication (variables described Section 4.4).

Tables will include:

- Type of antibiotic by class and by molecule
- Dose
- Duration (days)


Statistical Analysis Plan

- Frequency of administration
- Route of administration
- Reason for initiating
- Reason for discontinuation

#### 8.6.4 <u>Use of ceftazidime-avibactam</u>

Results will be presented overall, and stratified by country, indication, and bacteria (variables described Section 4.4).

# Tables will include:

- Dose
- Duration of treatment (days)
- Duration of dose administration
- Frequency of administration
- Route of administration
- Reason for initiating
- Reason for discontinuation

# 8.6.5 Concomitant antibiotic therapy during index hospitalization

Results will be presented and, overall, and stratified by country and indication (variables described Section 4.4).

#### Tables will include:

- Type of antibiotic by class and by molecule
- Dose
- Duration of treatment (days)
- Frequency of administration
- Route of administration
- Reason for initiating
- Reason for discontinuation

# 8.6.6 Antibiotic therapy after ceftazidime-avibactam during the index hospitalization:

Results will be presented and, overall, and stratified by country and indication.

#### Tables will include:

- Type of antibiotic by class and by molecule
- Dose
- Duration of treatment (days)
- Frequency of administration
- Route of administration
- Reason for initiating
- Reason for discontinuation


Statistical Analysis Plan

# 8.7 MICROBIOLOGICAL EVALUATION

This will capture pre-treatment microbiology sample and results, *i.e.* microbiological culture(s) of the index infection within 5 days prior to ceftazidime-avibactam initiation. Results will be presented, overall, and stratified by country and indication.

Frequency distributions of:

- Timing of sample collection,
- Type of specimen,
- Any fungal pathogens identified,
- Number of bacterial pathogens identified,
- Bacterial pathogens identified.

Frequency distributions of:

Resistance of pathogen to antibiotics identified by drug class and antibiotic.

Pathogen susceptibility Tables will include:

- Pathogens
- Antibiotic susceptibility tests

#### 8.8 EFFECTIVENESS

#### 8.8.1 Clinical outcomes

Clinical outcomes (success, failure, indeterminate) will be described at 30 days and at 60 days post-discharge according to the evaluation of the physician and based on the definitions mentioned in Section 5. In case of missing data for readmission to hospital (at 30 days or at 60 days post-discharge), the rules described in the Table 5 will be applied.

Table 5. Clinical Outcomes Missing Data Rules at 30 Days or at 60 Days Post-Discharge

| Clinical Outcome Missing Outcome | | Computed Clinical Outcome |
|---|---|---|
| Success (cure) | Readmission for index infection | Indeterminate |
| Failure | Readmission for index infection | Failure |
| Indeterminate | Readmission for index infection | Indeterminate |

Note: Readmission information based on paper by Casapao AM, Davis SL, Barr VO, et al. Large retrospective evaluation of the effectiveness and safety of ceftaroline fosamil therapy. Antimicrob Agents Chemother. 2014;58(5):2541-6.

Results will be presented stratified by country, indication and bacteria.

Frequency distributions of:

- Clinical evaluation: success, failure or indeterminate
- Reasons for failure, if applicable.

For logistic regression, outcomes will be coded as follows:

• 1 = Success


Statistical Analysis Plan

#### • 0 = Failure

Indeterminate set to missing for logistic regression.

Based on the number and reasons for indeterminate results in the data, analysis with indeterminate as a level in a multinomial logistic may also be performed. Variables with p < 0.20 in the univariate analysis will be included in multivariable regression analysis as potential risk factors will be used as covariates in the multivariable analysis, regardless of their univariate or multivariable p-value. The final model will include variables with p-value < 0.2, after backward selection.

Potential risk factors include age, gender, country, employment status, BMI, hospitalization within 90 days prior to the index date, LOS of recent hospitalization, history of antibiotic exposure (yes/no), treated with beta-lactam within the past 3 months duration, of recent antibiotic exposure (yes/no), recent healthcare procedure (yes/no), recent healthcare procedure (type), pre-treatment disease severity, foreign travel, DCCI, number of comorbidities, source of infection (HAI, HCAI, CAI), bacteria (*Escherichia coli, Klebsiella* spp., *Acinetobacter* spp., *Enterobacter* spp., *Pseudomonas* spp., and others), pregnancy (yes/no, for females), alcohol use (yes/no), smoker (yes/no), patient's infection by multi-resistant pathogen.

Note: Acinetobacter spp. a risk factor for failure as zavicefta is not active against the Acinetobacter spp.

# 8.8.2 Microbiological outcomes

Results will be presented, overall, and stratified by country, indication, and bacteria.

Microbiological treatment outcome is *stricto sensu*; it is solely evaluated within the hospital stay (actually only during 14 days following the first dose of zavicefta) and there are no microbiology or mandatory sampling, but failure may be assumed in case of hospital readmission due to same infection or secondary infection (see definitions in Section 5).

Reasons for initiating or discontinuing antibiotic therapy (any line) include but are not limited to AE, perceived clinical failure, isolation of a resistant pathogen, secondary infection requiring regimen change, switch to oral therapy, de-escalation, cure, death.

For a given patient, all lines of therapy that include ceftazidime-avibactam will be evaluated altogether for the final microbiological outcome. Results will be presented overall, stratified by country and the source of the index infection (HAI, HCAI, and CAI).


Statistical Analysis Plan

# 8.8.3 Prevalence of hospital readmissions

Prevalence of hospital readmissions for recurrence of the index infection within 30 and 60 days of hospital discharge among patients treated with ceftazidime-avibactam.

- Frequency distributions of:
  - o readmissions within 60 days
    - reason for readmission
  - o readmissions within 30 days
    - reason for readmission
- Summary of the number of days readmitted.
- Prevalence rates of readmission for index infection at 30 days and 60 days postdischarge.

Prevalence of hospital readmissions; analyzed as the proportion of patients readmitted to the hospital for recurrence of the index infection out of all patients discharged from the initial hospitalization.

Results will be presented overall, stratified by country, indication, and bacteria.

#### 8.9 MORTALITY

Descriptive analysis of in-hospital mortality, and 60-day and 30-day mortality post hospital discharge, following index hospitalization.

- 1. Frequency distributions of:
  - a. Time of death:
    - In-hospital, i.e. after treatment initiation but before hospital discharge
    - In-hospital and up to 30 days after hospital discharge
    - In-hospital and up to 60 days after hospital discharge
    - Unknown/lost to follow-up
    - After end of ceftazidime-avibactam treatment
    - After end of antibiotic treatment.
  - b. Cause of death
- 2. Number of days from treatment initiation with ceftazidime-avibactam to death, overall, and by cause of death.
- 3. Mortality rates in-hospital, and between hospital discharge and 30 and 60 days post-discharge.
- 4. Cumulative mortality rates up to 30 and 60 days post-discharge, including inhospital mortality.

Results will be presented stratified by country, indication, and bacteria.

#### 8.10 HEALTHCARE RESOURCE UTILIZATION

#### 8.10.1 Hospital length of stay

- Frequency distributions for initial hospitalization of:
  - o Mode of admission,
  - Source of admission,


- Ward admitted to,
- Wards visited.
- o Diagnosis at admission,
- o Diagnosis at discharge,
- o Patients discharge by end of study.
- Frequency distributions for ICU admission.
- Summary of consecutive hospital LOS from hospital admission to hospital discharge.
- Summary of hospital LOS from infection diagnosis to hospital discharge.
- Summary of hospital LOS from treatment initiation with ceftazidime-avibactam to hospital discharge.
- Summary of consecutive or non-consecutive ICU LOS from ICU admission to ICU discharge.
- Summary of ICU LOS from treatment initiation with ceftazidime-avibactam to ICU discharge.

Results will be presented overall, stratified by country, indication, and bacteria.

# 8.10.2 Resource utilization

Healthcare resource utilization data (medical/surgical/percutaneous procedures, CT/MRI imaging, days of mechanical ventilation, days of dialysis) will be abstracted from the patient medical records.

- Frequency distributions of healthcare resource utilization during initial hospitalization:
  - o any resource use,
  - o resource utilized:
    - mechanical ventilation
    - hemodialysis:
      - intermittent or continuous renal replacement therapy
        - o number of episodes
    - CTCT/MRI imaging
    - tracheostomy
  - o surgical intervention:
    - type
    - indication
    - procedure performed to control infection?
  - o percutaneous procedures:
    - type
    - was procedure performed to control infection?
  - o other procedures
    - type
    - was procedure performed to control infection?


Statistical Analysis Plan

- Summary of number of days on mechanical ventilation
- Summary of number of days on intermittent or continuous renal replacement therapy

Results will be presented overall, stratified by country and indication. Safety

#### 8.11 ADVERSE EVENTS

AEs and SAEs will be summarized as the proportion of patients with each safety event out of all treated patients. Results will be presented, overall, and stratified by country and indication. Tables will include:

- AE term
- LOS of AE
- Relationship with ceftazidime-avibactam
- Serious AE with criteria of seriousness

Safety data will be summarized by using counts and percentages.

### 9 PATIENTS WITH <72 HOURS OF CEFTAZIDIME-AVIBACTAM EXPOSURE

#### 9.1 DEMOGRAPHIC CHARACTESITICS

- Age
- Sex

#### 9.2 SOURCE OF INFECTION

Results will be presented, overall, and stratified by country and indication. Descriptive analysis of the source of infection (HAI, HCAI, and CAI).

#### 9.3 INDICATION FOR CEFTAZIDIME-AVIBACTAM

Results will be presented by country and indication.

Descriptive analysis of the indication for ceftazidime-avibactam:

- o cIAI, cUTI, HAP/VAP, other
- o Initial site of infection (organ).

Descriptive analysis of the Indication for ceftazidime-avibactam Other

- o Type of infection (e.g., SSI, CLABSI, primary BSI, meningitis, other)
- o Initial site of infection (organ).

#### 9.4 USE OF CEFTAZIDIME-AVIBACTAM

Results will be presented overall, stratified by country, indication, and bacteria. Variables described Section 4.4.

Tables will include:

- Dose
- Duration of treatment (days)
- Duration of dose administration


# C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

NIS Protocol C3591031

Statistical Analysis Plan

- Frequency of administration
- Route of administration
- Reason for initiating
- Reason for discontinuation

#### 9.5 IN-HOSPITAL MORTALITY

- In-hospital mortality occurring after treatment initiation but before hospital discharge.
  - o Numbers of days after treatment initiation
  - o Cause of death.

Results will be presented stratified by country, indication, and bacteria.

#### 10 SAFETY

AEs and SAEs will be summarized as the proportion of patients with each safety event out of all treated patients. Results will be presented overall, stratified by country and indication. Tables will include:

- AE term
- LOS of AE
- Relationship with ceftazidime-avibactam, concomitant drug or other Pfizer drug
- Serious AE with criteria of seriousness
- Outcome (recovered, resolved, fatal...)

.


Statistical Analysis Plan

#### 11 REFERENCES

- 1. Mazuski JE, Gasink LB, Armstrong J, Broadhurst H, Stone GG, Rank D, et al. Efficacy and Safety of Ceftazidime-Avibactam Plus Metronidazole Versus Meropenem in the Treatment of Complicated Intra-abdominal Infection: Results From a Randomized, Controlled, Double-Blind, Phase 3 Program. Clin Infect Dis. 2016;62(11):1380-9.
- 2. Torres A, Zhong N, Pachl J, Timsit JF, Kollef M, Chen Z, et al. Ceftazidime-avibactam versus meropenem in nosocomial pneumonia, including ventilator-associated pneumonia (REPROVE): a randomised, double-blind, phase 3 non-inferiority trial. Lancet Infect Dis. 2018;18(3):285-95.
- 3. Wagenlehner FM, Sobel JD, Newell P, Armstrong J, Huang X, Stone GG, et al. Ceftazidime-avibactam Versus Doripenem for the Treatment of Complicated Urinary Tract Infections, Including Acute Pyelonephritis: RECAPTURE, a Phase 3 Randomized Trial Program. Clin Infect Dis. 2016;63(6):754-62.
- 4. Clopper CJ, Pearson ES. The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Biometrika. 1934;26(4):404-13.


Statistical Analysis Plan

#### 12 LIST OF TABLE SHELLS

| Table 1 | Site Characteristics by Country (FAS) |
|---|---|
| Table 1.1 | Site Characteristics Gram-Negative Resistance Patterns by Country (FAS) |
| Table 2 | Patients Disposition by Indication Overall (ENR) |
| Table 2.1 | Patients Disposition by Indication in xxxxa (ENR) |
| Table 3 | Patients by Indication Overall (FAS72+ and FAS72-) |
| Table 3.1 | Patients by Indication in xxxxa (FAS72+ and FAS72-) |
| Table 4 | Demographic and Baseline Characteristics by Indication Overall (FAS72+) |
| Table 4.1 | Demographic and Baseline Characteristics by Indication in xxxxa (FAS72+) |
| Table 4.2 | Baseline Demographic Characteristics of Patients Exposed to Ceftazidime-Avibactam for <72 hours by Indication Overall (FAS72-) |
| Table 4.3 | Baseline Demographic Characteristics of Patients Exposed to Ceftazidime-<br>Avibactam for <72 Hours by Indication in xxxxa (FAS72-) |
| Table 5 | Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication Overall (FAS72+) |
| Table 5.1 | Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication in xxxxa (FAS72+) |
| Table 5.2 | Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication Overall (FAS72-) |
| Table 5.3 | Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication in xxxxa (FAS72-) |
| Table 6 | Additional Risk Factors by Indication Overall (FAS72+) |
| Table 6.1 | Additional Risk Factors by Indication in xxxxa (FAS72+) |
| Table 7 | Comorbidities by Indication Overall (FAS72+) |
| Table 7.1 | Comorbidities by Indication in xxxxa (FAS72+) |
| Table 8 | Source of Infection by Indication Overall (FAS72+) |
| Table 8.1 | Source of Infection by Indication in xxxxa (FAS72+) |
| Table 9 | Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) in Patients Infected by Bacteria Overall (FAS72+) |
| Table 9.1 | Diagnoses and symptoms associated with UTI (including pyelonephritis) in patients Infected by Bacteria in xxxxa (FAS72+) |
| Table 9.2 | Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) for Patients with Ceftazidime-Avibactam Exposure <72 Hours Bacteria Overall (FAS72-) |
| Table 9.3 | Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) for Patients with Ceftazidime-Avibactam Exposure <72 Hours Bacteria in xxxxa (FAS72-) |
| Table 10 | Diagnoses and Symptoms Associated with IAI in Patients Infected by Bacteria Overall (FAS72+) |
| Table 10.1 | Diagnoses and symptoms associated with IAI in Patients Infected by Bacteria in xxxxa (FAS72+) |
| Table 10.2 | Diagnoses and Symptoms Associated with IAI in Patients Infected by Bacteria for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-) |
| Table 10.3 | Diagnoses and Symptoms Associated with IAI in Patients Infected by Bacteria for Patients with Ceftazidime-Avibactam Exposure <72 Hours in xxxxa (FAS72-) |

Statistical Analysis Plan

| Table 11 | Diagnoses and Symptoms of NP Associated with HAP/VAP in Patients Infected by Bacteria Overall (FAS72+) |
|---|---|
| Table 11.1 | Diagnoses and Symptoms of NP Associated with HAP/VAP in Patients Infected by Bacteria in xxxxa (FAS72+) |
| Table 11.2 | Diagnoses and Symptoms of NP Associated with HAP/VAP in Patients Infected by Bacteria for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-) |
| Table 11.3 | Diagnoses and Symptoms of NP Associated with HAP/VAP in Patients Infected by Bacteria for Patients with Ceftazidime-Avibactam Exposure <72 Hours in xxxxa (FAS72-) |
| Table 12 | Diagnoses and Symptoms Associated with Other Indication in Patients Infected by Bacteria Overall (FAS72+) |
| Table 12.1 | Diagnoses and Symptoms Associated with Other Indication in Patients Infected by Bacteria in xxxxa (FAS72+) |
| Table 12.2 | Diagnoses and Symptoms of NP Associated with Other Indication in Patients Infected by Bacteria for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-) |
| Table 12.3 | Diagnoses and Symptoms of NP Associated with Other Indication in Patients Infected by Bacteria for Patients with Ceftazidime-Avibactam Exposure <72 Hours in xxxxa (FAS72-) |
| Table 13 | Initial Hospitalization by Indication Overall (FAS72+) |
| Table 13.1 | Initial Hospitalization by Indication in xxxxa (FAS72+) |
| Table 14 | Healthcare Resource Utilization by Indication Overall (FAS72+) |
| Table 14.1 | Healthcare Resource Utilization by Indication in xxxxa (FAS72+) |
| Table 15 | Antibiotic Therapy: Prior Lines of Treatment Prior to Ceftazidime-Avibactam by Indication Overall (FAS72+) |
| Table 15.1 | Antibiotic Therapy: Prior Lines of Treatment Prior to Ceftazidime-Avibactam by Indication in xxxxa (FAS72+) |
| Table 16 | Ceftazidime-Avibactam Usage by Indication Overall (FAS72+) |
| Table 16.1 | Ceftazidime-Avibactam Usage by Indication in xxxxa (FAS72+) |
| Table 16.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication Overall (FAS72-) |
| Table 16.3 | Ceftazidime-Avibactam Usage <72 Hours by Indication in xxxxa (FAS72-) |
| Table 17 | Ceftazidime-Avibactam by Indication in Patients Infected by Escherichia coli<br>Overall (FAS72+) |
| Table 17.1 | Ceftazidime-Avibactam by Indication in Patients Infected by Escherichia coli in xxxxa (FAS72+) |
| Table 17.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Escherichia coli Overall (FAS72-) |
| Table 17.3 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Escherichia coli in xxxxa (FAS72-) |
| Table 18 | Ceftazidime-Avibactam by Indication in Patients Infected by Klebsiella spp. Overall (FAS72+) |
| Table 18.1 | Ceftazidime-Avibactam by Indication in Patients Infected by Klebsiella spp. in xxxxa (FAS72+) |
| Table 18.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Klebsiella spp. Overall (FAS72-) |
| Table 18.3 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Klebsiella spp. in xxxxa (FAS72-) |


# C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| ` | NIS Protocol C3591031 | Statistical Analysis Plan |
|---|-----------------------|---------------------------|

| Table 19 | Ceftazidime-Avibactam by Indication in Patients Infected by Enterobacter spp. |
|---|---|
| 1 4016 19 | Overall (FAS72+) |
| Table 19.1 | Ceftazidime-Avibactam by Indication in Patients Infected by Enterobacter spp. in xxxxa (FAS72+) |
| Table 19.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Enterobacter spp. Overall (FAS72-) |
| Table 19.3 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Enterobacter spp. in xxxxa (FAS72-) |
| Table 20 | Ceftazidime-Avibactam by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72+) |
| Table 20.1 | Ceftazidime-Avibactam by Indication in Patients Infected by Pseudomonas spp. ir xxxxa (FAS72+) |
| Table 20.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72-) |
| Table 20.3 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Pseudomonas spp. in xxxxa (FAS72-) |
| Table 21 | Ceftazidime-Avibactam by Indication in Patients Infected by Other Bacteria Overall (FAS72+) |
| Table 21.1 | Ceftazidime-Avibactam by Indication in Patients Infected by Other Bacteria in xxxxa (FAS72+) |
| Table 21.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Other Bacteria Overall (FAS72-) |
| Table 21.3 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Other Bacteria in xxxxa (FAS72-) |
| Table 22 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Other Bacteria Overall (FAS72-) |
| Table 22.1 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Other Bacteria in xxxxa |
| Table 22.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Other Bacteria Overall (FAS72-) |
| Table 22.3 | Ceftazidime-Avibactam Usage <72 Hours by Indication in Patients Infected by Other Bacteria in xxxxa (FAS72-) |
| Table 23 | Concomitant Antibiotic Therapy During Index Hospitalization by Indication Overall (FAS72+) |
| Table 23.1 | Concomitant Antibiotic Therapy During Index Hospitalization by Indication in xxxxa (FAS72+) |
| Table 24 | Microbiological Evaluation Before Initial Antibiotic Therapy by Indication Overa (FAS72+) |
| Table 24.1 | Microbiological Evaluation Before Initial Antibiotic Therapy by Indication in xxxxa (FAS72+) |
| Table 25 | Pathogen Susceptibility to Antibiotics by Indication Overall (MOD) |
| Table 25.1 | Pathogen Susceptibility to Antibiotics by Indication in xxxxa (MOD) |
| Table 26 | Multi-Drug Resistance Before Initial Antibiotic Therapy by Indication Overall (FAS72+) |
| Table 26.1 | Multi-Drug Resistance Before Initial Antibiotic Therapy by Indication in xxxxa (FAS72+) |
| Table 26.2 | Multi-Drug Resistance Before Initial Antibiotic Therapy by Indication Overall (FAS72-) |


| NIS | Protocol | C3591031 |
|------|-----------|----------|
| LATO | 1 1010001 | C3331031 |

Statistical Analysis Plan

| Table 26.3 | Multi-Drug Resistance Before Initial Antibiotic Therapy by Indication in xxxxa (FAS72-) |
|---|---|
| Table 27 | Multi-Drug Resistance Before Initial Antibiotic Therapy by bacteria Overall (FAS72+) |
| Γable 27.1 | Multi-Drug Resistance Before Initial Antibiotic Therapy by Bacteria in xxxxa (FAS72+) |
| Γable 27.2 | Multi-Drug Resistance Before Initial Antibiotic Therapy by Bacteria Overall (FAS72-) |
| Table 27.3 | Multi-Drug Resistance Before Initial Antibiotic Therapy by Bacteria in xxxxa (FAS72-) |
| Γable 28 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication Overall (COD) |
| Table 28.1 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in xxxxa (COD) |
| Table 29 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Escherichia coli Overall (COD) |
| Table 29.1 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Escherichia coli in xxxxa (COD) |
| Table 30 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Klebsiella spp. Overall (COD) |
| Table 30.1 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Klebsiella spp. in xxxxa (COD) |
| Γable 31 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Enterobacter spp. Overall (COD) |
| Гable 31.1 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Enterobacter spp. in xxxxa (COD) |
| Γable 32 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Pseudomonas spp. Overall (COD) |
| Гable 32.1 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Pseudomonas spp. in xxxxa (COD) |
| Table 33 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Other Bacteria Overall (COD) |
| Table 33.1 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Other Bacteria in xxxxa (COD) |
| Table 34 | Logistic Regression Univariate Model for Clinical Success at Hospital Discharge by Indication Overall (COD) |
| Гable 34.1 | Logistic Regression Univariate Model for Clinical Success at Hospital Discharge by Indication in xxxxa (COD) |
| Γable 35 | Logistic Regression Univariate Model for Clinical Success by Indication at 30-<br>Days Post-Discharge by Indication Overall |
| Γable 35.1 | Logistic Regression Univariate Model for Clinical Success by Indication at 30-<br>Days Post-Discharge by Indication in xxxxa |
| Γable 36 | Logistic Regression Univariate Model for Clinical Success by Indication at 60-<br>Days Post-Discharge by Indication Overall |
| Table 36.1 | Logistic Regression Univariate Model for Clinical Success by Indication at 60-<br>Days Post-Discharge by Indication in xxxxa |
| Table 37 | Logistic Regression Multivariable Model for Clinical Success by Indication Overall (COD) |
| Γable 37.1 | Logistic Regression Multivariable Model for Clinical Success by Indication in |

#### Statistical Analysis Plan

| | xxxxa (COD) |
|---|---|
| Table 38 | Logistic Regression Multivariable Model for Clinical Success by Indication at 30 Days Post-Discharge by Indication Overall |
| Table 38.1 | Logistic Regression Multivariable Model for Clinical Success by Indication at 30 Days Post-Discharge by Indication in xxxxa |
| Table 39 | Logistic Regression Multivariable Model for Clinical Success by Indication at 60 Days Post-Discharge by Indication Overall |
| Table 39.1 | Logistic Regression Multivariable Model for Clinical Success by Indication at 60 Days Post-Discharge by Indication in xxxxa |
| Table 40 | Microbiological Evaluation Outcome (Success, Failure, Emergent Infections) by Indication Overall (MOD) |
| Table 40.1 | Microbiological Evaluation Outcome by Indication in xxxxa (MOD) |
| Table 41 | Microbiological Evaluation Outcome by Indication in Patients Infected by Escherichia Coli Overall (MOD) |
| Table 41.1 | Microbiological Evaluation Outcome by Indication in Patients Infected by Escherichia Coli in Xxxxa (MOD) |
| Table 42 | Microbiological Evaluation Outcome by Indication in Patients Infected by Klebsiella Spp. Overall (MOD) |
| Table 42.1 | Microbiological Evaluation Outcome by Indication in Patients Infected by Klebsiella Spp. in Xxxxa (MOD) |
| Table 43 | Microbiological Evaluation Outcome by Indication in Patients Infected by Enterobacter Spp. Overall (MOD) |
| Table 43.1 | Microbiological Evaluation Outcome by Indication in Patients Infected by Enterobacter Spp. In Xxxxa (MOD) |
| Table 44 | Microbiological Evaluation Outcome by Indication in Patients Infected by Pseudomonas Spp. Overall (MOD) |
| Table 44.1 | Microbiological Evaluation Outcome by Indication in Patients Infected by Other Bacteria in Xxxxa (MOD) |
| Table 45 | Prevalence of Hospital Readmissions by Indication Overall (FAS72+) |
| Table 45.1 | Prevalence of Hospital Readmissions by Indication in xxxxa (FAS72+) |
| Table 46 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Escherichia Coli Overall (FAS72+) |
| Table 46.1 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Escherichia Coli in xxxxa (FAS72+) |
| Table 47 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Klebsiella Spp. Overall (FAS72+) |
| Table 47.1 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Klebsiella Spp. in xxxxa (FAS72+) |
| Table 48 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Enterobacter spp. Overall (FAS72+) |
| Table 48.1 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Enterobacter Spp. in xxxxa (FAS72+) |
| Table 49 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Pseudomonas Spp. Overall (FAS72+) |
| Table 49.1 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Pseudomonas Spp. in xxxxa (FAS72+) |
| Table 50 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Other Bacteria Overall (FAS72+) |


Statistical Analysis Plan

| Table 50.1 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Other |
|---|---|
| | Bacteria in xxxxa (FAS72+) |
| Table 51 | Vital Status and Mortality Rates by Indication Overall (FAS72+) |
| Table 51.1 | Vital Status and Mortality Rates by Indication in xxxxa (FAS72+) |
| Table 52 | Vital Status and Mortality Rates by Indication in Patients Infected by Escherichia |
| - | Coli Overall (FAS72+) |
| Table 52.1 | Vital Status and Mortality Rates by Indication in Patients Infected by |
| | EscherichiaCcoli in xxxxa (FAS72+) |
| Table 53 | Vital Status and Mortality Rates by Indication in Patients Infected by Klebsiella |
| | spp. Overall (FAS72+) |
| Table 53.1 | Vital Status and Mortality Rates by Indication in Patients Infected by Klebsiella |
| | Spp. in xxxxa (FAS72+) |
| Table 54 | Vital Status and Mortality Rates by Indication in Patients Infected by Enterobacter |
| | spp. Overall (FAS72+) |
| Table 54.1 | Vital Status and Mortality Rates by Indication in Patients Infected by Enterobacter |
| | Spp. in xxxxa (FAS72+) |
| Table 55 | Vital Status and Mortality Rates by Indication in Patients Infected by |
| | Pseudomonas spp. Overall (FAS72+) |
| Table 55.1 | Vital Status and Mortality Rates by Indication in Patients Infected by |
| | Pseudomonas Spp. in xxxxa (FAS72+) |
| Table 56 | Vital Status and Mortality Rates by Indication in Patients Infected by Other |
| | Bacteria Overall (FAS72+) |
| Table 56.1 | Vital Status and Mortality Rates by Indication in Patients Infected by Other |
| | Bacteria in xxxxa (FAS72+) |
| Table 57 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure |
| | <72 Hours by Indication Overall (FAS72-) |
| Table 57.1 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure |
| T 11 50 | <72 Hours by Indication in xxxxa (FAS72-) |
| Table 58 | Vital Status and Mortality Rates for Patients with Ceftazidime-Avibactam |
| | Exposure <72 Hours by Indication in Patients Infected by Escherichia Coli Overall |
| T.11. 50.1 | (FAS72-) |
| Table 58.1 | Vital Status and Mortality Rates for Patients with Ceftazidime-Avibactam |
| | Exposure <72 Hours by Indication in Patients Infected by Escherichia Coli in |
| Table 50 | XXXXa (FAS72-) Vital Status and Mantality Patas for Patients with Coffee idina Avilantem |
| Table 59 | Vital Status and Mortality Rates for Patients with Ceftazidime-Avibactam Exposure <72 Hours by Indication in Patients Infected by Klebsiella Spp. Overall |
| | (FAS72-) |
| Table 59.1 | Vital Status and Mortality Rates for Patients with Ceftazidime-Avibactam |
| 1 autc 39.1 | Exposure <72 Hours by Indication in Patients Infected by Klebsiella Spp. in xxxxa |
| | (FAS72-) |
| Table 60 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure |
| Table 00 | <72 Hours by Indication in Patients Infected by Enterobacter spp. Overall (FAS72- |
| | ) |
| Table 60.1 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure |
| 14010 00.1 | <72 Hours by Indication in Patients Infected by Enterobacter Spp. in xxxxa |
| | (FAS72-) |
| Table 61 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure |
| 01 | <72 Hours by Indication in Patients Infected by Pseudomonas Spp. Overall |
| | (FAS72-) |
| | Tage 10 of 17 |

| NIS I | Protocol | C3591 | 031 |
|-------|----------|-------|-----|

#### Statistical Analysis Plan

| Table 61.1 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure |
|---|---|
| | <72 Hours by Indication in Patients Infected by Pseudomonas Spp. in xxxxa<br>(FAS72-) |
| Table 62 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure <72 Hours by Indication in Patients Infected by Other Bacteria Overall (FAS72-) |
| Table 62.1 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure <72 Hours by Indication in Patients Infected by Other Bacteria in xxxxa (FAS72-) |
| Table 63 | Antibiotic Therapy After Ceftazidime-Avibactam During the Index Hospitalization by Indication Overall (FAS72+) |
| Table 63.1 | Antibiotic Therapy After Ceftazidime-Avibactam During the Index Hospitalization by Indication in xxxxa (FAS72+) |
| Table 64 | Adverse Drug Reactions by Indication Overall (FAS) |
| Table 64.1 | Adverse Drug Reactions by Indication in xxxxa (FAS) |
| Table 65 | Fatal Serious Adverse Drug Reactions by Indication Overall (FAS) |
| Table 65.1 | Fatal Serious Adverse Drug Reactions by Indication in xxxxa (FAS) |
| Table 66 | Adverse Drug Reactions by System Organ Class by Indication Overall (FAS) |
| Table 66.1 | Adverse Drug Reactions by System Organ Class by Indication in xxxxa (FAS) |
| Table 67 | Serious Adverse Drug Reactions by System Organ Class by Indication Overall (FAS) |
| Table 67.1 | Serious Adverse Drug Reactions by System Organ Class by Indication in xxxxa (FAS) |
| Table 68 | Fatal Serious Adverse Drug Reactions by System Organ Class by Indication Overall (FAS) |
| Table 68.1 | Fatal Serious Adverse Drug Reactions by System Organ Class by Indication in xxxxa (FAS) |
| Table 69 | Fatal Serious Adverse Drug Reactions Leading to Discontinuation of Ceftazidime-Avibactam by System Organ Class by Indication Overall (FAS) |
| Table 69.1 | Fatal Serious Adverse Drug Reactions Leading to Discontinuation of Ceftazidime-Avibactam by System Organ Class by Indication in xxxxa (FAS) |


Statistical Analysis Plan

#### 13 LIST OF LISTINGS

| Listing 1 | Site Characteristics (1) |
|---|---|
| Listing 2 | Site Characteristics (2) |
| Listing 3 | Demographic |
| Listing 4 | Indication Diagnosis of UTI (ENR) |
| Listing 5 | Indication Clinical Diagnosis of IAI |
| Listing 6 | Indication Nosocomial Pneumonia (NP) HAP- Hospital Associated Pneumonia |
| | (HAP)/ Ventilator-Associated Pneumonia (VAP) |
| Listing 7 | Indication Other |
| Listing 8 | Subject with Comorbidities |
| Listing 9 | Prior Antibiotic Therapy |
| Listing 10 | Prior Hospitalization |
| Listing 11 | Prior Healthcare Procedures (1) |
| Listing 12 | Prior Healthcare Procedures (2) |
| Listing 13 | Additional Risk Factors |
| Listing 14 | Antibiotic Therapy: Prior Lines of Treatment |
| Listing 15 | Pattern of use of Ceftazidime-Avibactam |
| Listing 16 | Concomitant Antibiotic Therapy |
| Listing 17 | Antibiotic Treatment After Ceftazidime-Avibactam |
| Listing 18 | Initial Hospitalization |
| Listing 19 | Healthcare Resource Utilization (1) |
| Listing 20 | Healthcare Resource Utilization (2) |
| Listing 21 | Treatment Evaluation for Initial Hospitalization, at 30-days and at 60-Days Post Discharge |
| Listing 22 | Microbiological Evaluation Outcome |
| Listing 23 | Disease Severity |
| Listing 24 | Hospital Readmissions |
| Listing 25 | Microbiology Sample Taken |
| Listing 26 | Microbiology Bacterial Pathogens Identified in Specimen Sampled |
| Listing 27 | Pathogen Susceptibility (1) |
| Listing 28 | Pathogen Susceptibility (2) |
| Listing 29 | Pathogen Susceptibility (3) |
| Listing 30 | Mortality and Cumulative Mortality in-Hospital,30-Days and 60-Days Post Discharge |
| Listing 31 | Adverse Drug Reactions |
| Listing 32 | Serious Adverse Drug Reactions |
| Listing 33 | Adverse Drug Reactions Leading to Treatment Discontinuation |
| Listing 34 | End of Chart Review |


Statistical Analysis Plan

#### 14 APPENDIX

#### 14.1 PARTIAL DATE CONVENTIONS

Imputed dates will not be presented in the listings.

**Table 6. Algorithm for Treatment Emergence of Adverse Events** 

| START DATE | STOP | ACTION |
|---|---|---|
| | DATE | |
| Known | Known | If start date < study medication (medication) start |
| | | date, then not TEAE |
| | | If start date >= study medication start date, then |
| | | TEAE |
| | | If Zavicefta is discontinued, then the start date of |
| | | TEAE should be >= date of initiation of the antibiotic |
| | D 11.1 | and <= date of discontinuation + 1. |
| | Partial | If start date < study medication start date, then not |
| | | TEAE |
| | | If start date >= study medication start date, then TEAE |
| | Missing | If start date < study medication start date, then not |
| | wiissing | TEAE |
| | | If start date >= study medication start date, then |
| | | TEAE |
| Partial, but known | Known | Not TEAE |
| components show that it | | |
| cannot be on or after | | |
| study medication start | | |
| date [1] | 1 | |
| | Partial | Not TEAE |
| | Missing | Not TEAE |
| Partial, could be on or | Known | If stop date < study medication start date, then not |
| after study medication | | TEAE |
| start date | | If stop date >= study medication start date, then |
| | 1 | TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day |
| | | of month if day unknown or 31st December if day |
| | | and month are unknown), then: |
| | | If stop date < study medication start date, then not TEAE |
| | | If stop date >= study medication start date, then |
| | | TEAE |
| | Missing | Assumed TEAE |


Statistical Analysis Plan

| START DATE | STOP<br>DATE | ACTION |
|---|---|---|
| | DITTE | |
| Missing | Known | If stop date < study medication start date, then not TEAE If stop date >= study medication start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study medication start date, then not TEAE If stop date >= study medication start date, then TEAE |
| | Missing | Assumed TEAE |

<sup>[1]</sup> E.g. if treatment start date is 18-11-2019 and AE date is UNK-12-2019 and since from the "known component" we know that regardless of the actual day, AE started always after treatment start date, therefore, it is a TEAE.

AE: Adverse event; TEAE: Treatment emergent event; UNK: Unknown


#### Statistical Analysis Plan - SAP - 28-Aug-2020

#### **Electronic Signature Manifestation**

This page is a manifestation of the electronic signature(s) used in compliance with the organization's electronic signature policies and procedures.

| Signer Full Name | Meaning of Signature | Date and Time |
|---|---|---|
| Juzer Lotya | Document Approval (I certify that I have the education, training and experience to perform this task) | 06 Aug 2020 08:17:18 UTC |
| Richard Chambers | Document Approval (I certify that I have the education, training and experience to perform this task) | 28 Aug 2020 15:13:13 UTC |

#### NON-INTERVENTIONAL STUDY PROTOCOL C3591031

# REAL-WORLD OBSERVATIONAL STUDY OF ZAVICEFTA® (CEFTAZIDIME-AVIBACTAM) TO CHARACTERIZE USE PATTERNS, EFFECTIVENESS AND SAFETY - EZTEAM STUDY

#### ANNOTATED SHELLS

Version: 2.0

Author: Juzer Lotya

**Date:** 11 January 2022


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

#### Table of Contents

| Table 1.2 Site Characteristics Gram-Negative Resistance Patterns by Country (FAS) | Description | of Global Rules: | 12 |
|---|---|---|---|
| Table 2 Patients Disposition by Indication Overall (ENR) ADSL where ENRFL = "Y" | Table 1.1 | Site Characteristics by Country (FAS) | 14 |
| Patients by Indication Overall (FAS72+ and FAS72-) | Table 1.2 | Site Characteristics Gram-Negative Resistance Patterns by Country (FAS) | 20 |
| Table 4.1 Demographic and Baseline Characteristics by Indication Overall (FAS72+) | Table 2 | Patients Disposition by Indication Overall (ENR) ADSL where ENRFL = "Y" | 23 |
| Table 4.2 Baseline Demographic Characteristics of Patients Exposed to Ceftazidime-Avibactam for <72 hours by Indication Overall (FAS72-)30 Table 5 Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication Overall (FAS72+) | Table 3 | Patients by Indication Overall (FAS72+ and FAS72-) | 27 |
| Table 5 Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication Overall (FAS72+) | Table 4.1 | Demographic and Baseline Characteristics by Indication Overall (FAS72+) | 28 |
| Table 6 Additional Risk Factors by Indication Overall (FAS72+) | Table 4.2 | Baseline Demographic Characteristics of Patients Exposed to Ceftazidime-Avibactam for <72 hours by Indication Overall (F | FAS72-)30 |
| Table 7 Comorbidities by Indication Overall (FAS72+) | Table 5 | Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication Overall (FAS72+) | 31 |
| Table 8.1 Source of Infection by Indication Overall (FAS72+) | Table 6 | Additional Risk Factors by Indication Overall (FAS72+) | 34 |
| Table 8.2 Source of Infection by Indication Overall (FAS72-) | Table 7 | Comorbidities by Indication Overall (FAS72+) | 37 |
| Table 8.3 Indication for Ceftazidime-Avibactam Overall (FAS72+ and FAS72-)44 | Table 8.1 | Source of Infection by Indication Overall (FAS72+) | 43 |
| | Table 8.2 | Source of Infection by Indication Overall (FAS72-) | 43 |
| Table 9.1 Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) by Bacteria Overall (FAS72+) | Table 8.3 | Indication for Ceftazidime-Avibactam Overall (FAS72+ and FAS72-) | 44 |
| | Table 9.1 | Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) by Bacteria Overall (FAS72+) | 46 |


Document:

Title: Annotated TLF Shells

Version Number: Version Date: V2.0 11 January 2022

#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### PLAN

| Table 9.2 | Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) for Patients with Ceftazidime-Avibactam Exposure <72 Hours (FAS72-)49 |
|---|---|
| Table 10.1 | Diagnoses and Symptoms Associated with IAI by Bacteria Overall (FAS72+)51 |
| Table 10.2 | Diagnoses and Symptoms Associated with IAI for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-)54 |
| Table 11.1 | Diagnoses and Symptoms of NP Associated with HAP/VAP by Bacteria Overall (FAS72+)56 |
| Table 11.2 | Diagnoses and Symptoms of NP Associated with HAP/VAP for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-) |
| Table 12.1 | Diagnoses and Symptoms Associated with Other Indication by Bacteria Overall (FAS72+)59 |
| Table 12.2 | Diagnoses and Symptoms of NP Associated with Other Indication for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-) |
| Table 13 | Initial Hospitalization by Indication Overall (FAS72+)63 |
| Table 14 | Healthcare Resource Utilization by Indication Overall (FAS72+)66 |
| Table 15 | Antibiotic Therapy: Prior Lines of Treatment Prior to Ceftazidime-Avibactam by Indication Overall (FAS72+) |
| Table 16.1 | Ceftazidime-Avibactam Usage by Indication Overall (FAS72+) |
| Table 16.2 | Ceftazidime-Avibactam Usage <72 Hours by Indication Overall (FAS72-)75 |
| Table 17.1 | Ceftazidime-Avibactam by Indication in Patients Infected by Escherichia coli Overall (FAS72+) |
| Table 17.2 | Ceftazidime-Avibactam by Indication in Patients Infected by Klebsiella spp. Overall (FAS72+) |
| Table 17.3 | Ceftazidime-Avibactam by Indication in Patients Infected by Enterobacter spp. Overall (FAS72+) |
| | Page <b>3</b> of <b>159</b> |
| Document: | Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications Title: Annotated TLF Shells Version Number: V2.0 Version Date: 11 January 2022 |

#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### **PLAN**

| Table 17.4 | Ceftazidime-Avibactam by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72+) | 76 |
|---|---|---|
| Table 17.5 | Ceftazidime-Avibactam by Indication in Patients Infected by Other Gram-negative Bacteria Overall (FAS72+) | 76 |
| Table 17.6 | Ceftazidime-Avibactam Usage >72 Hours by Indication in Patients with no pathogen identified (FAS72+) | 76 |
| Table 18 | Immunocompromised patients by indication (FAS72+) | 77 |
| Table 19 | Patients with primary/secondary Bacteriemia by indication (FAS72+) | 79 |
| Table 20 | Patients with lower dose of Zavicefta by indication (FAS72+) | 81 |
| Table 21 | Clinical Outcome for patients with COVID-19 diagnosis (FAS72+) | 82 |
| Table 22.1 | Microbiological Evaluation Before Initial Antibiotic Therapy by Indication Overall (FAS72+) | 83 |
| Table 22.2 | Clinical Microbiological Evaluation after initial antibiotic therapy but before ceftazidime-avibactam therapy by Indication Overall (FAS72+) | 97 |
| Table 22.3 | Clinical Microbiological Evaluation after initiation or during ceftazidime-avibactam therapy by Indication Overall (FAS72+) | 97 |
| Table 22.4 | Clinical Microbiological Evaluation after end of ceftazidime-avibactam therapy by Indication Overall (FAS72+) | 97 |
| Table 22.5 | Clinical Microbiological Evaluation after end of any antibiotic therapy by Indication Overall (FAS72+) | 97 |
| Table 22.6 | Latest Microbiological Evaluation before start of ceftazidime-avibactam therapy by Indication Overall (FAS72+) | 97 |
| Table 23.1.1 | Gram-negative Pathogen Susceptibility to Antibiotics by cIAI Overall (FAS72+) | 98 |
| Table 23.1.2 | Gram-negative Pathogen Susceptibility to Antibiotics by cUTI Overall (FAS72+) | 101 |
| Table 23.1.3 | Gram-negative Pathogen Susceptibility to Antibiotics by HAP/VAP Overall (FAS72+) | 101 |


Document:

Title: Annotated TLF Shells

Version Number: Version Date: V2.0

11 January 2022

# C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Table 23.1.5 | Gram-negative Pathogen Susceptibility to Antibiotics by All indications Overall (FAS72+) | 101 |
|---|---|---|
| Table 23.2.1 | Gram-negative Multi Drug Resistance for cIAI Overall (FAS72+) | 101 |
| Table 23.2.2 | Gram-negative Multi Drug Resistance for cUTI Overall (FAS72+) | 103 |
| Table 23.2.3 | Gram-negative Multi Drug Resistance for HAP/VAP Overall (FAS72+) | 103 |
| Table 23.2.4 | Gram-negative Multi Drug Resistance for Other Overall (FAS72+) | 103 |
| Table 23.2.5 | Gram-negative Multi Drug Resistance for All indications Overall (FAS72+) | 103 |
| Table 24.1.1 | Gram-negative Pathogen Susceptibility to Antibiotics by cIAI Europe (FAS72+) | 103 |
| Table 24.1.2 | Gram-negative Pathogen Susceptibility to Antibiotics by cUTI Europe (FAS72+) | 103 |
| Table 24.1.3 | Gram-negative Pathogen Susceptibility to Antibiotics by HAP/VAP Europe (FAS72+) | 103 |
| Table 24.1.4 | Gram-negative Pathogen Susceptibility to Antibiotics by Other Europe (FAS72+) | 103 |
| Table 24.1.5 | Gram-negative Pathogen Susceptibility to Antibiotics by All Indications Europe (FAS72+) | 103 |
| Table 24.2.1 | Gram-negative Multi Drug Resistance for cIAI in Europe (FAS72+) | 103 |
| Table 24.2.2 | Gram-negative Multi Drug Resistance for cUTI Europe (FAS72+) | 103 |
| Table 24.2.3 | Gram-negative Multi Drug Resistance for HAP/VAP Europe (FAS72+) | 103 |
| Table 24.2.4 | Gram-negative Multi Drug Resistance for Others Europe (FAS72+) | 103 |
| Table 24.2.5 | Gram-negative Multi Drug Resistance for All Indications Europe (FAS72+) | 103 |
| | | Page <b>5</b> of <b>159</b> |
| Document: | Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications Title: Annotated TLF Shells | |
| | Version Number: | V2.0 |
| | Version Date: | 11 January 2022 |

#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### **PLAN**

| Table 25.1.1 | Gram-negative Pathogen Susceptibility to Antibiotics for cIAI in LATAM (FAS72+) | 103 |
|---|---|---|
| Table 25.1.2 | Gram-negative Pathogen Susceptibility to Antibiotics for cUTI LATAM (FAS72+) | 103 |
| Table 25.1.3 | Gram-negative Pathogen Susceptibility to Antibiotics for HAP/VAP LATAM (FAS72+) | 103 |
| Table 25.1.4 | Gram-negative Pathogen Susceptibility to Antibiotics for Others LATAM (FAS72+) | 103 |
| Table 25.1.5 | Gram-negative Pathogen Susceptibility to Antibiotics for All Indications LATAM (FAS72+) | 103 |
| Table 25.2.1 | Gram-negative Multi Drug Resistance for cIAI in LATAM (FAS72+) | 103 |
| Table 25.2.2 | Gram-negative Multi Drug Resistance for cUTI LATAM (FAS72+) | 103 |
| Table 25.2.3 | Gram-negative Multi Drug Resistance for HAP/VAP LATAM (FAS72+) | 103 |
| Table 25.2.4 | Gram-negative Multi Drug Resistance for Others LATAM (FAS72+) | 103 |
| Table 25.2.5 | Gram-negative Multi Drug Resistance for All Indications LATAM (FAS72+) | 103 |
| Table 26 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication Overall (COD) | 104 |
| Table 26.1 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Escherichia coli Overall (COD) | 107 |
| Table 26.2 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Klebsiella spp. Overall (COD) | 107 |
| Table 26.3 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Enterobacter spp. Overall (COD) | 107 |


Document:

 $\label{thm:path:local} Path: $$ \underline{\CBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$$ 

Title: Annotated TLF Shells


#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### PLAN

| Document: | Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications Title: Annotated TLF Shells Version Number: Version Date: | V2.0<br>11 January 2022 |
|---|---|---|
| Table 32.3 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Enterobacter spp. Overall (FAS72 | Page <b>7</b> of <b>159</b> |
| Table 32.2 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Klebsiella spp. Overall (FAS72+) | 131 |
| Table 32.1 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Escherichia Coli Overall (FAS72+). | 131 |
| Table 32 | Prevalence of Hospital Readmissions by Indication Overall (FAS72+) | 129 |
| Table 31.5 | Microbiological Evaluation Outcome by Indication in Patients Infected by Other Gram-negative bacteria Ov | erall (MOD)128 |
| Table 31.4 | Microbiological Evaluation Outcome by Indication in Patients Infected by Pseudomonas spp. Overall (MOD) | 128 |
| Table 31.3 | Microbiological Evaluation Outcome by Indication in Patients Infected by Enterobacter spp. Overall (MOD). | 128 |
| Table 31.2 | Microbiological Evaluation Outcome by Indication in Patients Infected by Klebsiella spp. Overall (MOD) | 128 |
| Table 31.1 | Microbiological Evaluation Outcome by Indication in Patients Infected by Escherichia Coli Overall (MOD) | 128 |
| Table 31 | Microbiological Evaluation Outcome (Success, Failure, Emergent Infections) by Indication Overall (MOD) – | 128 |
| Table 30 | Logistic Regression Multivariable Model 2 for Clinical Success by Indication at Initial Hospitalization | 122 |
| Table 29 | Regression Univariate Model 2 for Clinical Success at Initial Hospitalization by Indication Overall (COD) | 118 |
| Table 28 | Logistic Regression Multivariable Model 1 for Clinical Success by Indication Overall (COD) | 113 |
| Table 27 | Logistic Regression Univariate Model 1 for Clinical Success at Initial Hospitalization by Indication Overall (CC | DD)108 |
| Table 26.5 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Other Gr<br>Overall (COD) | |
| Table 26.4 | Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Pseudon Overall (COD) | • • |

#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### PLAN

| Table 32.4 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72+) | 13 |
|---|---|---|
| Table 32.5 | Prevalence of Hospital Readmissions by Indication in Patients Infected by Other Gram-negative Bacteria Overall (FAS72+) | 132 |
| Table 32.6 | Prevalence of Hospital Readmissions by Indication in Patients Infected by no Pathogen Identified Overall (FAS72+) | <b>13</b> 1 |
| Table 33 | Vital Status and Mortality Rates by Indication Overall (FAS72+) | 132 |
| Table 33.1 | Vital Status and Mortality Rates by Indication in Patients Infected by Escherichia Coli Overall (FAS72+) | 133 |
| Table 33.2 | Vital Status and Mortality Rates by Indication in Patients Infected by Klebsiella spp. Overall (FAS72+) | 133 |
| Table 33.3 | Vital Status and Mortality Rates by Indication in Patients Infected by Enterobacter spp. Overall (FAS72+) | 133 |
| Table 33.4 | Vital Status and Mortality Rates by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72+) | 133 |
| Table 33.5 | Vital Status and Mortality Rates by Indication in Patients Infected by Other Gram-negative Bacteria Overall (FAS72+) | 133 |
| Table 33.6 | Vital Status and Mortality Rates by Indication by no Pathogen Identified Overall (FAS72+) | 133 |
| Table 34 | Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure <72 Hours by Indication Overall (FAS72- | -)134 |
| Table 35 | Antibiotic Therapy After Ceftazidime-Avibactam During the Index Hospitalization by Indication Overall (FAS72+) | 135 |
| Table 36 | Adverse Events by Indication Overall (FAS) | 137 |
| Table 36.1 | Adverse Events Related to Ceftazidime-Avibactam by Indication Overall (FAS) | 138 |
| Table 37 | Adverse Events by System Organ Class by Indication Overall (FAS) | 139 |
| Table 37.1 | Adverse Events Related to Ceftazidime-Avibactam by System Organ Class by Indication Overall (FAS) | 140 |
| Table 38 | Serious Adverse Events by System Organ Class by Indication Overall (FAS) | 141 |
| | Pag | ge <b>8</b> of <b>15</b> 9 |
| Document: | Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications Title: Annotated TLF Shells | |

Version Number: Version Date: V2.0

n Date:

11 January 2022

#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### PLAN

| Document: | Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications | |
|---|---|---|
| | | of <b>15</b> 9 |
| Listing 7. | Healthcare Procedures within 30 days prior to ceftazidime-avibactam initiation | 150 |
| Listing 6. | Prior Hospitalization | 150 |
| Listing 5. | Prior Antibiotic Therapy | 150 |
| Listing 4. | Subject with Comorbidities | 149 |
| Listing 3.4. | Indication Other | 149 |
| Listing 3.3. | Indication Nosocomial Pneumonia (NP) HAP- Hospital Associated Pneumonia (HAP)/ Ventilator-Associated Pneumonia (VAP). | 149 |
| Listing 3.2. | Indication Clinical Diagnosis of IAI | 148 |
| Listing 3.1. | Indication Diagnosis of UTI (ENR) | 148 |
| Listing 2. | Demographic | 148 |
| Listing 1.2. | Site Characteristics (2) | 147 |
| Listing 1.1. | Site Characteristics (1) | 147 |
| Table 40.1 | Adverse Events Related to Ceftazidime-Avibactam Leading to Discontinuation of Ceftazidime-Avibactam by System Organ Cla Indication Overall (FAS) | • |
| Table 40 | Adverse Events Leading to Discontinuation of Ceftazidime-Avibactam by System Organ Class by Indication Overall (FAS) | 145 |
| Table 39.1 | Adverse Events Leading to Death Related to Ceftazidime-Avibactam by System Organ Class by Indication Overall (FAS) | 144 |
| Table 39 | Adverse Events Leading to Death by System Organ Class by Indication Overall (FAS) | 143 |
| Table 38.1 | Serious Adverse Events Related to Ceftazidime-Avibactam by System Organ Class by Indication Overall (FAS) | 142 |

Title: Annotated TLF Shells

#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### PLAN

| Listing 8. | Additional Risk Factors | 151 |
|---|---|---|
| Listing 9. | Antibiotic Therapy: Prior Lines of Treatment | 151 |
| Listing 10. | Pattern of use of Ceftazidime-Avibactam | 152 |
| Listing 11. | Concomitant Antibiotic Therapy | 152 |
| Listing 12. | Antibiotic Treatment After Ceftazidime-Avibactam | 152 |
| Listing 13. | Initial Hospitalization | 153 |
| Listing 13.1. | Disease Severity | 153 |
| Listing 14.1. | Healthcare Resource Utilization During Hospitalization (1) | 153 |
| Listing 14.2. | Healthcare Resource Utilization During Hospitalization - Percutaneous procedures (2) | 153 |
| Listing 14.3. | Healthcare Resource Utilization During Hospitalization – Surgical Interventions(3) | 154 |
| Listing 15. | Hospital Readmissions | 154 |
| Listing 16. | Treatment Evaluation for Initial Hospitalization and at 60-Days Post-Discharge | 155 |
| Listing 17. | Microbiology Sample Taken | 155 |
| Listing 18. | Microbiology Bacterial Pathogens Identified in Specimen Sampled | 156 |
| Listing 18.1. | Pathogen Susceptibility | 156 |
| Listing 19. | Mortality and Cumulative Mortality in-Hospital,30-Days and 60-Days Post Discharge | 157 |
| Listing 20. | Adverse Events | 158 |
| | | Page <b>10</b> of <b>159</b> |
| Document: | Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications Title: Annotated TLF Shells | |

Document:

#### ${\tt C3591031\ NON-INTERVENTIONAL\ FINAL\ STUDY\ REPORT-APPENDIX\ 4\ STATISTICAL\ ANALYSIS}$

#### **PLAN**

| Listing 21. | Serious Adverse Events | 158 |
|---|---|---|
| Listing 22. | Adverse Events Leading to Discontinuation of Ceftazidime-Avibactam | 158 |
| Listing 23. | Patient Disposition | 159 |
| Listing 24. | End of Chart Review | 159 |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

#### **PLAN**

#### **Description of Global Rules:**

| Global Rules | Description |
|---|---|
| General information | <ul> <li>All Tables will be performed overall, by region, and then by country.</li> <li>First, overall;</li> <li>Then only for EUFL = "Y"</li> <li>Afterwards, only for LATAMFL = "Y"</li> <li>Finally, for each country.</li> <li>Follow the same logic detailed in Table 2.</li> </ul> |
| Decimal place rules | <ul> <li>Minimum, Maximum – Same decimal places as raw data</li> <li>Mean, Median, Q1, Q3- 1 more decimal places than the raw data</li> <li>SD – 2 more decimal places than the raw data</li> <li>Percentages, 95% CI – 1 decimal place</li> <li>P-values – 3 decimal places</li> </ul> |
| Standard deviation rules | <ul> <li>2 more decimal places than the raw data</li> <li>If n=1, SD displayed as "-"</li> </ul> |
| Percentages | <ul> <li>Based on the number of number of patients with no missing data</li> <li>For zero, only count and no percentage will be displayed.</li> <li>For 100, it shall be displayed as an integer (100)</li> </ul> |
| Lack of observations | <ul> <li>If there is no observation, summary statistics will be displayed as "-"</li> <li>Table completely empty will be prepared with the respective title and a footnote, but with the text "- No Observations -" in the body of the output</li> <li>If a column has N=0, percentages should be represented by "(-)"</li> <li>If a Country has N=0 in ADSL, then it should not be presented in tables</li> </ul> |
| P-values | <ul> <li>3 decimal places</li> <li>P-values rounded to less than 0.001 will be reports as &lt;0.001</li> </ul> |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

# C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Global Rules | Description |
|----------------------|-------------------------------------------------------|
| Confidence intervals | Presented as "xx.x, xx.x" |
| Listings | Sorted by subject number, unless specified otherwise. |


 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

Document:

Table 1.1 Site Characteristics by Country (FAS)

| Characteristic | | tria | Fra | nce | Ger | many | Gre | ece | Ita | ly | Rus | sia | Sp | ain | Uni | ted | Ove | rall |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (N=xx) | | (N=xx) | | (N=xx) | | (N=xx) | | (N=xx) | | (N=xx) | | (N=xx) | | Kingdom<br>(N=xx) | | (N=xx) | |
| Physician<br>specialty, n | | | | | | | | | | | | | | | | | | |
| (%) [1] | | | | | | | | | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx | | xx | | xx | | xx | | xx |
| Infectious<br>disease | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | хx | (xx.x |
| Microbiology | хx | (xx.x) | хx | (xx.x) | ХX | (xx.x) | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x |
| Surgery | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x |
| Internal medicine | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хх | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x |
| Intensive care | xx | (xx.x) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| Anesthesiology | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x |
| Other | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хх | (xx.x |
| Total # of physician | | хх | | xx | | xx | | xx | | xx | | xx | | xx | | xx | | хх |
| Missing, n | | xx | | xx | | xx | | xx | | xx | | xx | | xx | | xx | | xx |
| Hospital care<br>level, n (%)[1] | | | | | | | | | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx | | xx | | xx | | xx | | xx |
| Secondary | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x |
| Tertiary | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | xx | (xx.x |
| Missing, n | | хx | | жx | | хх | | жx | | xx | | хх | | хх | | хx | | хx |
| Hospital type, n<br>(%)[3] | | | | | | | | | | | | | | | | Page | · 14 | of <b>15</b> |

Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


PFIZER 

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Characteristic | Austria | France | Germany | Greece | Italy | Russia | Spain | United | Overall |
|---|---|---|---|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | Kingdom<br>(N=xx) | (N=xx) |
| n | xx | хх | xx | xx | хх | xx | хх | xx | хх |
| Teaching | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-teaching | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total number of beds, n(%) | | | | | | | | | |
| n | xx | хх | xx | xx | жx | xx | жx | xx | хх |
| <500 | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| [500-1000) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| [1000-1500) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| [1500-2000) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| ≥2000 | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| Missing, n | xx | хх | хх | хх | хх | xx | хх | xx | xx |
| Total number of beds | | | | | | | | | |
| n | xx | жx | xx | xx | xx | xx | жx | xx | хх |
| Mean (SD) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Characteristic | Austria | France | Germany | Greece | Italy | Russia | Spain | United | Overall |
|---|---|---|---|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | Kingdom<br>(N=xx) | (N=xx) |
| Q1, Q3 | xx.x, | хх.х, | хх.х, | жж.ж, | хх.х, | хх.х, | хх.х, | жж.ж, | xx.x, |
| | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx.x, | xx.x, | xx.x, | жж.ж, | xx.x, | хх.х, | xx.x, | жж.ж, | xx.x, |
| | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Unknown, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Missing, n | xx | жж | жx | жx | xx | жж | жж | xx | xx |
| CU beds | vv | vv | ** | ** | ** | ** | ** | ** | vv |
| CU beds<br>n | xx | хх | хх | хх | xx | хх | хх | xx | xx |
| CU beds | xx.x | xx.x | xx.x | xx.x | <b>xx.x</b> | xx.x | xx.x | <b>xx.x</b> | xx.x |
| CU beds<br>n<br>Mean (SD) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| CU beds<br>n | xx.x | xx.x | xx.x | xx.x | <b>xx.x</b> | xx.x | xx.x | <b>xx.x</b> | xx.x |
| CCU beds<br>n<br>Mean (SD) | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) | xx.x<br>(xx.xx) |
| Mean (SD) | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x | xx.x<br>(xx.xx)<br>xx.x |
| CCU beds<br>n<br>Mean (SD)<br>Median | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | жж.ж<br>(жж.жж)<br>жж.ж<br>жж.ж, | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | жж.ж<br>(жж.жж)<br>жж.ж<br>жж.ж, | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, |
| CU beds<br>n<br>Mean (SD)<br>Median<br>Q1, Q3 | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x, | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x |
| CU beds<br>n<br>Mean (SD)<br>Median<br>Q1, Q3 | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x | xx.x<br>(xx.xx)<br>xx.x<br>xx.x,<br>xx.x,<br>xx.x |

#### FAS-Full analysis set

Document:


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


TAT

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three, Min- Minimum, Max- Maximum. ICU-Intensive care unit

<sup>[1]</sup> n Number of physicians by specialty. Percentages computed among the total number of physicians (only principal investigator) by Country.

<sup>[2]</sup> n Number of hospitals by level. Percentages computed among the total number of hospitals by Country.

<sup>[3]</sup> n Number of hospitals by type. Percentages computed among the total number of hospitals by Country.

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Characteristic | Argentina (N=xx) | Brazil (N=xx) | Colombia (N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Physician specialty, n (%)[1] | | | | |
| Infectious disease | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Microbiology | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgery | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Internal medicine | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intensive care | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anesthesiology | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total # of physician | xx | xx | xx | жж |
| Missing, n | xx | xx | xx | жж |
| Hospital care level, n (%)[1] | | | | |
| n | xx | xx | xx | xx |
| Secondary | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tertiary | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx |
| <pre>Hospital type, n (%)[3]</pre> | | | | |
| Teaching | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-teaching | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total number of beds, n(%) | | | | |
| n | xx | xx | xx | xx |
| <500 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN** 

| Characteristic | Argentina (N=xx) | Brazil (N=xx) | Colombia (N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| [500-1000) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| [1000-1500) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| [1500-2000) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| ≥2000 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Missing, n | xx | xx | хx | xx |
| Total number of beds | | | | |
| n | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Unknown, n | xx | xx | xx | xx |
| Missing, n | xx | xx | xx | хх |
| Total number of ICU beds | | | | |
| n | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Unknown, n | xx | xx | xx | xx |
| Missing, n | xx | xx | xx | xx |

FAS-Full analysis set


 $\label{thm:lem:path$ Document: Title: Annotated TLF Shells

Version Number: Version Date:

V2.0 11 January 2022

PFIZER 

Document:

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three, Min- Minimum, Max- Maximum. ICU-Intensive care unit [1] n Number of physicians by specialty. Percentages computed among the total number of physicians (only principal investigator) by Country.

- [2] n Number of hospitals by level. Percentages computed among the total number of hospitals by Country.
- [3] n Number of hospitals by type. Percentages computed among the total number of hospitals by Country.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Characteristic | Austria | France | Germany | Greece | Italy | Russia | Spain | United | Overall |
|---|---|---|---|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | Kingdom (N=xx) | (N=xx) |
| Sites with information | | | | | | | | (=: ====, | |
| on percentage of | | | | | | | | | |
| gram-negative | | | | | | | | | |
| isolates that exhibit | | | | | | | | | |
| resistance to the | | | | | | | | | |
| following | | | | | | | | | |
| antibiotics, n(%) | | | | | | | | | |
| n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| 3 <sup>rd</sup> generation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| cephalosporins [1] | | | | | | | | | |
| Carbapenems [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 <sup>rd</sup> generation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| cephalosporins and | | | | | | | | | |
| carbapenems (cross- | | | | | | | | | |
| resistance) [1] | | | | | | | | | |
| Colistin | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | хx | xx | хx | xx | хх | xx | xx |
| If yes, for which | | | | | | | | | |
| year? [2] | | | | | | | | | |
| YYYY | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| YYYY | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| YYYY | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <b>YYYY</b> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Rate of resistance to | | | | | | | | | |
| 3 <sup>rd</sup> generation | | | | | | | | | |
| cephalosporins | | | | | | | | | |
| n(%)[3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Q1, Q3 | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x |
| Min, Max | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, |
| | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Unknown, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Missing, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Characteristic | Austria<br>(N=xx) | France<br>(N=xx) | Germany<br>(N=xx) | Greece<br>(N=xx) | Italy<br>(N=xx) | Russia<br>(N=xx) | Spain<br>(N=xx) | United<br>Kingdom<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|---|
| Rate of resistance to | | | | | | | | | |
| carbapenems | | | | | | | | | |
| n(%)[3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, x.x | xx.x, x.x | <b>xx.x</b> , <b>x.x</b> | <b>xx.x</b> , <b>x.x</b> | xx.x,xx.x | <b>xx.x</b> , <b>x.x</b> | xx.x,xx.x | xx.x, x.x | xx.x,xx.x |
| Min, Max | xx.x,<br>xx.x | xx.x,<br>xx.x | xx.x,<br>xx.x | xx.x,<br>xx.x | xx.x,<br>xx.x | xx.x,<br>xx.x | xx.x,<br>xx.x | xx.x,<br>xx.x | xx.x,<br>xx.x |
| Unknown, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Missing, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Rate of cross-<br>resistance to 3rd<br>generation<br>cephalosporins and<br>carbapenems | | | | | | | | | |
| n(%)[3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, x.x | xx.x,xx.x | xx.x, x.x | xx.x,xx.x | xx.x, x.x | xx.x,xx.x | xx.x, x.x | xx.x,xx.x | xx.x, x.x |
| Min, Max | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, |
| | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Unknown, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Missing, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Rate of resistance to colistin | | | | | | | | | |
| n(%)[3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, |
| | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, | xx.x, |
| | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Unknown, n | xx | xx | xx | xx | xx | xx | xx | xx | хx |
| Missing, n | xx | xx | xx | xx | xx | xx | xx | xx | xx |


 $Path: $$ \Path: $$ \Path: $$ Path: $$ P$ 

Title: Annotated TLF Shells

Document:


PFIZER 

Document:

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

- SD- Standard deviation, Q1- Quartile one, Q3- Quartile three, Min- Minimum, Max- Maximum.
- [1] Percentages computed among the total number of sites by Country.
- [2] The latest available rates.
- [3] Percentages computed among the total number of sites within the sub-category.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Version Number: V2.0 Version Date: 11 January 2022
Table 2 Patients Disposition by Indication Overall (ENR)

| Characteristic | cIAI<br>(N=xx) | cUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL [1]<br>(N=xx) |
|---|---|---|---|---|---|
| Overall (N=xxx) | | | | | |
| Signed informed consent, n(%) | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Applicable as per local | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Applicable as per Local<br>Regulations | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Informed consent provided by, n(%) | | | | | |
| Patient | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Next of kin | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient followed through medical records up to 60 days after hospital discharge, n(%) | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reasons patient not followed<br>through medical records up to 60<br>days after hospital discharge, n(%) | , , | , , | , , | | , , |
| In-hospital death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal from the study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Analysis Population, n (%)

Document:


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| ENR | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|---|
| FAS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS72+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS72- | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| COD | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MOD | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Europe (N=xx) | | | | | |
| Signed informed consent, n (%) | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | AA (AA.A) | AA (AA.A) | AA (AA.A) | AA (AA.A) | AA (AA.A) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Applicable as per Local | | | | | |
| Regulations | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Informed consent provided by, n(%) | | | | | |
| Patient | | | | | |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Next of kin | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient followed through medical records up to 60 days after | | | | | |
| hospital discharge, n(%) | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reasons patient not followed | | | | | |
| through medical records up to 60 | | | | | |
| days after hospital discharge, n(%) | | | | | |
| In-hospital death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal from the study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| Analysis Population datasets, n (%) | | | | | |
|---|---|---|---|---|---|
| ENR | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS72+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS72- | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| COD | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MOD | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Latin America (N=xx) | | | | | |
| Signed informed consent, n (%) | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Applicable as per Local | | | | | |
| Regulations | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre>Informed consent provided by, n(%)</pre> | | | | | |
| Patient | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Next of kin | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient followed through medical | | | | | |
| records up to 60 days after | | | | | |
| hospital discharge, n(%) Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | (, | (, | (, | (, | (, |
| Reasons patient not followed<br>through medical records up to 60<br>days after hospital discharge, n(%) | | | | | |
| In-hospital death [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal from the study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


### Zavicefta

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

### **PLAN**

Document:

| Analysis Population, n (%) | | | | | |
|---|---|---|---|---|---|
| ENR | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS72+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FAS72- | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| COD | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MOD | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> There is xx patient with indication missing.

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

The enrolled set (ENR) has all patients who complied with local requirements of informed consent (provided signed informed consent or informed consent was not applicable per local regulations).

The full analysis set (FAS) has all eligible patients.

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours

FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.

The clinical outcomes analysis set (COD) has all patients exposed to ceftazidime-avibactam  $\geq$  72 hours and  $\geq$  1 non-missing clinical outcome.

The microbiological outcomes analysis set (MOD) has all exposed to ceftazidime-avibactam  $\geq$  72 hours and  $\geq$  1 non-missing microbiological outcome.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


V2.0 11 January 2022

Table 3 Patients by Indication Overall (FAS72+ and FAS72-)

| Characteristic | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Exposure to ceftazidime-avibactam, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| Duration of exposure ≥ 72 hours | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Duration of exposure < 72 hours | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Missing, n | xx | xx | xx | хx | xx |

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.

Table 4.1 Demographic and Baseline Characteristics by Indication Overall (FAS72+)

| Characteristic | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Exposure to ceftazidime-avibactam, n | | | | | |
| (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| Missing, n | хх | xx | xx | xx | xx |
| Age (years) | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | жx | xx | xx | xx | хх |
| Age group, n(%) | | | | | |
| n | жx | xx | хх | xx | xx |
| <40 | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| 40-49 | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| 50-59 | xx (xx) | xx (xx) | xx (xx) | xx(xx) | xx(xx) |
| 60-69 | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| 70-79 | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| 80-89 | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| >=90 | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx(xx) |
| Missing, n | xx | xx | xx | xx | хх |
| Gender, n(%) | | | | | |
| n | xx | xx | xx | xx | xx |
| Male | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Female | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN** 

| Characteristic | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Missing, n | xx | xx | xx | xx | xx |
| Height, cm | | | | | |
| n | хx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | хx |
| Weight, kg | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | хx | хх |
| BMI (kg/m²) | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | XX.X | xx.x |
| Q1, Q3<br>Min, Max | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx.x, xx.x<br>xx | xx.x, xx.x<br>xx | xx.x, xx.x<br>xx | xx.x, xx.x<br>xx | xx.x, xx.x<br>xx |
| Employment status | | | | | |
| n | xx | xx | xx | xx | хx |
| Full Time | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Part Time | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Unemployed | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Retired | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (x |


 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

Document:


11 January 2022

V2.0

## Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Characteristic | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|----------------|---------|---------|---------|---------|---------|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Not Available | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Missing, n | xx | xx | xx | xx | xx |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three, Min- minimum, Max- Maximum.

Table 4.2 Baseline Demographic Characteristics of Patients Exposed to Ceftazidime-Avibactam for <72 hours by Indication Overall (FAS72-)

FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.

Programming Note: Besides Overall, Europe, and LATAM; repeat for each Country. Each section will start in a new page. Possible countries:


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Version Number:

V2.0

Version Date:

11 January 2022

Table 5 Prior Hospitalizations, Healthcare Resource Utilization and Antibiotic Exposure by Indication Overall (FAS72+)

| Characteristic | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any prior hospitalizations within 90 days prior to | | | | | |
| date of current hospitalization, n (%) PRIORHP | | | | | |
| count unique (SUBNUM) | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Hospital LOS for prior hospitalization (days)[1] HOSPDUR | | | | | |
| n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Any healthcare procedure within the 30 days prior to index date, n (%) [3] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing/Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Type of procedure, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| Mechanical ventilation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dialysis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tracheostomy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgical intervention | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Percutaneous procedure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| omer | (, | | (, | (, | (, |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Characteristic | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Antibiotic exposure within 90 days prior to index | | | | | |
| hospitalization, n (%) | | | | | |
| Antibiotic | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing/unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic Class and name [4] | | | | | |
| n | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 3 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Duration of antibiotic treatment (days) | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Reason for antibiotic treatment, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| Therapeutic | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Prophylactic | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | _ | age <b>32</b> of <b>159</b> |

Document:

 $Path: \underline{\Quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$ 

Title: Annotated TLF Shells

### Zavicefta

Document:

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

### **PLAN**

| Characteristic | CIAI<br>(N=xx) | cUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|
| Missing, n | xx | xx | xx | xx | xx |

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

- SD- Standard deviation, Q1- Quartile one, Q3- Quartile three, Min- minimum, Max- Maximum, LOS- Length of Stay.
- [1] Hospital LOS: (Date of hospital discharge Date of hospital admission)
- [2] n for LOS for prior hospitalization, is the number of patients with a prior hospitalization.
- [3] A patient may have had more than one procedure during this period.
- [4] Some patients may be administered multiple antibiotics; the Antibiotic totals may exceed the number of patients. Likewise, the sum of percentages may exceed 100%.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 6 Additional Risk Factors by Indication Overall (FAS72+)

| Risk Factors | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | |
| Travel to foreign country within the last 3 | | | | | |
| months, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Country [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | хх | xx | xx | xx |
| Travel duration [3] | | | | | |
| n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | хх | жx | xx | xx | хx |
| Subject hospitalized during travel, n (%)[2] | xx | хx | хx | xx | хx |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | хх | xx | xx | хx |
| Pregnancy, n (%)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Applicable | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Number of weeks of gestation since last menstrua | 11 | | | | |
| period | | | | | |
| n (%)[4] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |


Document:

 $Path: $$ \Parm = \Parm$ 

Title: Annotated TLF Shells


V2.0


11 January 2022

Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Risk Factors | CIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | хх | xx | xx |
| Does the patient drink alcohol, n (%)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Alcohol use > 14 drinks/week | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Number of drinks per week | | | | | |
| n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Tobacco use, n (%) [1] | | | | | |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Current Smoker | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Previous Smoker | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Never Smoked | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cigarettes per day for current smokers | | | | | |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | хx | хх | xx | хx |


Document:

 $Path: \underline{\Quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$ 

Title: Annotated TLF Shells

Version Number: Version Date: V2.0

11 January 2022

## Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Risk Factors | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | |
| Cigarettes per day for previous smokers | | | | | |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Number of years smoking | | | | | |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

- SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum
- [1] Percentages computed among the total number of patients by Country.
- [2] Percentages computed among the total number of patients within the category.
- [3] Duration of travel = [End date of travel Start date of travel]

Document:

[4] Percentages computed among the total number of pregnant patients.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications
Title: Annotated TLF Shells


Table 7 Comorbidities by Indication Overall (FAS72+)

| Comorbidities | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| ny comorbidities, n (%) [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| o comorbidities, n (%) [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of comorbidities by patient, | | | | | |
| n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| Min, Max | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| Missing, n | xx | xx | xx | xx | xx |
| Any Deyo-Charlson comorbidity, n (%) | | | | | |
| n [1] | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| Missing, n | xx | xx | xx | xx | xx |
| Deyo-Charlson comorbidity score [3], n (%) | | | | | |
| 0 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| 1 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| 2 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| 3 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| >=4 | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| Deyo-Charlson comorbidity score | | | | | |
| n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Deyo-Charlson comorbidities | | | | | |
| Myocardial Infarction, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | Page <b>37</b> of <b>15</b> |
| Document: Path: \\quintiles.net\Enterprise\S | Sites\USCBG\ Dents\ Pio | Stat\ Dfizer\ Zavicofta\ C | Occumentation\Specifics | ations | |
| Title: Annotated TLF Shells | <u> </u> | otat (i lizei (zaviceita) | ocumentation (Specifica | <u> </u> | |


11 January 2022

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Comorbidities | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Congestive heart failure, n (%) [2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Peripheral vascular disease, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Chronic obstructive pulmonary Disease, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Rheumatologic disease, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) |
| Peptic ulcer disease, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderate or severe renal disease, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Skin ulcers/cellulitis, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AIDS, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cerebrovascular disease (except<br>nemiplegia), n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | • • • | • • • | , , | • • • | |
| | | | | | Page <b>38</b> of <b>15</b> 9 |

Document:

 $Path: \underline{\Quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$ 

Title: Annotated TLF Shells

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| V | /3- | | | | |
|---|---|---|---|---|---|
| 7 | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Hemiplegia, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Paraplegia, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mild liver disease, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderate to severe liver disease, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dementia, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Use of warfarin, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Depression, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hypertension, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Diabetes mild to moderate, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | vv /v·· ··\ |
| | • • | • | • | | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Diabetes + complications, n (%)[2] | | | | | |
| | | | | | Page <b>39</b> of <b>15</b> |

Document:

 $\label{thm:path:local} Path: $$ \underline{\CBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$$ 

Title: Annotated TLF Shells


Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Comorbidities | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Malignancy (solid tumor, non-metastic, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Metastatic solid tumor, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hematological malignancy/leukemia or<br>lymphoma, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Bone marrow transplant, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other transplant (solid organ), n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) |
| Any Non-Deyo-Charlson comorbidity , n (%) | | | | | |
| Yes. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No , | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reduced consciousness, n (%)[2] | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 165 | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Document:

 $Path: \underline{\Quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$ 

Title: Annotated TLF Shells


11 January 2022

V2.0

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Comorbidities | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| n | xx | xx | xx | xx | xx |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) |
| 9 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) |
| 10 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) |
| 11 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) |
| 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 13 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 14 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not done | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other, n (%)[2] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | хх | xx | xx | xx |
| Indwelling devices at the time of the infection diagnosis, n $(%)$ | | | | | |
| Any Indwelling device n | хх | хх | xx | xx | xx |
| None [2] | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intravenous peripheric catheter [2] | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intravenous central catheter [2] | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Urinary catheter[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Arterial catheter [2] | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Arteriovenous cannula [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tracheal intubation [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tracheal cannula [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any drain [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam  $\geq$  72 hours.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


### Zavicefta

## C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

- SD- Standard deviation, Q1- Quartile one, Q3- Quartile three, Min- minimum, Max- Maximum
- [1] Percentages computed among the total number of patients by Country.
- [2] Percentages computed among the total number of patients within the category.
- [3] Deyo-Charlson comorbidity score is a derived variable. For the comorbidities to be included and the corresponding weights please refer to the SAP.


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Table 8.1 Source of Infection by Indication Overall (FAS72+)

| Characteristic | cIAI | cuti | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Source of infection, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| HCAI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| HAI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CAI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

HCAI-Healthcare-Associated Infection, HAI-Hospital-Acquired Infection, CAI-Community-Acquired Infection

Note: HCAI and HAI are not mutually exclusive, in principle HCAI include the HAI

Table 8.2 Source of Infection by Indication Overall (FAS72-)

| Characteristic | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Source of infection, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| HCAI | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| HAI | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| CAI | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Missing, n | xx | xx | xx | xx | xx |

FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

HCAI-Healthcare-Associated Infection, HAI-Hospital-Acquired Infection, CAI-Community-Acquired Infection Note: HCAI and HAI are not mutually exclusive, in principle HCAI include the HAI.


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 8.3 Indication for Ceftazidime-Avibactam Overall (FAS72+ and FAS72-)

| Indication for ceftazidime-<br>avibactam | FAS+ (N=XX) | FAS- (N=XX) | Total |
|---|---|---|---|
| Complicated Urinary Tract<br>Infection (cUTI), n (%)[1] | xx (xx.x) | <b>жж</b> (жж.ж) | жж (жж.ж) |
| Complicated Intra-Abdominal Infection (cIAI),n (%)[1] | xx (xx.x) | xx (xx.x) | хх (хх.х) |
| Hospital-Acquired Pneumonia/Ventilator- Associated Pneumonia (HAP/VAP),n (%)[1] | xx (xx.x) | жж (жж.ж) | жж (жж.ж) |
| Other, n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Was the patient diagnosed<br>with COVID-19?<br>Yes<br>No | xx (xx.x)<br>xx (xx.x) | жж (жж.ж)<br>жж (жж.ж) | жж (жж.ж)<br>жж (жж.ж) |
| Not applicable | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| If yes, indication for ceftazidime-avibactam Complicated Urinary Tract Infection (cUTI), n (%)[2] Complicated Intra-Abdominal Infection (cIAI),n (%)[2] Hospital-Acquired Pneumonia/Ventilator- | xx (xx.x)<br>xx (xx.x) | жж (жж.ж)<br>жж (жж.ж) | жж (жж.ж)<br>жж (жж.ж) |
| Associated Pneumonia (HAP/VAP), n (%)[2] | xx (xx.x) | жж (жж.ж) | xx (xx.x) |
| Other, n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

### Zavicefta

Document:

## C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| If No, indication : | | | | | | | |
|---|---|---|---|---|---|---|---|
| Complicated Urinary Infection (cUTI), | y Tract | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Complicated Intra-<br>Infection (cIAI),n | | хх | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Hospital-Acquired Pneumonia/Ventila | | | | | | | |
| Associated<br>(HAP/VAP), n (%)[ | Pneumonia | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Other, n (%)[1] | | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.

cIAI-Complicated Intra-Abdominal Infection; cUTI-Complicated Urinary Tract Infection; HAP-Hospital-Acquired Pneumonia; VAP-Ventilator-Associated Pneumonia.

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

- [1] Percentages computed among the total number of patients by Country.
- [2] Percentages computed among the total number of patients within the category.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Table 9.1 Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) by Bacteria Overall (FAS72+)

| Overall/Region/Country | Escherichia<br>coli<br>(N=xx) | Klebsiella<br>spp.<br>(N=xx) | Enterobacter spp. (N=xx) | Pseudomonas<br>spp.<br>(N=xx) | Other<br>pathogen<br>(N=xx) | No pathogen identified (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|---|
| Indication for ceftazidime-avibactam | | | | | | | |
| Complicated Urinary Tract<br>Infection (cUTI), n<br>(%)[1] INDIC =2 | хх (хх.х) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) | хх (хх.х) | xx (xx.x) |
| Primary diagnosis of UTI (including pyelonephritis) that occurs associated with, n (%) [2] | жж (жж.ж) | хх (хх.х) | xx (xx.x) | жж (жж.ж) | хх (хх.х) | хх (хх.х) | жж (жж.ж) |
| Calculi/Stone | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indwelling catheter or other drainage device | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) | xx (xx.x) |
| Obstruction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Immunosuppression | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Renal failure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Renal transplantation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Functional or anatomical abnormalities of the urinary tract | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) | хх (хх.х) | xx (xx.x) |
| Partial obstructive<br>uropathy (Acquired<br>or congenital) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Elevated postvoidal residual volume (>100 mL residual) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Established diagnosis of neurogenic bladder | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Instrumentation of the urinary tract | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Overall/Region/Country | Escherichia<br>coli<br>(N=xx) | Klebsiella<br>spp.<br>(N=xx) | Enterobacter<br>spp.<br>(N=xx) | Pseudomonas<br>spp.<br>(N=xx) | Other<br>pathogen<br>(N=xx) | No pathogen identified (N=xx) | TOTAL<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Secondary diagnosis of<br>UTI (including<br>pyelonephritis), n (%)[1]<br>Secondary diagnosis of<br>UTI (including<br>pyelonephritis) that<br>occurs associated with, n<br>(%)[2] | хх (хх.х) | жж (жж.ж) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) | жж (жж.ж) |
| Calculi/Stone | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indwelling catheter or other drainage device | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Obstruction | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Immunosuppression | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Renal failure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Renal transplantation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Functional or anatomical abnormalities of the urinary tract | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Partial obstructive uropathy (Acquired or congenital) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Elevated postvoidal residual volume (>100 mL residual) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) | хх (хх.х) |
| Established diagnosis of neurogenic bladder | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Instrumentation of the urinary tract | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Symptoms of UTI, n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fever | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

### Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN**

| Overall/Region/Country | Escherichia<br>coli<br>(N=xx) | Klebsiella<br>spp.<br>(N=xx) | Enterobacter spp. (N=xx) | Pseudomonas<br>spp.<br>(N=xx) | Other<br>pathogen<br>(N=xx) | No pathogen identified (N=xx) | TOTAL<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Flank pain or suprapubic pain or costovertebral angle (CVA) tenderness on examination | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) |
| Dysuria, urgency,<br>frequency, incontinence<br>or nausea/vomiting with<br>no other recognized<br>cause | хж (хж.ж) | жж (жж.ж) | xx (xx.x) | хж (хх.х) | хх (хх.х) | xx (xx.x) | хх (хх.х) |
| Pyuria | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Symptoms of UTI: Positive dipstick for leukocyte esterase and/or nitrite, n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | жж (жж.ж) | xx (xx.x) | жж (жж.ж) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Symptoms of UTI: Did the patient have a secondary bacteremia, n (%)[2] | | | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours. UTI-Urinary tract infection


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications Title: Annotated TLF Shells


SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

<sup>[1]</sup> Percentages computed among the total number of patients by Country. [2] Percentages computed among the total number of patients within the category.

Patients may have more than one pathogen identified.

Document:

Table 9.2 Diagnoses and Symptoms Associated with UTI (Including Pyelonephritis) for Patients with Ceftazidime-Avibactam Exposure <72 Hours (FAS72-)

| Overall/Region/Country | TOTAL |
|---|---|
| | (N=xx) |
| Indication for ceftazidime-avibactam | |
| Complicated Urinary Tract Infection (cUTI), n (%)[1] | xx (xx.x) |
| Primary diagnosis of UTI (including pyelonephritis) that occurs associated with, n (%) [2] | xx (xx.x) |
| Calculi/Stone | xx (xx.x) |
| Indwelling catheter or other drainage | xx (xx.x) |
| device | |
| Obstruction | xx (xx.x) |
| Immunosuppression | xx (xx.x) |
| Renal failure | xx (xx.x) |
| Renal transplantation | xx (xx.x) |
| Pregnancy | xx (xx.x) |
| Functional or anatomical | xx (xx.x) |
| abnormalities of the urinary tract | |
| Partial obstructive uropathy (Acquired | xx (xx.x) |
| or congenital) | , , |
| Elevated postvoidal residual volume (>100 mL residual) | xx (xx.x) |
| Established diagnosis of neurogenic bladder | xx (xx.x) |
| Instrumentation of the urinary tract | xx (xx.x) |
| Other | xx (xx.x) |
| Secondary diagnosis of UTI (including pyelonephritis), n (%)[1] | xx (xx.x) |
| Secondary diagnosis of UTI (including pyelonephritis) that occurs associated with, n | |
| Calculi/Stone | xx (xx.x) |
| Indwelling catheter or other drainage device | xx (xx.x) |
| Obstruction | xx (xx.x) |
| Immunosuppression | xx (xx.x) |
| Renal failure | xx (xx.x) |
| | Page <b>49</b> of : |

Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


### Zavicefta

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

### **PLAN**

| Overall/Region/Country | TOTAL |
|---|---|
| | (N=xx) |
| Renal transplantation | xx (xx.x) |
| Pregnancy | xx (xx.x) |
| Functional or anatomical abnormalities of the urinary tract | xx (xx.x) |
| Partial obstructive uropathy (Acquired or congenital) | xx (xx.x) |
| Elevated postvoidal residual volume (>100 mL residual) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) |
| Established diagnosis of neurogenic bladder | xx (xx.x) |
| Instrumentation of the urinary tract | xx (xx.x) |
| Other | xx (xx.x) |
| Symptoms of UTI, n (%)[2] | xx (xx.x) |
| Fever | xx (xx.x) |
| Flank pain or suprapubic pain or costovertebral angle (CVA) tenderness on examination | xx (xx.x) |
| Dysuria, urgency, frequency, incontinence or nausea/vomiting with no other recognized cause | xx (xx.x) |
| Pyuria | xx (xx.x) |

UTI-Urinary tract infection

Document:


 $\label{thm:linear} Path: $$ \underline{\cline{Conditions}} \ Path: $\underline{\cline{Conditions}} \ Path: $\underline{\cl$ 

Title: Annotated TLF Shells


SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

<sup>[1]</sup> Percentages computed among the total number of patients by Country.

<sup>[2]</sup> Percentages computed among the total number of patients within the category.

Table 10.1 Diagnoses and Symptoms Associated with IAI by Bacteria Overall (FAS72+)

| Overall/Region/Country | Escherichia<br>coli<br>(N=xx) | Klebsiella<br>spp.<br>(N=xx) | Enterobacter spp. (N=xx) | Pseudomonas<br>spp.<br>(N=xx) | Other<br>pathogen<br>(N=xx) | No pathogen identified (N=xx) | TOTAL<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Indication for ceftazidime-avibactam | | | | | | | |
| Complicated Intra-<br>Abdominal Infection<br>(cIAI),n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary diagnosis of<br>IAI, n (%)[2] | xx (xx.x) | хх (хх.х) | xx (xx.x) | хх (хх.х) | хх (хх.х) | хх (хх.х) | xx (xx.x) |
| Peritonitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intraperitoneal abscess | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Liver abscess | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pancreatic abscess | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Appendicitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Diverticulitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gastric or duodenal ulcers | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cholecystitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cholangitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Traumatic population | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Secondary diagnosis of IAI, n (%)[2] | | | | | | | |
| Peritonitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intraperitoneal abscess | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Liver abscess | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pancreatic abscess | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Overall/Region/Country | Escherichia<br>coli | Klebsiella<br>spp. | Enterobacter spp. | Pseudomonas<br>spp. | Other pathogen | No pathogen identified | TOTAL (N=xx) |
|---|---|---|---|---|---|---|---|
| Appendicitis | (N=xx)<br>xx (xx.x) | (N=xx)<br>xx (xx.x) | (N=xx)<br>xx (xx.x) | (N=xx)<br>xx (xx.x) | (N=xx)<br>xx (xx.x) | (N=xx)<br>xx (xx.x) | xx (xx.x) |
| Diverticulitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gastric or duodenal ulcers | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cholecystitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cholangitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Traumatic population | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Symptoms of IAI, n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fever | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hypothermia | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abdominal pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tenderness on palpation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Guarding and rebound tenderness | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abdominal fullness or/ distension | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Nausea or vomiting | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ileus | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Diarrhea | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tachycardia | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hypotension | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Shock | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Symptoms of IAI: Did the patient have a secondary bacteremia? | | | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | | Page <b>52</b> of <b>15</b> |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


PFIZER 

## Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Overall/Region/Country | Escherichia | Klebsiella | Enterobacter | Pseudomonas | Other | No pathogen | TOTAL |
|---|---|---|---|---|---|---|---|
| | coli | spp. | spp. | spp. | pathogen | identified | (N=xx) |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

IAI-Intra-abdominal infection

Document:

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

- [1] Percentages computed among the total number of patients by Country.
- [2] Percentages computed among the total number of patients within the category.

Patients may have more than one pathogen identified.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 10.2 Diagnoses and Symptoms Associated with IAI for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-)

| Overall/Region/Country | TOTAL | |
|---|---|---|
| Indication for ceftazidime-avibactam | (N=xx) | |
| Complicated Intra-Abdominal Infection (cIAI),n (%)[1] | xx (xx.x) | |
| Primary diagnosis of IAI, n (%)[2] | xx (xx.x) | |
| Peritonitis | xx (xx.x) | |
| Intraperitoneal abscess | xx (xx.x) | |
| Liver abscess | xx (xx.x) | |
| Pancreatic abscess | xx (xx.x) | |
| Appendicitis | xx (xx.x) | |
| Diverticulitis | xx (xx.x) | |
| Gastric or duodenal ulcers | xx (xx.x) | |
| Cholecystitis | xx (xx.x) | |
| Cholangitis | xx (xx.x) | |
| Traumatic population | xx (xx.x) | |
| Other | xx (xx.x) | |
| Secondary diagnosis of IAI, n (%)[2] | | |
| Peritonitis | xx (xx.x) | |
| Intraperitoneal abscess | xx (xx.x) | |
| Liver abscess | xx (xx.x) | |
| Pancreatic abscess | xx (xx.x) | |
| Appendicitis | xx (xx.x) | |
| Diverticulitis | xx (xx.x) | |
| Gastric or duodenal ulcers | xx (xx.x) | |
| Cholecystitis | xx (xx.x) | |
| Cholangitis | xx (xx.x) | |
| | Page <b>5</b> - | 4 of <b>15</b> 9 |
| Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Depts\Dept | | |

Title: Annotated TLF Shells

# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Overall/Region/Country | TOTAL |
|-----------------------------------|-----------|
| | (N=xx) |
| Traumatic population | xx (xx.x) |
| Other | xx (xx.x) |
| Symptoms of IAI, n (%)[2] | xx (xx.x) |
| Fever | xx (xx.x) |
| Hypothermia | xx (xx.x) |
| Abdominal pain | xx (xx.x) |
| Tenderness on palpation | xx (xx.x) |
| Guarding and rebound tenderness | xx (xx.x) |
| Abdominal fullness or/ distension | xx (xx.x) |
| Nausea or vomiting | xx (xx.x) |
| Ileus | xx (xx.x) |
| Diarrhea | xx (xx.x) |
| Tachycardia | xx (xx.x) |
| Hypotension | xx (xx.x) |
| Shock | xx (xx.x) |

FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


Table 11.1 Diagnoses and Symptoms of NP Associated with HAP/VAP by Bacteria Overall (FAS72+)

| Overall/Region/Country | Escherichia<br>coli<br>(N=xx) | Klebsiella<br>spp.<br>(N=xx) | Enterobacter spp. (N=xx) | Pseudomonas<br>spp.<br>(N=xx) | Other<br>pathogen<br>(N=xx) | No pathogen identified (N=xx) | TOTAL[3] (N=xx) |
|---|---|---|---|---|---|---|---|
| Indication for ceftazidime-avibactam | | | | | | | |
| Hospital-Acquired<br>Pneumonia/Ventilator-<br>Associated Pneumonia<br>(HAP/VAP),n (%)[1] | хх (хх.х) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hospital acquired pneumonia, n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) |
| Ventilator-associated pneumonia, n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Symptoms of NP diagnosis, n (%)[2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fever | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| White blood cell | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| For adults 70 years or older, | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| A new onset of cough | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| New onset of purulent sputum | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Auscultatory findings consistent with pneumonia/pulmonary consolidation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) | жж (жж.ж) |
| Dyspnea, tachypnea or hypoxemia | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| A need for mechanical ventilation | хх (хх.х) | xx (xx.x) | хх (хх.х) | хх (хх.х) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

## Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Overall/Region/Country | Escherichia<br>coli<br>(N=xx) | Klebsiella<br>spp.<br>(N=xx) | Enterobacter spp. (N=xx) | Pseudomonas<br>spp.<br>(N=xx) | Other<br>pathogen<br>(N=xx) | No pathogen identified (N=xx) | TOTAL[3]<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Symptoms of NP: Did<br>the patient have a<br>secondary bacteremia?,<br>n (%) [2] | | | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown, n | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

HAP- Hospital Associated Pneumonia; VAP- Ventilator-Associated Pneumonia.


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications
Title: Annotated TLF Shells


V2.0


SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

<sup>[1]</sup> Percentages computed among the total number of patients by Country.

<sup>[2]</sup> Percentages computed among the total number of patients with Hospital-Acquired Pneumonia/Ventilator-Associated

<sup>[3]</sup> The total column are unique patients with the specific characteristic. Patients may have more than one pathogen identified.

Document:

Table 11.2 Diagnoses and Symptoms of NP Associated with HAP/VAP for Patients with Ceftazidime-Avibactam Exposure <72 Hours
Overall (FAS72-)

| | = = |
|---|---|
| | (N=xx) |
| Indication for ceftazidime-avibactam | |
| Hospital-Acquired Pneumonia/Ventilator-Associated Pneumonia (HAP/VAP),n (%)[1] | xx (xx.x) |
| Hospital acquired pneumonia, n (%)[1] | xx (xx.x) |
| Ventilator-associated pneumonia, n (%)[1] | xx (xx.x) |
| Symptoms of NP diagnosis, n (%)[2] | xx (xx.x) |
| Fever | xx (xx.x) |
| White blood cell | xx (xx.x) |
| For adults 70 years or older, | xx (xx.x) |
| A new onset of cough | xx (xx.x) |
| New onset of purulent sputum | xx (xx.x) |
| Auscultatory findings consistent with pneumonia/pulmonary consolidation | xx (xx.x) |
| Dyspnea, tachypnea or hypoxemia | xx (xx.x) |
| A need for mechanical ventilation | xx (xx.x) |
| Symptoms of NP: Did the patient have a secondary bacteremia?, n (%) [2] | |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| Unknown, n | xx (xx.x) |

FAS72-: is a subset of the FAS patients with <72 hours exposure to ceftazidime-avibactam


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells
Table 12.1 Diagnoses and Symptoms Associated with Other Indication by Bacteria Overall (FAS72+)

| | Escherichia<br>coli<br>(N=xx) | Klebsiella Enterobact Pseudomonas<br>spp. er spp. spp.<br>(N=xx) (N=xx) (N=xx) | | Other Gram- negative pathogen (N=xx) | No pathogen identified (N=xx) | TOTAL [3]<br>(N=xx) | |
|---|---|---|---|---|---|---|---|
| Indication for ceftazidime-avibactam: | | | | | | | |
| Other n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SSI [2] INDICOTH | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CLABSI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BSI/Sepsis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Meningitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Endocarditis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Osteomyelitis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Febrile neutropenia | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Initial site of infection (organ), n (%) [1] Appendix [2] | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Bladder | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Kidney | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Large Intestine | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lungs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Liver | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gall Bladder | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pancreas | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Peritoneum | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Small Intestine | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stomach | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Urethra | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | Escherichia<br>coli<br>(N=xx) | Klebsiella<br>spp.<br>(N=xx) | Enterobact<br>er spp.<br>(N=xx) | Pseudomonas<br>spp.<br>(N=xx) | Other Gram- negative pathogen (N=xx) | No pathogen identified (N=xx) | TOTAL [3]<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Did the patient have a secondary bacteremia? [1] | | | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

- [1] Percentages computed among the total number of patients by Country.
- [2] Percentages computed among the total number of patients within the category.
- [3] The total column are unique patients with the specific characteristic.

Patients may have more than one pathogen identified.


 $\label{thm:linear} Path: $$ \underline{\cline{Conditions}} \ Path: $$\underline{\cline{Conditions}} \ Path: $\underline{\cline{Conditions}} \ Path: $\underline{\cline{C$ 

Title: Annotated TLF Shells

Document:


Title: Annotated TLF Shells

Table 12.2 Diagnoses and Symptoms of NP Associated with Other Indication for Patients with Ceftazidime-Avibactam Exposure <72 Hours Overall (FAS72-)

| | TOTAL [3] |
|---|---|
| Indication for ceftazidime-avibactam: | (N=xx) |
| Other n (%)[1] | xx (xx.x) |
| SSI [2] | xx (xx.x) |
| CLABSI | xx (xx.x) |
| BSI/Sepsis | xx (xx.x) |
| Meningitis | xx (xx.x) |
| Endocarditis | xx (xx.x) |
| Osteomyelitis | xx (xx.x) |
| Febrile neutropenia | xx (xx.x) |
| Other | xx (xx.x) |
| Initial site of infection (organ), n (%) [1] | xx (xx.x) |
| Appendix [2] | xx (xx.x) |
| Bladder | xx (xx.x) |
| Kidney | xx (xx.x) |
| Large Intestine | xx (xx.x) |
| Lungs | xx (xx.x) |
| Liver | xx (xx.x) |
| Gall Bladder | xx (xx.x) |
| Pancreas | xx (xx.x) |
| Peritoneum | xx (xx.x) |
| Small Intestine | xx (xx.x) |
| Stomach | xx (xx.x) |
| Urethra | xx (xx.x) |
| Other | xx (xx.x) |
| Did the patient have a secondary bacteremia? [1] | |
| | Page <b>61</b> of <b>1</b> ! |


V2.0

11 January 2022

## Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

**PLAN** 

Document:

| TOTAL [3] (N=xx) |
|------------------|
| (H-XX) |
| xx (xx.x) |
| xx (xx.x) |
| xx (xx.x) |

FAS72-: is a subset of the FAS patients with <72 hours exposure to ceftazidime-avibactam


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


11 January 2022

V2.0

Table 13 Initial Hospitalization by Indication Overall (FAS72+)

| | | CIAI | | cUTI | H.Z | P/VAP | C | Other | 7 | TOTAL |
|---|---|---|---|---|---|---|---|---|---|---|
| | ( | N=xx) | ( | N=xx) | ( | N=xx) | ( | N=xx) | ( | N=xx) |
| Mode of admission, n (%)[1] | | | | | | | | | | |
| Emergency | | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) |
| Scheduled | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Missing, n | | xx | | xx | | xx | | xx | | xx |
| Source of admission, n (%)[1] | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx |
| Outpatient | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Long-term care facility | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Transfer from acute care hospital | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Other | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Missing, n | | xx | | xx | | xx | | xx | | xx |
| Initial ward admitted at hospitalization, n (%)[1] | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx |
| Surgical | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Medical | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Onco-hematology | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Infectious disease | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| ICU | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Other | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Missing, n | | xx | | xx | | хх | | xx | | хx |
| All wards attended during hospitalization, n | | | | | | | | | | |
| (%) [1,2] | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx |
| Surgical | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Medical | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Onco-hematology | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Infectious disease | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| ICU | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Other | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Missing, n | | xx | | xx | | xx | | xx | | хx |
| LOS from hospital admission [3] | | | | | | | | | | |
| LOS ITOM NOSPITAL ACMISSION [3] | | | | | | | | Б | age <b>63</b> | o f |


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


| | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| LOS from start of Ceftazidime-avibactam [4] | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Was the patient admitted to the ICU, n(%)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing/Unknown | xx | xx | xx | xx | xx |
| Cumulative ICU LOS from hospital admission [5] | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | хх | xx | xx |
| Was APACHE II evaluated upon admission to ICU?, | | | | | |
| n(%)[3] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| APACHE II Score | | | | | |
| | | | | P | age <b>64</b> of <b>159</b> |

Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications
Title: Annotated TLF Shells


### Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN**

| | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Was another disease severity score evaluated? | | | | | |
| [1] | | | | | |
| n | xx | xx | xx | xx | xx |
| | | | () | xx (xx.x) | / |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | AA (AA.A) | xx (xx.x) |
| Yes<br>No | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum, LOS- Length of Stay, ICU-Intensive care unit

- [1] Percentages computed among the total number of patients by Country.
- [2] A subject can attend more than one ward during hospitalization.

Document:

- [3] Consecutive Hospital LOS: (Date of hospital discharge Date of hospital admission)
- [4] Hospital LOS from treatment initiation: (Date of hospital discharge Date of ceftazidime-avibactam initiation)
- [5] Consecutive or non-consecutive ICU LOS: (Date of ICU discharge Date of ICU admission)
- [6] ICU LOS from treatment initiation: (Date of ICU discharge Date of ceftazidime-avibactam initiation)


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications Title: Annotated TLF Shells


V2.0 11 January 2022


Table 14 Healthcare Resource Utilization by Indication Overall (FAS72+)

| | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Did the patient use any healthcare resources during the index hospitalization? n (%) [1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | хx |
| Healthcare resource utilized during the index | | | | | |
| hospitalization, n (%) [1] | | | | | |
| Mechanical ventilation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hemodialysis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CT/MRI imaging | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tracheostomy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgical intervention | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Percutaneous procedures | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mechanical ventilation: number of Days (for patients who received ventilation) [2] | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | хх | xx | xx | xx | хх |
| Hemodialysis (including intermittent or continuous renal replacement therapy), n (%) [1] | | | | | |
| n, (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intermittent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Continuous | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hemodialysis: number of days [2] | | | | | |
| n | xx | xx | xx | xx | xx |
| | | | | Pag | ge <b>66</b> of <b>159</b> |
| Oocument: Path: \\quintiles.net\Enterprise\Sites\USCBG\Dep | ts\BioStat\Pfizer\Zavio | cefta\Documentation | \Specifications | | |
| Title: Annotated TLF Shells | | | | | |

Ve

| | cIAI<br>(N=xx) | cUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL<br>(N=xx) |
|---|---|---|---|---|---|
| Mean (SD) xx.x | | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | жж | xx | жж | хx |
| Surgical intervention, n (%)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Number of surgical interventions, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Percutaneous procedure, n (%)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | хх | хх | xx | хх | хх |
| Number of percutaneous procedures, n (%) | | | | | |
| n | xx | xx | xx | xx | xx |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other procedure, n (%)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Number of other procedures, n (%) | | | | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


PFIZER 

| | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| n | xx | xx | xx | xx | xx |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Procedure performed to control infection? , n (%)[ | 3] | | | | |
| Any procedure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgical intervention | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Percutaneous procedure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other procedure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of surgical interventions to control | | | | | |
| infection, n (%) | | | | | |
| n | xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of percutaneous procedures to control infection, n(%) | | | | | |
| n | xx | xx | xx | xx | xx |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Number of other procedures to control infection, n | 1(%) | | | | |
| n | xx | xx | xx | xx | xx |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

- [1] Percentages computed among the total number of patients by Country.
- [2] Number of Days = Stop Date Start Date
- [3] Percentages computed among the total number of patients.

Table 15 Antibiotic Therapy: Prior Lines of Treatment Prior to Ceftazidime-Avibactam by Indication Overall (FAS72+)


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications
Title: Annotated TLF Shells


11 January 2022

V2.0

| Repeat table for each of | cIAI | cIAI cUTI | | Other | TOTAL |
|---|---|---|---|---|---|
| Gram-Negative/ Gram-Positive/ | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Anaerobic/ other (include antifungal, antiviral, other) | | | | | |
| table | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Antibiotic class and name (generic name, n(%) [2] | | | | | |
| n | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 1 | xx (xx. | (xx.xx) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx. | (xx.xx) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 | xx (xx. | (xx.xx) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 3 etc. | xx (xx. | (xx.xx) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 2 | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 3 | xx (xx.x | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 4 | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 5 | xx (xx. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx. | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | • | | | | |
| Total duration (days) of antibiotics used for current | | | | | |
| infection up to the start of Ceftazidime-avibactam [3] | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x | xx.x | xx.x | xx.x | xx.x |
| | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx. | x xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx. | x xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| n | xx | xx | xx | xx | xx |
| | | | | F | Page <b>69</b> of <b>15</b> 9 |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


PFIZER 

| Repeat table for each of | | cIAI<br>(N=xx) | | cUTI | | AP/VAP | Other | | TOTAL | |
|---|---|---|---|---|---|---|---|---|---|---|
| Gram-Negative/ Gram-Positive/ | ( | N=xx) | ( | N=xx) | ( | N=xx) | ( | N=xx) | (1 | N=xx) |
| Anaerobic/ other (include antifungal, antiviral, other) | | | | | | | | | | |
| Reason for initiating per antibiotic, n(%)[2] | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| n | | xx | | хх | | xx | | xx | | xx |
| Clostridium difficile | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Disease progression | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Empiric treatment | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Failure of antimicrobial therapy | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Infection | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Microbiology | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Prophylaxis | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Other | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Missing, n | | xx | | xx | | xx | | xx | | xx |
| Reason for discontinuation per antibiotic, n(%) [2] | | | | | | | | | | |
| n . | | xx | | xx | | xx | | xx | | xx |
| AE | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Perceived clinical failure/disease progression | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Isolation of a resistant pathogen | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Preference for empiric coverage | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Secondary infection requiring regimen change | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Switch to oral therapy | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| De-escalation | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Cure | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Death | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Other | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Missing, n | | xx | | хх | | xx | | xx | | хх |
| Antibiotics that were continued after start of | | | | | | | | | | |
| ceftazidime-avibactam | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx |
| Therapeutic class 1 | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Antibiotic 1 | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Antibiotic 2 | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Antibiotic 3 etc. | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| | | | | | | | | | D <b>7</b> | 0 af 1E0 |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Repeat table for each of<br>Gram-Negative/ Gram-Positive/<br>Anaerobic/ other (include antifungal, antiviral, other) | cIAI<br>(N=xx) | CUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL<br>(N=xx) |
|---|---|---|---|---|---|
| Therapeutic class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 3 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 3 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

AE - Adverse event, SD - Standard deviation, Q1- Quartile one, Q3 - Quartile three. Min - minimum, Max - Maximum

- [1] Percentages computed among the total number of patients by Country.
- [2] Percentages computed among the total number of patients within the category. For the variable, "Reason for initiating per Antibiotic", percentages may exceed 100% due to cases where one individual was treated with more than one antibiotic.
- [3] Duration of Antibiotic = [Stop Date of Antibiotic Start Date of Antibiotic]


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Version Date: 11

11 January 2022

V2.0

Table 16.1 Ceftazidime-Avibactam Usage by Indication Overall (FAS72+)

| | cIAI | cUTI | HAP/VAP (N=xx) | Other | Total |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | | (N=xx) | (N=xx) |
| Use of ceftazidime-avibactam overall, n(%)[2] | | | | | |
| Monotherapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Combination Therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative coverage | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other coverage | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative and Other coverage | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fotal Duration of administration of ceftazidime-avibactam (days), n(%) | | | | | |
| 1 | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.x |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Outcome/Reason for discontinuation of ceftazidime-avibactam, n (%) [1] | | | | | |
| n | xx | xx | xx | xx | xx |
| AE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Perceived clinical failure/disease progression | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Isolation of a resistant pathogen | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preference for empiric coverage | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Secondary infection requiring regimen change | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Switch to oral therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| De-escalation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| riroarity, ii | AA | AA | ** | AA | ** |

 $Path: $$ \Path: \underline{\Documentation\Specifications} $$ Path: \underline{\Documentat$ 

Title: Annotated TLF Shells

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

| PΙ | _AN |
|----|-----|
|----|-----|

| Dose and frequency of ceftazidime-avibactam, | | | | | |
|---|---|---|---|---|---|
| duration of infusion and treatment duration for | | | | | |
| <pre>each dosage n (%) Dose1*Frequency1</pre> | | | | | |
| Duration of Infusion | | | | | |
| 2 hours | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 hours | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment duration (days) | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | хх | хх | xx |
| Total dose of ceftazidime-avibactam | | | | | |
| n | xx | xx | xx | хх | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | xx | xx |
| Daily dose of ceftazidime-avibactam (mg) | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | xx | xx | хх | xx |
| Antibiotics combined with ceftazidime-avibactam, | | | | | |
| by WHO Drug Class and preferred term | | | | | |
| Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | Page | <b>73</b> of <b>159</b> |

Document:

 $\label{thm:likes$ 

Title: Annotated TLF Shells


## C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Antibiotic name | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|---|
| Antibiotic name | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic name | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic name | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for initiation of antibiotics combined with | | | | | |
| ceftazidime-avibactam | | | | | |
| Clostridium difficile | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Empiric treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Failure of antimicrobial treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Infection | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Microbiology | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Prophylaxis | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Please order Antibiotics by: Gram-negative coverage (GRAMNFL = `Y'), Gram-positive | | | | | |
| coverage (GRAMPFL = \text{\text{Y}}), Anaerobe coverage | | | | | |
| (ANAEFL = 'Y') and Other (OTHFL = 'Y') | | | | | |
| Reason for discontinuation of antibiotics combined with ceftazidime-avibactam | | | | | |
| Reason 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc | | | | | |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

- [1] Percentages computed among the total number of patients within the category.
- [2] Percentages computed among the total number of patients by Country.

Antibiotic class and name are sorted by Therapeutic class and antibiotics by alphabetical order.

'Other agents' class are in the order: 1. Polymyxins, 2. Sulfonamides and Trimethoprim, 3. Other antibiotics, 4. Antiviral drugs, 5. Antimycotic drugs, 6. Antiparasitic drugs.

Reason for initiation/discontinuation of antibiotics is sorted by alphabetical order.


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


#### Zavicefta

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

Table 16.2 Ceftazidime-Avibactam Usage <72 Hours by Indication Overall (FAS72-) FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.

Footnote: Antibiotic class and name is sorted by Therapeutic class and antibiotics by alphabetical order.

'Other agents' class are in the order: 1. Polymyxins, 2. Sulfonamides and Trimethoprim, 3. Other antibiotics, 4. Antiviral drugs, 5. Antimycotic drugs, 6. Antiparasitic drugs.

Reason for initiation/discontinuation will be sorted by alphabetical order.


Document: Path:\\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 17.1 Ceftazidime-Avibactam by Indication in Patients Infected by Escherichia coli Overall (FAS72+)

Table 17.2 Ceftazidime-Avibactam by Indication in Patients Infected by Klebsiella spp. Overall (FAS72+)

Table 17.3 Ceftazidime-Avibactam by Indication in Patients Infected by Enterobacter spp. Overall (FAS72+)

Table 17.4 Ceftazidime-Avibactam by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72+)

Table 17.5 Ceftazidime-Avibactam by Indication in Patients Infected by Other Gram-negative Bacteria Overall (FAS72+)

Table 17.6 Ceftazidime-Avibactam Usage >72 Hours by Indication in Patients with no pathogen identified (FAS72+)


Document:

 $Path: $$ \ \underline{\CBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications} $$$ 

Title: Annotated TLF Shells

Version Number: Version Date: V2.0

ate: 11 January 2022

Table 18. Immunocompromised patients by indication (FAS72+)

| Yes | | cIAI (N=xx) | cuti (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | Total (N=xx) |
|---|---|---|---|---|---|---|
| No | Immunocompromised patients overall, n(%) | | | | | |
| Subgroups by Comorbidities AIDS diagnosis, n(%) Yes | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AIDS diagnosis, n(%) Yes | No | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | Subgroups by Comorbidities AIDS diagnosis, n(%) | | | | | |
| Malignancy (solid tumor, non-metastatic), n(%) Yes XX (XX.X) XX | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (x | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | Malignancy (solid tumor, non-metastatic), n(%) | | | | | |
| Chemotherapy received in the last 3 months? n(%) Yes | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No xx (xx.x) < | | | | | | |
| Yes xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) No xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Chemotherapy received in the last 3 months? n(%) xx (xx.x) Yes xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Hematological malignancy/Leukaemia or lymphoma, n(%) Yes xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | Metastatic solid tumor, n(%) | | | | | |
| Chemotherapy received in the last 3 months? n(%) Yes No Hematological malignancy/Leukaemia or lymphoma, n(%) Yes xx (xx.x) | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n(%) Yes xx (xx.x) xx (xx. | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | | | | | | |
| Hematological malignancy/Leukaemia or lymphoma, n(%) Yes xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | Yes | • • | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n(%) Yes | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ( | Hematological malignancy/Leukaemia or lymphoma, $n(%)$ | | | | | |
| No | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


#### Zavicefta

Document:

## C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Chemotherapy received in the last 3 months? | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| n (%) | | | | | | | | | | |
| Yes | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| No | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Bone marrow transplant, n(%) | | | | | | | | | | |
| Yes | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| No | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | ХX | (xx.x) | хx | (xx.x) |
| Other transplant (Solid organ), n(%) | | | | | | | | | | |
| Yes | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| No | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Overall outcome of ceftazidime-avibactam for | | | | | | | | | | |
| immunocompromised patients | | | | | | | | | | |
| n (%) | | xx | | xx | | xx | | xx | | xx |
| Treatment Success | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Treatment Failure | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Indeterminate | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Overall outcome of ceftazidime-avibactam for Non- | | | | | | | | | | |
| immunocompromised patients | | | | | | | | | | |
| n (%) | | xx | | xx | | xx | | xx | | xx |
| Treatment Success | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Treatment Failure | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Indeterminate | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 19. Patients with primary/secondary Bacteriemia by indication (FAS72+)

| | cIAI | (N=xx) | cUTI | (N=xx) | HAP/VA | P (N=xx) | Other | (N=xx) | Tota: | l (N=xx |
|---|---|---|---|---|---|---|---|---|---|---|
| Patients with bacteriemia overall, n(%) | | | | | | | | | | |
| Primary | | | | | | | | | xx | (xx.x) |
| Secondary | vv | (xx.x) | vv | (xx.x) | ** | (xx.x) | vv | (xx.x) | | (xx.x) |
| No or Unknown | | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) |
| NO OI OIRIIONII | AA | (AA.A) | AA | (AA.A) | AA | (AA.A) | AA | (AA.A) | AA | (AA.A) |
| Patients with primary bacteriemia overall, n(%) | | | | | | | | | | |
| Yes | | | | | | | | | xx | (xx.x) |
| No | | | | | | | | | xx | (xx.x) |
| Patients with secondary bacteriemia overall, n(%) | | | | | | | | | | |
| Yes | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| No | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Unknown | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | хx | (xx.x) |
| Overall outcome of ceftazidime-avibactam for patients | | | | | | | | | | |
| with primary bacteriemia | | | | | | | | | | |
| n(%) | | xx | | xx | | xx | | xx | | xx |
| Treatment Success | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Treatment Failure | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Indeterminate | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Overall outcome of ceftazidime-avibactam for patients without primary bacteriemia | | | | | | | | | | |
| n (%) | | xx | | xx | | xx | | xx | | xx |
| Treatment Success | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Freatment Failure | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Indeterminate | хx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Overall outcome of ceftazidime-avibactam for patients | | | | | | | | | | |
| with secondary bacteriemia | | | | | | | | | | |
| n (%) | | xx | | хx | | хх | | хх | | xx |
| Treatment Success | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Treatment Failure | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Indeterminate | | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


#### Zavicefta

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### **PLAN**

Document:

| Overall outcome of ceftazidime-avibactam for | XX | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| patients without secondary bacteriemia | | | | | | | | | | |
| n (%) | | xx | | xx | | xx | | xx | | xx |
| Treatment Success | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Treatment Failure | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Indeterminate | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Overall outcome of ceftazidime-avibactam for | | | | | | | | | | |
| patients without primary or secondary bacteriemia | | | | | | | | | | |
| n(%) | | xx | | xx | | xx | | xx | | xx |
| Treatment Success | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Treatment Failure | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Indeterminate | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

V2.0 Version Number: Version Date: 11 January 2022

PFIZER 

Table 20. Patients with lower dose of Ceftazidime-Avibactam by indication (FAS72+)

| | cIAI (N=xx) | cuti (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | Total (N=xx) |
|---|---|---|---|---|---|
| Patients with lower dose of | | | | | |
| Ceftazidime-Avibactam overall, n(%) | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Overall outcome of ceftazidime- | | | | | |
| vibactam for patients with lower | | | | | |
| lose of Ceftazidime-Avibactam | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| Treatment Success | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment Failure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indeterminate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| verall outcome of ceftazidime- | | | | | |
| vibactam for patients without lower | | | | | |
| ose of Ceftazidime-Avibactam | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| Treatment Success | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment Failure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indeterminate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Population with lower dose of Cef | tazidime-Avibactam | will include those | subjects with average | ≤4 q. | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

Table 21. Clinical Outcome for patients with COVID-19 diagnosis (FAS72+)

| Overall outcome of ceftazidime-<br>avibactam for patients with COVID-19<br>diagnosis | cIAI N=xx) | cuti (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | Total (N=xx) |
|---|---|---|---|---|---|
| n(%) | xx | xx | xx | xx | xx |
| Treatment Success | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment Failure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indeterminate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Overall outcome of ceftazidime- | | | | | |
| avibactam for patients without COVID- | | | | | |
| 19 diagnosis | | | | | |
| n(%) | xx | xx | xx | xx | xx |
| Treatment Success | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment Failure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indeterminate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


 $\label{thm:linear} Path: $$ \underline{\cline{Conditions}} \ Path: $$\underline{\cline{Conditions}} \ Path: $\underline{\cline{Conditions}} \ Path: $\underline{\cline{C$ 

Title: Annotated TLF Shells

Document:

Table 22.1 Microbiological Evaluation Before Initial Antibiotic Therapy by Indication Overall (FAS72+)

| | cIAI | (N=xx) | cUTI | (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (1 | N=x |
|---|---|---|---|---|---|---|---|---|
| Patient Level | | | | | | | | |
| Samples taken, n(%) | | | | | | | | |
| N | | жж | | xx | xx | xx | xx | ĸ |
| Yes | xx | (xx.x) | хx | (xx.x) | xx (xx.x) | xx (xx.x) | хх (х | ж.х |
| No | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (x | ж.х |
| Missing, n | | xx | | xx | xx | xx | xx | ĸ |
| Number of bacterial pathogens, n(%) | | | | | | | | |
| N | | xx | | xx | xx | xx | xx | x |
| 0 | xx | (xx.x) | ж | (xx.x) | xx (xx.x) | xx (xx.x) | хх (х | ж.х |
| 1 | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (x | ж.х |
| 2 | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (x | ж.х |
| >2 | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (x: | ж.х |
| Not Known | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (x: | ж.х |
| Same pathogen in >1 sample | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | хх (х | ж.х |
| Was a fungal pathogen identified?, n(%) | | | | | | | | |
| N | | xx | | xx | xx | xx | xx | |
| Yes | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх | к. ж) |
| No | xx | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx | |
| Missing, n | | xx | | xx | xx | xx | xx | |
| Type of specimen, n(%) | | | | | | | | |
| N | | xx | | xx | xx | xx | xx | |
| Blood | | (xx.x) | | (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх | |
| Catheter tip | | (xx.x) | | (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх | - |
| | | (xx.x) | | (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх | - |
| Urine | | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx | к.х) |
| Bronchoalveolar lavage | | - | | | and the second s | | | |
| | | (xx.x) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх | K.X) |

 $\label{thm:path:local} Path: $$ \underline{\CBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$$ 

Title: Annotated TLF Shells

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| Swab | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Surgical/biopsy specimen | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pathogens identified | | | | | | |
| <pre>Gram-negative, Escherichia Coli, n(%)</pre> | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Klebsiella pneumoniae, | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n(%) | | | | | | |
| Gram-negative, Klebsiella spp. | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre>Gram-negative, Proteus mirabilis, n(%)</pre> | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre>Gram-negative, Proteus spp., n(%)</pre> | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Acinetobacter baumanii, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Acinetobacter spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Enterobacter cloacae, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Enterobacter spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Citrobacter spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Serratia spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Morganella morganii, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Salmonella spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Shigella spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Pseudomonas aeruginosa, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Pseudomonas spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Haemophilus influenzae, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Haemophilus spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Other, n(%) | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram positive, Staphylococcus aureus, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram positive, Enterococcus spp., n(%) | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mycobacterium abscessus | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, Bacteroides spp. | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, Peptostreptococcus spp. | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, Clostridium spp. | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, Prevotella spp. | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, other | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, other specify | XX | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pathogen Level | | | | | | |
| Gram-negative, Escherichia Coli, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | Page <b>84</b> of <b>1</b> 5 |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | | | | | |
| | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Klebsiella pneumoniae, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n<br>- | | xx | xx | xx | xx | XX . |
| A | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | Page <b>85</b> of <b>159</b> |

rage 85 or 15

Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, <i>Klebsiella</i> spp. Beta-lactamase identified: | хх | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Proteus Mirabilis, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | Page <b>86</b> of |

Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | CIAI | (N=xx) | cUTI | (N=xx) | HAP/VA | P (N=xx) | Othe | r (N=xx) | TOTA | L (N=x |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| 2 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| 3 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| >3 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Unknown/not tested | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | хx | (xx.x) |
| Ambler's class, n(%) | | | | | | | | | | |
| N | | xx | | xx | | xx | | xx | | xx |
| A | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| В | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| С | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| D | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Ambler's type, n(%) | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx |
| Carba-R | | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| KPC | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| NDM | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| Oxa-48 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| MBL | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| ESBL | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| Other | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| ram-negative, Proteus spp., n(%)<br>Beta-lactamase identified: | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| 0 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| 1 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| 2 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| 3 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| >3 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Unknown/not tested | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x |
| Ambler's class, n(%) | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx |
| A | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| В | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| С | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |
| D | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x |


 $Path: $$ \Path: $$ \operatorname{Local} BioStat Pfizer \array* Documentation \array* Descriptions $$ Path: $$ \array* Descriptions $$ Path: $$ \array* Description \array* Descri$ 

Title: Annotated TLF Shells

Document:

Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN** 

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Acinetobacter baumanii, n(%) | хx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| C | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Acinetobacter spp., n(%) | | | | | | |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | Page <b>88</b> of |

 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

V2.0 Version Number: Version Date: 11 January 2022

Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN** 

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Enterobacter cloacae, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | Page <b>89</b> of |

 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

V2.0 Version Number: Version Date: 11 January 2022

Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN** 

| | cIAI | (N=xx) | cuti (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Enterobacter spp., n(%) | | | | | | |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Citrobacter spp, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | Page <b>90</b> of |

 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

V2.0 Version Number: Version Date: 11 January 2022

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| <u> </u> | | | | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| Unknown/not tested | xx | (xx.x) | хх (хх.х) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Serratia spp., n(%)<br>Beta-lactamase identified: | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

 $Path: \underline{\Quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$ 

Title: Annotated TLF Shells


Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx |
|---|---|---|---|---|---|---|
| 0xa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Morganella morganii, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Salmonella spp., n(%) Beta-lactamase identified: | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


PFIZER 

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Shigella spp, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | | | Page <b>93</b> of |

 $Path: \underline{\Quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$ 

Title: Annotated TLF Shells

Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN** 

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-negative, Pseudomonas aeruginosa, n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Pseudomonas spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Beta-lactamase identified: | | | | | | |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| | | | | | | Page <b>94</b> of 1 |

 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

Document:

V2.0 Version Number: Version Date: 11 January 2022

PFIZER 
Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS **PLAN** 

| | cIAI | (N=xx) | cuti (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CTM-X | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | хx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Haemophilus influenzae, n(%) | хx | (xx.x) | xx (xx.x) | хх (хх.х) | xx (xx.x) | xx (xx.x) |
| ram-negative, Haemophilus spp., n(%) | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ram-negative, Other, n(%) Beta-lactamase identified: | хx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 0 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >3 | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/not tested | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's class, n(%) | | | | | | |
| n | | хx | xx | xx | xx | xx |
| A | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| С | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| D | хx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ambler's type, n(%) | | | | | | |
| n | | xx | xx | xx | xx | xx |
| Carba-R | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| KPC | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | - | • | - | Page <b>95</b> of <b>1</b> |

 $\label{thm:lem:path$ Document:

Title: Annotated TLF Shells

V2.0 Version Number: Version Date: 11 January 2022

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | cIAI | (N=xx) | cUTI (N=xx) | HAP/VAP (N=xx) | Other (N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|---|
| NDM | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxa-48 | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ESBL | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CTM-X | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre>Gram positive, Staphylococcus aureus, n(%) Is it an MRSA (methicillin-resistant S. aureus)?</pre> | ж | (xx.x) | хх (хх.х) | xx (xx.x) | жж (жж.ж) | xx (xx.x) |
| Yes | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown, n | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre>Gram positive, Enterococcus spp., n(%) Is it a VRE (vancomycin resistant Enterococcus)?</pre> | хх | (xx.x) | хх (хх.х) | <b>хх</b> (хх.х) | xx (xx.x) | хх (хх.х) |
| Yes | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown, n | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram positive, Streptococcus spp. | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gram-positive, other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mycobacterium abscessus | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, Bacteroides spp. | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anareobes, Peptostreptococcus spp. | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, Clostridium spp. | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, Prevotella spp. | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, other | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anaerobes, other specify | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other Bacterial Agent | xx | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


#### Zavicefta

C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

**PLAN** 

The microbiological outcomes analysis set (MOD) has all exposed to ceftazidime-avibactam  $\geq$  72 hours and  $\geq$  1 non-missing microbiological outcome.

Table 22.2 Clinical Microbiological Evaluation after initial antibiotic therapy but before ceftazidime-avibactam therapy by Indication Overall (FAS72+)

Table 22.3 Clinical Microbiological Evaluation after initiation or during ceftazidime-avibactam therapy by Indication

Overall (FAS72+)

Table 22.4 Clinical Microbiological Evaluation after end of ceftazidime-avibactam therapy by Indication Overall (FAS72+)

Table 22.5 Clinical Microbiological Evaluation after end of any antibiotic therapy by Indication Overall (FAS72+)
Table 22.6 Latest Microbiological Evaluation before start of ceftazidime-avibactam therapy by Indication Overall (FAS72+)


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Version Number: Version Date: V2.0

11 January 2022

Table 23.1.1 Gram-negative Pathogen Susceptibility to Antibiotics by cIAI Overall (FAS72+)

| Timing on Sample collection | Before initial<br>antibiotic<br>Therapy | After initial antibiotic therapy but before ceftazidime-avibactam therapy | After initiation<br>or during<br>ceftazidime-<br>avibactam<br>therapy | After end of<br>ceftazidime-<br>avibactam<br>therapy | After end of an antibiotic therapy |
|---|---|---|---|---|---|
| Overall | | <b></b> | | | |
| All Gram-negative bacterial pathogens, | | | | | |
| n [1] | | | | | |
| Pathogen identified and tested for susceptibility | XX | XX | xx | XX | XX |
| Antibiotic resistance by Gram-negative bacterial pathogens (all pathogens,) n | | | | | |
| (%) [2] | | | | | |
| n [1] (pathogens) | XX | XX | xx | XX | XX |
| Aminoglycosides | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Amphenicol | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Carbapenems | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cephalosporins | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cephalosporin/beta-lactamase inhibitor | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Glycopeptides | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Glycylcicline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lipopeptides | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Macrolides | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mono Bactam | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Nitroimidazole | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxalolidinones | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Penicillins | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Penicillins and beta-lactamase | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| inhibitors | | | | | |
| individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Quinolones | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Streptogramins | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tetracycline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


#### Zavicefta

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

PLAN

Other Agents xx (xx.x) x

Repeat this table for the following specific pathogens:

- Antibiotic resistance by Gram negative, Escherichia Coli, n (%)[2]
- Antibiotic resistance by Gram negative, Proteus spp. , n (%)[2]
- Antibiotic resistance by Gram negative, Klebsiella spp., n (%)[2]
- Antibiotic resistance by Gram negative, Enterobacter spp., n (%)[2]
- Antibiotic resistance by Gram negative, Citrobacter spp., n (%)[2]
- Antibiotic resistance by Gram negative, Serratia spp., n (%)[2]
- Antibiotic resistance by Gram negative, Haemophilus spp., n (%)[2]
- Antibiotic resistance by Gram negative, Morganella morganii , n (%)[2]
- Antibiotic resistance by Gram negative, Acinetobacter spp. , n (%)[2]
- Antibiotic resistance by Gram negative, Pseudomonas aeruginosa, n (%)[2]
- Antibiotic resistance by Gram negative, Salmonella spp., n (%)[2]


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


PFIZER 

#### Zavicefta

Document:

## C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

- Antibiotic resistance by Gram negative, Shigella spp., n (%)[2]
- Antibiotic resistance by Gram negative, Other, n (%)[2]

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

- [1] The n is the number of pathogens identified and tested for pathogen susceptibility.
- [2] The n and percentage in each table cell are: number of pathogens tested against the particular antibiotic (or class), and the percentage which were found resistant to the particular antibiotic (or class), respectively.

Antibiotic resistance is sorted by Therapeutic class, and antibiotics by alphabetical order.

Antibiotics are sorted by therapeutic class and antibiotics within the class are sorted by alphabetical order.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 23.1.2 Gram-negative Pathogen Susceptibility to Antibiotics by cUTI Overall (FAS72+)
Table 23.1.3 Gram-negative Pathogen Susceptibility to Antibiotics by HAP/VAP Overall (FAS72+)
Table 23.1.4 Gram-negative Pathogen Susceptibility to Antibiotics by Other Overall (FAS72+)
Table 23.1.5 Gram-negative Pathogen Susceptibility to Antibiotics by All indications Overall (FAS72+)
Table 23.2.1 Gram-negative Multi Drug Resistance for cIAI Overall (FAS72+)

| Timing on Sample collection | Before<br>initial<br>antibiotic<br>Therapy | After initial antibiotic therapy but before ceftazidime- avibactam therapy | After initiation or during ceftazidime- avibactam therapy | After end of<br>ceftazidime-<br>avibactam<br>therapy | After end of<br>any<br>antibiotic<br>therapy |
|---|---|---|---|---|---|
| Overall | | cherapy | | | |
| Gram-negative Multi-resistant | | | | | |
| pathogen n (%)[1] | | | | | |
| n [1] (pathogens) | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n [1](pathogens) Aminoglycosides Amphenicol | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx (xx.x)<br>xx (xx.x) |
| Carbapenems | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cephalosporins | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cephalosporin/beta-lactamase<br>inhibitor | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Glycopeptides | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Glycylcicline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lipopeptides | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Macrolides | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Mono Bactam | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Nitroimidazole | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oxalolidinones | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

#### Zavicefta

## C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Penicillins | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|---|
| Penicillins and beta-lactamase | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| inhibitors | | | | | |
| Individual antibiotics | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Quinolones | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Streptogramins | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tetracycline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other Agents | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Repeat this table for the following specific pathogens:

- Gram negative, Escherichia Coli
- Gram negative, Proteus spp.
   Gram negative, Klebsiella spp.
- Gram negative, Enterobacter spp.
- Gram negative, Citrobacter spp.
- Gram negative, Serratia spp.
- Gram negative, Haemophilus spp.
- Gram negative, Morganella morganii
- Gram negative, Acinetobacter spp.
- Gram negative, Pseudomonas aeruginosa
- Gram negative, Salmonella spp.
- Gram negative, Shigella spp.
- Gram negative, Other

Document:

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

- [1] The n is the number of pathogens identified and tested for multi-drug resistance.
- [2] The n and percentage in each table cell are: number of pathogens tested against the particular antibiotic (or class), and the percentage which were found resistant to the particular antibiotic (or class), respectively.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Table 23.2.2 Gram-negative Multi Drug Resistance for cUTI Overall (FAS72+)
Table 23.2.3 Gram-negative Multi Drug Resistance for HAP/VAP Overall (FAS72+)
Table 23.2.4 Gram-negative Multi Drug Resistance for Other Overall (FAS72+)
Table 23.2.5 Gram-negative Multi Drug Resistance for All indications Overall (FAS72+)
Table 24.1.1 Gram-negative Pathogen Susceptibility to Antibiotics by cIAI Europe (FAS72+)
Table 24.1.2 Gram-negative Pathogen Susceptibility to Antibiotics by cUTI Europe (FAS72+)
Table 24.1.3 Gram-negative Pathogen Susceptibility to Antibiotics by HAP/VAP Europe (FAS72+)
Table 24.1.4 Gram-negative Pathogen Susceptibility to Antibiotics by Other Europe (FAS72+)
Table 24.1.5 Gram-negative Pathogen Susceptibility to Antibiotics by All Indications Europe (FAS72+)

Table 24.2.1 Gram-negative Multi Drug Resistance for cIAI in Europe (FAS72+)

Table 24.2.2 Gram-negative Multi Drug Resistance for cUTI Europe (FAS72+)

Table 24.2.3 Gram-negative Multi Drug Resistance for HAP/VAP Europe (FAS72+)

Table 24.2.4 Gram-negative Multi Drug Resistance for Others Europe (FAS72+)

Table 24.2.5 Gram-negative Multi Drug Resistance for All Indications Europe (FAS72+)

Table 25.1.1 Gram-negative Pathogen Susceptibility to Antibiotics for cIAI in LATAM (FAS72+)

Table 25.1.2 Gram-negative Pathogen Susceptibility to Antibiotics for cUTI LATAM (FAS72+)

Table 25.1.3 Gram-negative Pathogen Susceptibility to Antibiotics for HAP/VAP LATAM (FAS72+)

Table 25.1.4 Gram-negative Pathogen Susceptibility to Antibiotics for Others LATAM (FAS72+)

Table 25.1.5 Gram-negative Pathogen Susceptibility to Antibiotics for All Indications LATAM (FAS72+)

Table 25.2.1 Gram-negative Multi Drug Resistance for cIAI in LATAM (FAS72+)
Table 25.2.2 Gram-negative Multi Drug Resistance for cUTI LATAM (FAS72+)
Table 25.2.3 Gram-negative Multi Drug Resistance for HAP/VAP LATAM (FAS72+)
Table 25.2.4 Gram-negative Multi Drug Resistance for Others LATAM (FAS72+)
Table 25.2.5 Gram-negative Multi Drug Resistance for All Indications LATAM (FAS72+)


Document:

 $Path: \underline{\downward{\downw$ 

Title: Annotated TLF Shells


V2.0 11 January 2022

| | | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Clinical outcome fo | r the initial hospitalization | | | | | |
| Overall outcome of | ceftazidime-avibactam (any therapy) | | | | | |
| n(%) | | xx | xx | xx | хх | xx |
| Treatment Succes | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment Failur | e [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indeterminate | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| herapy type | | | | | | |
| n (%) | | xx | xx | xx | xx | xx |
| Monotherapy | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Combination ther | гару | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| overall outcome of<br>All monotherapy re | ceftazidime-avibactam in monotherapy<br>gimens) | | | | | |
| n (%) | | xx | xx | xx | xx | xx |
| Treatment Succes | s | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | хх ( хх.х |
| Treatment Failur | re | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x |
| Indeterminate | | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| | ceftazidime-avibactam in combined therap | У | | | | |
| (All combined thera | py regimens) | | | | | |
| n (%) | | xx | xx | xx | xx | xx |
| Treatment Succes | SS | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | хх ( хх.х |
| Treatment Failu | re | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x |
| Indeterminate | | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x |
| linical outcome at | 60 days post-discharge [b] | | | | | |
| verall Outcome of | ceftazidime-avibactam (any therapy) | | | | | |
| | | | | | Pag | ge <b>104</b> of <b>1</b> |
| ocument: | Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioSta | at\Pfizer\Zavicefta\Dc | cumentation\Spe | ecifications | | |
| | Title: Annotated TLF Shells | | | | | |
| | | | Version Number: | : | | V2 |
| | | | Version Date: | | | 11 January 20 |

| | cIAI<br>(N=xx) | cUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|
| n (%) | xx | xx | xx | xx | xx |
| Treatment success | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment failure | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Indeterminate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapy type | | | | | |
| n (%) | xx | xx | хх | xx | xx |
| Monotherapy | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Combination Therapy | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Overall outcome of ceftazidime-avibactam in monotherapy (All monotherapy regimens) | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| Treatment Success | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Treatment Failure | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Indeterminate | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | хх ( хх.х) |
| Overall outcome of ceftazidime-avibactam in combined therapy (All combined therapy regimens) | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| Treatment Success | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Treatment Failure | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Indeterminate | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Clinical outcome at 60 days post-treatment [a] | | | | | |
| Overall Outcome of ceftazidime-avibactam (any therapy) | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment success | xx (xx.x) | AA (AA.A) | 1111 (1111:11) | 1111 (1111:11) | 1111 (1111:11) |
| Treatment success Treatment failure | xx (xx.x)<br>xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | cIAI<br>(N=xx) | cUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|
| Therapy type | | · | · | · | |
| n (%) | xx | xx | xx | xx | xx |
| Monotherapy | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Combination Therapy | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Overall outcome of ceftazidime-avibactam in monotherapy | | | | | |
| (All monotherapy regimens) | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| Treatment Success | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Treatment Failure | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Indeterminate | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Overall outcome of ceftazidime-avibactam in combined therapy | | | | | |
| (All combined therapy regimens) | | | | | |
| n (%) | | xx | xx | xx | xx |
| | xx | | | | |
| Treatment Success | | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| | xx ( xx.x) | | | | |
| Treatment Failure | | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | жж ( жж.ж) |
| | xx ( xx.x) | | | | |
| Indeterminate | | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| | xx ( xx.x) | | | | |

The clinical outcomes analysis set (COD) has all patients exposed to ceftazidime-avibactam  $\geq$  72 hours and  $\geq$  1 non-missing clinical outcome.

cIAI: Complicated Intra-Abdominal Infection; cUTI: Complicated Urinary Tract Infection; HAP: Hospital-Acquired Pneumonia; VAP: Ventilator-Associated Pneumonia.

125 patients not evaluated (97 died during initial hospitalization, 10 died after discharge, 12 missing evaluation/death date, 6 criteria not met).


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Version Number: Version Date: V2.0 11 January 2022 Table 26.1 Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Escherichia coli Overall (COD)

Table 26.2 Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Klebsiella spp. Overall (COD)

Table 26.3 Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Enterobacter spp. Overall (COD)

Table 26.4 Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Pseudomonas spp. Overall (COD)

Table 26.5 Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients Infected by Other Gramnegative Bacteria Overall (COD)

Table 26.6 Clinical Evaluation Outcome (Success, Failure, Indeterminate) by Indication in Patients with no Pathogens identified (COD)


Document: Path: \quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


V2.0


11 January 2022

Table 27 Logistic Regression Univariate Model 1 for Clinical Success at Initial Hospitalization (COD)

| | n (%) | Odds Ratio | 95% CI | p-value |
|-------------------------------|----------|------------|------------|---------|
| Age at Baseline | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Baseline BMI kg/m²) | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Gender | x (xx.x) | | | |
| Male | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Female | x (xx.x) | Reference | | |
| Region | x (xx.x) | | | |
| Latam | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Europe | x (xx.x) | Reference | | |
| Country | x (xx.x) | | | |
| Austria | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Germany | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| France | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Italy | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Russia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Spain | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Argentina | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Brazil | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Colombia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| UK | x (xx.x) | Reference | | |
| Employment status | x (xx.x) | | | |
| Full Time | x.xx | x.xx, x.xx | x.xxx | x.xxx |
| Part Time | x.xx | x.xx, x.xx | x.xxx | x.xxx |
| Retired | x.xx | x.xx, x.xx | x.xxx | x.xxx |
| Unemployed | x (xx.x) | Reference | | |
| Recent hospitalization | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| LOS of recent hospitalization | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| History of antibiotic exposure | x (xx.x) | | | <del>_</del> |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Treated with betalactam within the past 3 months | x (xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Recent healthcare procedure | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Healthcare Resource Utilization during Initial | x (xx.x) | | | |
| Hospitalization | | | | |
| Mechanical ventilation | x(xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Dialysis | x(xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Tracheostomy | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Surgical intervention | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Percutaneous procedure | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Other | x (xx.x) | Reference | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Foreign travel in the past 3 months | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pre-treatment disease severity (APACHE II score) | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| Any Deyo-Carlson Comorbidity | | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| DCCI score | x (xx.x) | | | |
| 0 | x(xx.x) | Reference | | |
| 1 | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 2 | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 3 | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ≥4 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Any non Deyo-Carlson Comorbidity | | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Indication | x (xx.x) | | | |
| Other | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| CIAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| HAP/VAP | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| cUTI | x (xx.x) | Reference | | |
| Source of admission | x (xx.x) | | | |
| Outpatient | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Long-term care facility | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Transfer from acute care hospital | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Other | x (xx.x) | Reference | | |
| Ward admitted for initial hospitalization | x (xx.x) | | | |
| Surgical | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Medical | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Onco-hematology | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Infectious disease | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ICU | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Other | x (xx.x) | Reference | | |
| Patient attended ICU during hospitalization, n (%) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|------------------------------|----------|------------|------------|---------|
| Source of infection | x (xx.x) | | | |
| HAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| HCAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| CAI | x (xx.x) | Reference | | |
| Bacteria (categorical) | | | | |
| Escherichia coli | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Klebsiella spp., | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Enterobacter spp. | x (xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Pseudomonas spp. | x(xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Other Gram-negative bacteria | x (xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pregnancy (only Female) | x (xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use > 14 drinks/week | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Smoker | x (xx.x) | | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Smoker status | | | | |
| Current smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Previous smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Unknown | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Never smoked | x (xx.x) | Reference | | |
| Patient's infection by multi-resistant pathogen | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |

BMI-body mass index

Document:

LOS- Length of Stay, VAP- Ventilator-associated pneumonia

n represents the number of non-Missing, n values per regression variable.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


V2.0

11 January 2022

Table 28 Logistic Regression Multivariable Model 1 for Clinical Success (COD)

| | n (%) | Odds Ratio | 95% CI | p-value |
|-------------------------------|----------|------------|------------|---------|
| Age at Baseline | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Baseline BMI kg/m²) | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Gender | x (xx.x) | | | |
| Male | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Female | x (xx.x) | Reference | | |
| Region | x (xx.x) | | | |
| Latam | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Europe | x (xx.x) | Reference | | |
| Country | x (xx.x) | | | |
| Austria | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Germany | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| France | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Italy | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Russia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Spain | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Argentina | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Brazil | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Colombia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| UK | x (xx.x) | Reference | | |
| Employment status | x (xx.x) | | | |
| Full Time | x.xx | x.xx, x.xx | x.xxxx | x.xxx |
| Part Time | x.xx | x.xx, x.xx | x.xxxx | x.xxx |
| Retired | x.xx | x.xx, x.xx | x.xxxx | x.xxx |
| Unemployed | x (xx.x) | Reference | | |
| Recent hospitalization | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| LOS of recent hospitalization | x (xx.x) | x.xx | x.xx, x.xx | x.xxxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

| History of antibiotic exposure | x (xx.x) | | | |
|---|---|---|---|---|
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Treated with betalactam within the past 3 months | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | · | |
| Recent healthcare procedure | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | 22.1.1.7 | |
| Healthcare Resource Utilization during Initial | x (xx.x) | | | |
| Hospitalization | A (AA.A) | | | |
| Mechanical ventilation | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Dialysis | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Tracheostomy | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Surgical intervention | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Percutaneous procedure | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Other | x (xx.x) | Reference | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Foreign travel in the past 3 months | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pre-treatment disease severity (APACHE II score) | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Any Deyo-Carlson Comorbidity | | | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
|---|---|---|---|---|
| No | x (xx.x) | Reference | | |
| DOOT | / | | | |
| DCCI score | x (xx.x) | | | |
| 0 | x (xx.x) | Reference | | |
| 1 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 2 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 3 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ≥4 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Any non Deyo-Carlson Comorbidity | | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Indication | / | | | |
| Other | x (xx.x)<br>x (xx.x) | x.xx | V VV V V | x.xxxx |
| CIAI | x (xx.x) | x.xx<br>x.xx | x.xx, x.xx | x.xxxx |
| HAP/VAP | | · | x.xx, x.xx | |
| | x (xx.x) | X.XX | x.xx, x.xx | x.xxx |
| CUTI | x (xx.x) | Reference | | |
| Source of admission | x (xx.x) | | | |
| Outpatient | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Long-term care facility | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Transfer from acute care hospital | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Other | x (xx.x) | Reference | | |
| Ward admitted for initial hospitalization | x (xx.x) | | | |
| Surgical | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Medical | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Onco-hematology | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Infectious disease | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ICU | x (xx.x) | x.xx | x.xx, x.xx | x.xxxx |
| Other | x (xx.x) | Reference | | |
| Deticat attended TON dening beginning to | () | | | |
| Patient attended ICU during hospitalization, n (%) | x (xx.x) | | | |
| Yes | x (xx . x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Source of infection | x (xx.x) | | | |
| HAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| HCAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
|------------------------------|----------|-----------|------------|-------|
| CAI | x (xx.x) | Reference | | |
| Bacteria (categorical) | | | | |
| Escherichia coli | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Klebsiella spp., | x(xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Enterobacter spp. | x(xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pseudomonas spp. | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Other Gram-negative bacteria | x(xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pregnancy (only Female) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use > 14 drinks/week | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Smoker | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | · | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

#### Zavicefta

Document:

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### **PLAN**

| Smoker status | | | | |
|---|---|---|---|---|
| Current smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Previous smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Unknown | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Never smoked | x (xx.x) | Reference | | |
| Patient's infection by multi-resistant pathogen | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |

[1] Note: Since Zavicefta is not active against Acinetobacter; it's then a good factor for failure The clinical outcomes analysis set (COD) has all patients exposed to ceftazidime-avibactam  $\geq$  72 hours and  $\geq$  1 non-missing clinical outcome.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 29 Logistic Regression Univariate Model 2 for Clinical Success at Initial Hospitalization (COD)

| | n (%) | Odds Ratio | 95% CI | p-value |
|-------------------------------|----------|------------|------------|---------|
| Age at Baseline | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Baseline BMI kg/m²) | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Gender | x (xx.x) | | | |
| Male | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Female | x (xx.x) | Reference | | |
| Region | x (xx.x) | | | |
| Latam | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Europe | x (xx.x) | Reference | | |
| Country | x (xx.x) | | | |
| Austria | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Germany | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| France | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Italy | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Russia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Spain | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Argentina | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Brazil | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Colombia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| UK | x (xx.x) | Reference | | |
| Employment status | x (xx.x) | | | |
| Full Time | x.xx | x.xx, x.xx | x.xxx | x.xxx |
| Part Time | x.xx | x.xx, x.xx | x.xxx | x.xxx |
| Retired | x.xx | x.xx, x.xx | x.xxx | x.xxx |
| Unemployed | x (xx.x) | Reference | | |
| Recent hospitalization | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| LOS of recent hospitalization | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| History of antibiotic exposure | x (xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Treated with betalactam within the past 3 months | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Recent healthcare procedure | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Healthcare Resource Utilization during Initial | x (xx.x) | | | |
| Hospitalization | | | | |
| Mechanical ventilation | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Dialysis | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Tracheostomy | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Surgical intervention | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Percutaneous procedure | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Other | x (xx.x) | Reference | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Foreign travel in the past 3 months | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pre-treatment disease severity (APACHE II score) | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| Any Deyo-Carlson Comorbidity | | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| DCCI score | x (xx.x) | | | |
| 0 | x(xx.x) | Reference | | |
| 1 | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 2 | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 3 | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ≥4 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Any non Deyo-Carlson Comorbidity | | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Indication | x (xx.x) | | | |
| Other | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| CIAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| HAP/VAP | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| cUTI | x (xx.x) | Reference | | |
| Source of admission | x (xx.x) | | | |
| Outpatient | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Long-term care facility | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Transfer from acute care hospital | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Other | x (xx.x) | Reference | | |
| Ward admitted for initial hospitalization | x (xx.x) | | | |
| Surgical | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Medical | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Onco-hematology | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Infectious disease | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ICU | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Other | x (xx.x) | Reference | | |
| Patient attended ICU during hospitalization, n (%) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|------------------------------|----------|------------|------------|---------|
| Source of infection | x (xx.x) | | | |
| HAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| HCAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| CAI | x (xx.x) | Reference | | |
| Bacteria (categorical) | | | | |
| Escherichia coli | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Klebsiella spp., | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Enterobacter spp. | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pseudomonas spp. | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Other Gram-negative bacteria | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pregnancy (only Female) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use > 14 drinks/week | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Smoker | x (xx.x) | | | |


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Smoker status | | | | |
| Current smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Previous smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Unknown | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Never smoked | x (xx.x) | Reference | | |
| Patient's infection by multi-resistant pathogen | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Was the patient diagnosed with COVID-19? | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Not applicable | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Patients with bacteriemia overall, n(%) | | | | |
| Primary | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Secondary | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Immunocompromised patients overall, n(%) | x (xx.x) | | | |
| l'es | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Patients with lower dose of Zavicefta overall, | x (xx.x) | | | |
| n (%) | | | | |
| les es | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |

Table 30 Logistic Regression Multivariable Model 2 for Clinical Success at Initial Hospitalization

| Age at Baseline | x (xx.x) | x.xx | X.XX, X.XX | y-varue<br>x.xxxx |
|-----------------|----------|------------|------------|-------------------|
| | n (%) | Odds Ratio | 95% CI | p-value |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Zavicefta
C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| Baseline BMI kg/m²) | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Gender | x (xx.x) | | | |
| Male | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Female | x (xx.x) | Reference | | |
| Region | x (xx.x) | | | |
| Latam | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Europe | x (xx.x) | Reference | | |
| Country | x (xx.x) | | | |
| Austria | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Germany | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| France | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Italy | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Russia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Spain | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Argentina | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Brazil | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Colombia | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| UK | x (xx.x) | Reference | | |
| Employment status | x (xx.x) | | | |
| Full Time | x.xx | x.xx, x.xx | x.xxxx | x.xxx |
| Part Time | x.xx | x.xx, x.xx | x.xxxx | x.xxx |
| Retired | x.xx | x.xx, x.xx | x.xxxx | x.xxx |
| Unemployed | x (xx.x) | Reference | | |
| Recent hospitalization | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| LOS of recent hospitalization | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| History of antibiotic exposure | x (xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Treated with betalactam within the past 3 months | x (xx.x) | | | |


 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Recent healthcare procedure | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Healthcare Resource Utilization during Initial | x (xx.x) | | | |
| Mechanical ventilation | x(xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Dialysis | x(xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Tracheostomy | x(xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Surgical intervention | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Percutaneous procedure | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x(xx.x) | Reference | | |
| Other | x(xx.x) | Reference | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Foreign travel in the past 3 months | x (xx.x) | | | |
| Yes | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Pre-treatment disease severity (APACHE II score) | x(xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Any Deyo-Carlson Comorbidity | | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| DCCI score | x (xx.x) | | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| 0 | x (xx.x) | Reference | 350 01 | p varac |
| 1 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 2 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| 3 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ≥4 | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Any non Deyo-Carlson Comorbidity | | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Indication | x (xx.x) | | | |
| Other | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| cIAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| HAP/VAP | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| CUTI | x (xx.x) | Reference | | |
| Source of admission | x (xx.x) | | | |
| Outpatient | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Long-term care facility | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Transfer from acute care hospital | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Other | x (xx.x) | Reference | | |
| Ward admitted for initial hospitalization | x (xx.x) | | | |
| Surgical | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Medical | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Onco-hematology | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Infectious disease | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| ICU | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Other | x (xx.x) | Reference | | |
| Patient attended ICU during hospitalization, n (%) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Source of infection | x (xx.x) | | | |
| HAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| HCAI | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| CAI | x (xx.x) | Reference | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|------------------------------|----------|------------|------------|---------|
| Bacteria (categorical) | | | | |
| Escherichia coli | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Klebsiella spp., | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Enterobacter spp. | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | • | |
| Pseudomonas spp. | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | , | |
| Other Gram-negative bacteria | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | , | |
| Pregnancy (only Female) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Alcohol use > 14 drinks/week | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Smoker | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Smoker status | | | | |
| Current smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |

Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


| | n (%) | Odds Ratio | 95% CI | p-value |
|---|---|---|---|---|
| Previous smoker | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Unknown | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Never smoked | x (xx.x) | Reference | | |
| Patient's infection by multi-resistant pathogen | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Was the patient diagnosed with COVID-19? | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Not applicable | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Patients with bacteriemia overall, n(%) | | | | |
| Primary | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| Secondary | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Immunocompromised patients overall, n(%) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |
| Patients with lower dose of Zavicefta overall, n(%) | x (xx.x) | | | |
| Yes | x (xx.x) | x.xx | x.xx, x.xx | x.xxx |
| No | x (xx.x) | Reference | | |

<sup>[1]</sup> Note: Since Zavicefta is not active against Acinetobacter; it's then a good factor for failure The clinical outcomes analysis set (COD) has all patients exposed to ceftazidime-avibactam  $\geq$  72 hours and  $\geq$  1 non-missing clinical outcome.

The logistic regression is modelling clinical success versus failure with clinical indeterminate set to missing.


V2.0

Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Version Number: Version Date: 11 January 2022

Table 31 Microbiological Evaluation Outcome (Success, Failure, Emergent Infections) by Indication Overall (MOD) - Since few patients had samples taken after start of Zavicefta, table will not me produced.

Table 31.1 Microbiological Evaluation Outcome by Indication in Patients Infected by Escherichia Coli Overall (MOD)

Since few patients had samples taken after start of Zavicefta, table will not me produced.

Table 31.2 Microbiological Evaluation Outcome by Indication in Patients Infected by *Klebsiella* spp. Overall (MOD) Since few patients had samples taken after start of Zavicefta, table will not me produced.

Table 31.3 Microbiological Evaluation Outcome by Indication in Patients Infected by *Enterobacter* spp. Overall (MOD) Since few patients had samples taken after start of Zavicefta, table will not me produced.

Table 31.4 Microbiological Evaluation Outcome by Indication in Patients Infected by *Pseudomonas* spp. Overall (MOD) Since few patients had samples taken after start of Zavicefta, table will not me produced.

Table 31.5 Microbiological Evaluation Outcome by Indication in Patients Infected by Other Gram-negative bacteria Overall (MOD)

Since few patients had samples taken after start of Zavicefta, table will not me produced.


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


11 January 2022

V2.0

Table 32 Prevalence of Hospital Readmissions by Indication Overall (FAS72+)

| | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| he number of patients readmitted to hospital within 0 days post-initial discharge, n (%) | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown, n | <b>xx</b> ( <b>xx</b> . <b>x</b> ) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | хх | хх | xx | хх | |
| he number of hospital readmissions within 60 days ost-initial discharge, n | | | | | |
| n | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| atient readmitted within, n (%) | | | | | |
| Discharge-30 Days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 31-60 days | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| uration of re-hospitalization (Days)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Missing, n | xx | хх | хх | xx | хх |
| eason for readmission | | | | | |
| n | хx | xx | хx | хx | xx |
| | | | | Dage 1 | <b>29</b> of <b>159</b> |

Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

| | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Unrelated to the infection | хх (хх.х) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Infection recurrence | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Secondary infection | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Missing, n | xx | xx | xx | xx | xx |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

Version Date: 11 J

11 January 2022

V2.0

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum

<sup>[1]</sup> Duration of Re-hospitalization = Date of discharge - Date of readmission
#### Zavicefta

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

**PLAN** 

Table 32.1 Prevalence of Hospital Readmissions by Indication in Patients Infected by Escherichia Coli Overall (FAS72+)

For all tables 34.1 through 34.6: add the footnotes: FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours. SD- Standard deviation, Q1- Quartile one, Q3- Quartile three. Min- minimum, Max- Maximum [1] Duration of Re-hospitalization = Date of discharge - Date of readmission

Table 32.2 Prevalence of Hospital Readmissions by Indication in Patients Infected by Klebsiella spp. Overall (FAS72+)

Table 32.3 Prevalence of Hospital Readmissions by Indication in Patients Infected by Enterobacter spp. Overall (FAS72+)

Table 32.4 Prevalence of Hospital Readmissions by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72+)

Table 32.5 Prevalence of Hospital Readmissions by Indication in Patients Infected by Other Gram-negative Bacteria Overall (FAS72+)

Table 32.6 Prevalence of Hospital Readmissions by Indication in Patients Infected by no Pathogen Identified Overall (FAS72+)


Document: Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


V2.0


Table 33 Vital Status and Mortality Rates by Indication Overall (FAS72+)

| | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Patient status at date of last available record | | | | | |
| n(%) | XX | XX | XX | XX | XX |
| Alive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient Died | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx | XX | XX | XX | xx |
| Timing of death (if patient died)[1] | | | | | |
| n (%) | XX | XX | XX | XX | XX |
| During Index hospitalization | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Within 30 days of discharge | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Within 60 days of discharge | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx | xx | XX | XX | xx |
| Total in-hospital mortality rate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 95% CI | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |
| Cumulative mortality rate at 30 days post- | | | | | |
| discharge [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 95% CI | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |
| Cumulative mortality rate at 60 days post- | | | | | |
| discharge [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 95% CI | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |

#### FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

- [1] The post-discharge timing of death are from 1-30 days and is 31-60 days, inclusive.
- [2] Cumulative mortality up to 30 days post-discharge, including in-hospital mortality
- [3] Cumulative mortality up to 60 days post-discharge, including in-hospital mortality


 $\label{thm:path:local} Path: $$ \underline{\CBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$$ 

Title: Annotated TLF Shells

Document:

#### Zavicefta

Document:

C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

Table 33.1 Vital Status and Mortality Rates by Indication in Patients Infected by Escherichia Coli Overall (FAS72+)

For all tables 35.1 through 35.6: add the footnotes:

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam  $\geq$  72 hours.

- [1] The post-discharge timing of death are from 1-30 days and is 31-60 days, inclusive.
- [2] Cumulative mortality up to 30 days post-discharge, including in-hospital mortality
- [3] Cumulative mortality up to 60 days post-discharge, including in-hospital mortality

Table 33.2 Vital Status and Mortality Rates by Indication in Patients Infected by Klebsiella spp. Overall (FAS72+)

Table 33.3 Vital Status and Mortality Rates by Indication in Patients Infected by Enterobacter spp. Overall (FAS72+)

Table 33.4 Vital Status and Mortality Rates by Indication in Patients Infected by Pseudomonas spp. Overall (FAS72+)

Table 33.5 Vital Status and Mortality Rates by Indication in Patients Infected by Other Gram-negative Bacteria Overall (FAS72+)

Table 33.6 Vital Status and Mortality Rates by Indication by no Pathogen Identified Overall (FAS72+)


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


11 January 2022

V2.0

### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### **PLAN**

Table 34 Vital Status and Mortality Rates in Patients with Ceftazidime-Avibactam Exposure <72 Hours by Indication Overall (FAS72-)

| | cIAI<br>(N=xx) | CUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL<br>(N=xx) |
|---|---|---|---|---|---|
| Patient status at date of last available | | | | | |
| record | | | | | |
| n (%) | xx | xx | xx | xx | xx |
| Alive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient Died | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx | xx | xx | xx | xx |
| Total in-hospital mortality rate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 95% CI | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |

FAS72- analysis set has all patients exposed to ceftazidime-avibactam < 72 hours.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

SD- Standard deviation, Q1- Quartile one, Q3- Quartile three, Min- Minimum, Max- Maximum.

<sup>[1]</sup> Percentages computed among the total number of patients by Country.

<sup>[2]</sup> Date of death - Date of treatment initiation.

<sup>[3]</sup> Percentages computed among the total number of patients within the category.

Table 35 Antibiotic Therapy After Ceftazidime-Avibactam During the Index Hospitalization by Indication Overall (FAS72+)

| First create Overall table. Repeat table for each of Gram-Negative/ Gram-Positive/ | cIAI<br>(N=xx) | cUTI<br>(N=xx) | HAP/VAP<br>(N=xx) | Other<br>(N=xx) | TOTAL (N=xx) |
|---|---|---|---|---|---|
| Anaerobic/ other (include antifungal, antiviral, other) | | | | | |
| Any antibiotic(s) used for current infection after | | | | | |
| Ceftazidime-avibactam, n (%)[1] | | | | | |
| n | xx | xx | xx | xx | xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing, n | xx | xx | xx | xx | xx |
| Antibiotic class and name (generic name, n(%) [2] | | | | | |
| n | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 3 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic class 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Antibiotic 2 etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total duration of antibiotics used for current infection | | | | | |
| after Ceftazidime-avibactam [3] | | | | | |
| n | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x | xx.x | xx.x | xx.x | xx.x |
| | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| Q1, Q3 | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | | | | Pā | age <b>135</b> of <b>15</b> |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| First create Overall table. | c | IAI | | cUTI | H. | AP/VAP | ( | Other | 7 | TOTAL |
|---|---|---|---|---|---|---|---|---|---|---|
| Repeat table for each of Gram-Negative/ Gram-Positive/ | (I) | N=xx) | ( | N=xx) | ( | N=xx) | ( | N=xx) | ( | N=xx) |
| Anaerobic/ other (include antifungal, antiviral, other) | | | | | | | | | | |
| Missing, n | | хх | | xx | | xx | | xx | | хх |
| n | | xx | | xx | | xx | | xx | | xx |
| Reason for initiating per antibiotic, n(%)[2] | хх | (xx.x) | хх | (xx.x) | хх | (xx.x) | хх | (xx.x) | хx | (xx.x) |
| n | | xx | | xx | | xx | | xx | | xx |
| Clostridium difficile | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| De-escalation | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Disease progression | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Empiric treatment | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Failure of antimicrobial therapy | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Infection | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Microbiology | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Prophylaxis | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Relapse | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Other | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Missing, n | | хх | | xx | | хх | | xx | | хх |
| Reason for discontinuation per antibiotic, n(%) [2] | | | | | | | | | | |
| n | | xx | | xx | | xx | | xx | | xx |
| AE | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | ХX | (xx.x) | xx | (xx.x) |
| Perceived clinical failure/disease progression | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| Isolation of a resistant pathogen | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | ХX | (xx.x) | xx | (xx.x) |
| Preference for empiric coverage | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) | ХX | (xx.x) | xx | (xx.x) |
| Secondary infection requiring regimen change | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Switch to oral therapy | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | хx | (xx.x) | xx | (xx.x) |
| De-escalation | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Cure | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Death | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Other | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| Missing, n | | xx | | xx | | xx | | xx | | xx |

FAS72+ analysis set has all patients exposed to ceftazidime-avibactam ≥ 72 hours.

AE - Adverse event, SD - Standard deviation, Q1- Quartile one, Q3 - Quartile three. Min - minimum, Max - Maximum

[1] Percentages computed among the total number of patients by Country.

Document:

- [2] Percentages computed among the total number of patients within the category.
- [3] Duration of Antibiotic = [Stop Date of Antibiotic Start Date of Antibiotic]


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications
Title: Annotated TLF Shells

Table 36 Adverse Events by Indication Overall (FAS)

| | | CIAI | | CUTI | HA | P/VAP | Other | | 1 | 'OTAL |
|---|---|---|---|---|---|---|---|---|---|---|
| | ( | N=xx) | (1 | N=xx) | (1 | N=xx) | ( | N=xx) | (1 | N=xx) |
| Any adverse event | | | | | | | | | | |
| Patients, n (%) | xx | (xx.x) | хx | (xx.x) | хx | (xx.x) | ХX | (xx.x) | хx | (xx.x) |
| Events, n | | xx | | xx | | ХХ | | xx | | хх |
| Any adverse event leading to discontinuation of | | | | | | | | | | |
| ceftazidime-avibactam | | | | | | | | | | |
| Patients, n (%) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| Events, n | | xx | | хх | | XX | | xx | | XX |
| Any serious adverse event | | | | | | | | | | |
| Patients, n (%) | ХX | (xx.x) | хх | (xx.x) | хx | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| Events, n | | xx | | хх | | XX | | XX | | хх |
| Any fatal serious adverse event | | | | | | | | | | |
| Patients, n (%) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Events, n | | xx | | хх | | XX | | xx | | хх |
| Any non-fatal serious adverse event | | | | | | | | | | |
| Patients, n (%) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| Events, n | | XX | | ХХ | | XX | | XX | | XX |
| Any serious adverse event leading to discontinuation | | | | | | | | | | |
| of ceftazidime-avibactam | | | | | | | | | | |
| Patients, n (%) | ХX | (xx.x) | хх | (xx.x) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| Events, n | | xx | | хх | | xx | | xx | | xx |

The full analysis set (FAS) has all eligible patients.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


11

Table 36.1 Adverse Events Related to Ceftazidime-Avibactam by Indication Overall (FAS)

| | | cIAI<br>N=xx) | | CUTI<br>N=xx) | | AP/VAP<br>N=xx) | Other<br>(N=xx) | | _ | OTAL<br>N=xx) |
|---|---|---|---|---|---|---|---|---|---|---|
| | , | N-AA) | , | N-AA) | , | N-XX) | , | N-AA) | ( | N-AA) |
| Any adverse event | | | | | | | | | | |
| Patients, n (%) | ХX | (xx.x) | хx | (xx.x) | хx | (xx.x) | ХX | (xx.x) | хx | (xx.x) |
| Events, n | | ХХ | | xx | | ХХ | | хх | | ХХ |
| Any adverse event leading to discontinuation of | | | | | | | | | | |
| ceftazidime-avibactam | | | | | | | | | | |
| Patients, n (%) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Events, n | | XX | | XX | | XX | | XX | | xx |
| Any serious adverse event | | | | | | | | | | |
| Patients, n (%) | ХX | (xx.x) | хx | (xx.x) | ХX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| Events, n | | xx | | xx | | xx | | xx | | ХХ |
| Any fatal serious adverse event | | | | | | | | | | |
| Patients, n (%) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) | хx | (xx.x) |
| Events, n | | xx | | xx | | xx | | xx | | xx |
| Any non-fatal serious adverse event | | | | | | | | | | |
| Patients, n (%) | хx | (xx.x) | ХX | (xx.x) | хх | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| Events, n | | xx | | xx | | xx | | xx | | ХХ |
| Any serious adverse event leading to discontinuation of ceftazidime-avibactam | | | | | | | | | | |
| Patients, n (%) | ХX | (xx.x) | хx | (xx.x) | хх | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| Events, n | | XX | | XX | | XX | | XX | | ХХ |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:


Table 37 Adverse Events by System Organ Class by Indication Overall (FAS)

| System organ class | CIAI | CUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any adverse event | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| System organ class 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | хх | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | ХХ | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | хх | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| System organ class 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | хх | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | ХХ | ХХ |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | XX |
| Etc | | | | | |

Document:


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 37.1 Adverse Events Related to Ceftazidime-Avibactam by System Organ Class by Indication Overall (FAS)

| System organ class | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any adverse event | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | XX | XX | XX | xx | ХХ |
| System organ class 1 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | ХХ |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | XX | XX | XX | xx |
| System organ class 2 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | ХХ |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | XX | XX | xx | xx |
| Etc | | | | | |

Document:


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Table 38 Serious Adverse Events by System Organ Class by Indication Overall (FAS)

| (N= xx () x () x () x () x () | (x.x)<br>x | xx | N=xx) (xx.x) xx (xx.x) | xx | N=xx) (xx.x) xx | | N=xx)<br>(xx.x)<br>xx | | (xx.x)<br>xx |
|---|---|---|---|---|---|---|---|---|---|
| xx (2<br>x | x (x . x) | | xx | | | xx | | xx | |
| xx (2<br>x | x (x . x) | | xx | | | xx | | xx | |
| xx (2<br>x | (X.X) | xx | | | XX | | XX | | xx |
| х | | ХХ | (xx.x) | | | | | | |
| х | | xx | (xx.x) | | | | | | |
| | x | | | XX | (xx.x) | ХX | (xx.x) | ХX | (xx.x) |
| /- | | | xx | | xx | | xx | | xx |
| /- | | | | | | | | | |
| XX (2 | (x.x) | ХX | (xx.x) | XX | (xx.x) | ХХ | (xx.x) | ХX | (xx.x) |
| х | x | | xx | | хх | | хх | | хх |
| xx () | (x.x) | ХX | (xx.x) | ХХ | (xx.x) | xx | (xx.x) | ХX | (xx.x) |
| х | x | | xx | | хх | | хх | | хх |
| хх (з | (x.x) | хx | (xx.x) | ХХ | (xx.x) | хх | (xx.x) | хx | (xx.x) |
| x | x | | xx | | xx | | xx | | xx |
| xx () | (x.x) | ХX | (xx.x) | ХХ | (xx.x) | xx | (xx.x) | ХX | (xx.x) |
| × | x | | xx | | хх | | хх | | хх |
| xx () | (x.x) | ХX | (xx.x) | ХХ | (xx.x) | xx | (xx.x) | ХX | (xx.x) |
| × | x | | xx | | хх | | хх | | хх |
| хх (з | (x.x) | ХX | (xx.x) | хх | (xx.x) | хх | (xx.x) | хx | (xx.x) |
| x | x | | xx | | хх | • | xx | | хх |
| | | | | | | • | | | |
| хх (з | (x.x) | хx | (xx.x) | xx | (xx.x) | хх | (xx.x) | хx | (xx.x) |
| x | x | | xx | | xx | | xx | | хх |
| | xx () xx () xx () xx () xx () xx () xx () | xx (xx.x) xx xx (xx.x) xx xx (xx.x) xx xx (xx.x) xx xx (xx.x) xx xx (xx.x) xx xx (xx.x) xx | XX (XX.X) | XX (XX.X) | xx (xx.x) xx (xx.x) xx xx xx xx xx (xx.x) xx (xx.x) xx xx xx xx xx (xx.x) xx (xx.x) xx xx (xx.x) xx (xx.x) xx xx (xx.x) xx xx xx (xx.x) xx xx xx (xx.x) xx xx xx (xx.x) xx xx xx (xx.x) xx xx | xx (xx.x) xx (xx.x) xx xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | xx (xx.x) xx (xx.x) xx (xx.x) xx xx xx xx xx xx (xx.x) xx (xx.x) xx xx xx (xx.x) xx (xx.x) xx xx xx (xx.x) xx (xx.x) xx xx xx (xx.x) xx (xx.x) xx xx xx (xx.x) xx (xx.x) xx xx xx (xx.x) xx xx xx xx (xx.x) xx xx xx xx (xx.x) xx xx xx | xx (xx.x) xx (xx.x) xx (xx.x) xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx xx xx xx xx xx | xx (xx.x) xx (xx.x) xx (xx.x) xx xx xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx xx (xx.x) xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx xx (xx.x) xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx xx (xx.x) xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx xx (xx.x) xx xx xx xx (xx.x) xx (xx.x) xx xx xx (xx.x) xx (xx.x) xx xx |

Document:


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


| System organ class | CIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any serious adverse event | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | XX | xx | xx |
| System organ class 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | XX | XX | xx | xx | xx |
| System organ class 2 | | | | | • |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | ХХ | xx | ХХ | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Etc | | | | | |

The full analysis set (FAS) has all eligible patients.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Table 39 Adverse Events Leading to Death by System Organ Class by Indication Overall (FAS)

| (N=xx) xx (xx.x) xx xx | (N=xx) xx (xx.x) xx | (N=xx)<br>xx (xx.x)<br>xx | (N=xx)<br>xx (xx.x)<br>xx |
|---|---|---|---|
| xx | | | |
| xx | | | |
| | xx | xx | XX |
| xx (xx.x) | | | |
| xx (xx.x) | | | |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | xx | xx |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | xx | xx |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | xx | ХХ |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | xx | xx |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | XX | xx |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | xx | ХХ |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | xx | ХХ |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| xx | xx | xx | xx |
| | <del>-</del> | | |

Document:


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

| System organ class | CIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any adverse event | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| System organ class 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| System organ class 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | XX | xx | xx |
| Etc | | | | | |

The full analysis set (FAS) has all eligible patients.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Table 40 Adverse Events Leading to Discontinuation of Ceftazidime-Avibactam by System Organ Class by Indication Overall (FAS)

| System organ class | CIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any adverse event | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| System organ class 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | XX | XX | XX | xx | xx |
| System organ class 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | XX | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | XX | XX | XX | xx | xx |
| Etc | | | | | |

The full analysis set (FAS) has all eligible patients.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Table 40.1 Adverse Events Related to Ceftazidime-Avibactam Leading to Discontinuation of Ceftazidime-Avibactam by System
Organ Class by Indication Overall (FAS)

| System organ class | cIAI | cUTI | HAP/VAP | Other | TOTAL |
|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Any adverse event | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| System organ class 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| System organ class 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 1 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 2 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | xx | xx | xx |
| Preferred term 3 | | | | | |
| Patients, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events, n | xx | xx | XX | xx | xx |
| Etc | | | | | |

The full analysis set (FAS) has all eligible patients.


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

### List of Listings

Document:

#### Listing 1.1. Site Characteristics (1)

| Site | Physician<br>specialty/<br>Other,<br>specify | Care<br>level | Hospital<br>type | Total<br>number<br>of beds | Total<br>number<br>of ICU<br>beds | Is the percentage of Gram-negative isolates that exhibit resistance to 3rd generation cephalosporins known? | If,<br>Yes/<br>Rate | Time period<br>start<br>date/Time<br>period end<br>date |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xx | xx | xx | xx | xx | xx | xx | xx |

#### Listing 1.2. Site Characteristics (2)

| Site | Is the percentage of Gram-negative isolates that exhibit resistance to carbapenems known? | If,<br>Yes/<br>Rate | Time period start date/Time period end date | Is the percentage of Gram-negative isolates that exhibit resistance to 3rd generation cephalosporins and carbapenems known? | If,<br>Yes/<br>Rate | Time period start date/Time period end date | Is the percentage of Gramnegative isolates that exhibit resistance to colistin known? | If,<br>Yes/<br>Rate | Time period start date/Time period end date |
|---|---|---|---|---|---|---|---|---|---|
| xx | хх | хх | xx | xx | хх | xx | xx | xxx | хх |


 $\label{thm:linear} Path: $$ \operatorname{Local} \operatorname{Coc} \operatorname{Coc$ 

Title: Annotated TLF Shells

#### Listing 2. Demographic

| Subjid | Date of informed consent /Did the patient pass all eligibility criteria? | Age/Sex | Height (cm) | Weight(kg) | BMI (kg/m^2) | Current employment status |
|---|---|---|---|---|---|---|
| xx | xx | xx | xx | xx | xx | xx |

#### Listing 3.1. Indication Diagnosis of UTI (ENR)

| Subjid | Age/Sex | Source of infection | Diagnosis<br>of UTI<br>Primary<br>diagnosis | Diagnosis<br>of UTI<br>Secondary<br>diagnosis | Sympt<br>oms | Date of<br>sampling | Positive dipstick for leukocyte esterase and/or nitrite | Date of<br>diagnosis | Patient<br>have a<br>secondary<br>bacteremia | Did the patient test positive for COVID-19 at admission or during hospitalization? |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | xx/F | xx | xx | | | DDMMMYYYY | | DDMMMYYYY | No | |

#### Listing 3.2. Indication Clinical Diagnosis of IAI

| Subjid | Age/Sex | Source of infection | Diagnosis of<br>IAI Primary<br>diagnosis | Diagnosis of<br>IAI<br>Secondary<br>diagnosis | Symptoms | Date of<br>diagnosis | Patient have<br>a secondary<br>bacteremia | Did the patient test positive for COVID-19 at admission or during hospitalization? |
|---|---|---|---|---|---|---|---|---|
| xx | xx/F | xx | | | | DDMMMYYYY | Yes | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Listing 3.3. Indication Nosocomial Pneumonia (NP) HAP- Hospital Associated Pneumonia (HAP) / Ventilator-Associated Pneumonia (VAP)

| Subjid | Age/Sex | Source of infection | HAP<br>Diagnosis | VAP<br>Diagnosis | Symptoms | Date of<br>diagnosis | Explain other; initial site of infection (organ) | Patient have<br>a secondary<br>bacteremia | Did the patient<br>test positive<br>for COVID-19 at<br>admission or<br>during<br>hospitalization? |
|---|---|---|---|---|---|---|---|---|---|
| хх | xx/F | xx | xx | xx | xxxxx | DDMMMYYYY | xxxxxxxx | xxxx | |

[1] CAI: Community-Acquired Infection; HAI: Hospital-Acquired Infection; HCAI: Healthcare-Associated Infection

#### Listing 3.4. Indication Other

| Subjid | Age/Sex | Source of infection | Indication for<br>ceftazidime-<br>avibactam<br>other | Symptoms | Explain other; initial site of infection (organ) | Patient have a<br>secondary<br>bacteremia | Did the patient test positive for COVID-19 at admission or during hospitalization? |
|---|---|---|---|---|---|---|---|
| хх | xx/F | xx | xx | xxxxx | xxxxxxxx | xxxx | |

#### Listing 4. Subject with Comorbidities

Document:

| Subjid | Age/Sex | Comorbidities | Deyo-Charlson<br>score<br>calculated | Diagnosis | Diagnosis<br>date | Chemotherapy received in the last 3 months? | Indwelling devices that the patient had at the time of the infection diagnosis |
|---|---|---|---|---|---|---|---|
| xx | xx/F | жx | XX | xx | Dd/mmm/yy | xx | xxxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

### **PLAN**

Document:

#### Listing 5. Prior Antibiotic Therapy

| Subjid | Age/Sex | Any antibiotic(s) used within 90 days prior to date of admission for the current hospitalization? | Antibiotic/ other | Start date/ Stop<br>date | Reason for<br>treatment |
|---|---|---|---|---|---|
| хх | xx/F | xx | xx | xx | xxxxxxxxx |

#### Listing 6. Prior Hospitalization

| Subjid | Age/Sex | Any prior hospitalizations within 90 days prior to date of admission for the current hospitalization? | Date of<br>admission | Date of<br>discharge | Primary diagnosis at<br>discharge SOC | Primary diagnosis at<br>discharge: Preferred Term |
|---|---|---|---|---|---|---|
| xx | xx/F | xx | xx | xx | xxxxxxx | ххххххх |

#### Listing 7. Healthcare Procedures within 30 days prior to ceftazidime-avibactam initiation

| Subjid | Age/Sex | Any prior healthcare procedures within 30 days prior to ceftazidime-avibactam initiation? | Date of healthcare procedure | Type of healthcare procedure | Other, specify |
|---|---|---|---|---|---|
| xx | xx/F | хх | xx | xx | xxxxxxxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

#### Listing 8. Additional Risk Factors

| Subjid | Age/Sex | Has the patient<br>travelled to any<br>foreign country in<br>the last 3 months?<br>/ Country | Start date/<br>Return date | Was subject<br>hospitalized<br>during travel? | Is the<br>patient<br>pregnant? | Number of<br>weeks of<br>gestation<br>since last<br>menstrual<br>period | Does the patient drink alcohol? / Number of drinks per week | Tobacco use |
|---|---|---|---|---|---|---|---|---|
| xx | xx/F | xx | xx | xx | | | | |

#### Listing 9. Antibiotic Therapy: Prior Lines of Treatment

| Subjid | Age/Sex | Any antibiotic(s) used for current infection before ceftazidime- avibactam initiation? | Antibiotic/<br>other | Start<br>date/<br>stop<br>date | Dose/<br>unit | Frequency | Route of administration | Reason for initiating | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|---|
| xx | xx/F | хх | | xx | xx | | | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Document:

#### **PLAN**

Document:

Listing 10. Pattern of use of Ceftazidime-Avibactam

| Subjid | Age/Sex | Use of<br>Ceftazidime-<br>avibactam<br>reported in<br>patient<br>records? | Start<br>date/<br>stop date | Dose/<br>unit | Frequency | Duration of<br>Administration<br>(hours) | Route of administration | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| xx | xx/F | xx | | xx | | | | |

#### Listing 11. Concomitant Antibiotic Therapy

| Subji<br>d | Age/Se<br>x | Any antibiotic(s) used concurrently with ceftazidime- avibactam? | Antibioti<br>c | Star<br>t<br>date<br>/<br>stop<br>date | Dose<br>/<br>unit | Frequenc<br>Y | Duration of<br>Administratio<br>n (days) | Route of administration | Reason<br>for<br>initiatin<br>g | Reason for<br>discontinuatio<br>n |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | xx/F | xx | | | xx | | | | | |

#### Listing 12. Antibiotic Treatment After Ceftazidime-Avibactam

| Subji<br>d | Age/Se<br>x | Any antibiotic(s) used directly after ceftazidime- avibactam? | Antibioti<br>c | Star<br>t<br>date<br>/<br>stop<br>date | Dose<br>/<br>unit | Frequenc<br>Y | Duration of Administration (days) | Route of administration | Reason<br>for<br>initiatin<br>g | Reason for<br>discontinuatio<br>n |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | xx/F | xx | | | xx | | | | | |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells


Listing 13. Initial Hospitalization

| Subj | Age/S | Date | Mode | Source | Ward | Date of | Diagno | Wards | Was the | Date | Diagno |
|---|---|---|---|---|---|---|---|---|---|---|---|
| id | ex | of<br>hospit<br>al<br>admiss<br>ion | of<br>admiss<br>ion | of<br>admissi<br>on/<br>Other | admitted<br>for initial<br>hospitaliza<br>tion | initial hospitaliza tion admission | sis at<br>admiss<br>ion | admitted/transf<br>erred to during<br>hospital stay | patient<br>dischar<br>ged by<br>the end<br>of the<br>study<br>period<br>(30 Jun<br>2019)? | of<br>hospit<br>al<br>discha<br>rge | sis at<br>discha<br>rge |
| хx | xx/F | xx | | | xx | | | | | | |

#### Listing 13.1. Disease Severity

Document:

| Subjid | Age/Sex | Was the patient<br>admitted to the<br>ICU | If yes, was APACHE II completed? | Score | If yes, was Score another disease severity score completed?/ Type of Score |
|---|---|---|---|---|---|
| xx | xx/F | Yes/NO | xx | xxx | xx |

#### Listing 14.1. Healthcare Resource Utilization During Hospitalization (1)

| Subjid | Age/Sex | Healthcare<br>resource<br>utilized | Mechanical<br>ventilation<br>Start date /<br>Stop date | Hemodialysis (including intermittent or continuous renal replacement therapy) | Start date / Stop<br>date / Number of<br>episodes | CT/MRI date/<br>Tracheostomy date |
|---|---|---|---|---|---|---|
| xx | xx/F | | | xx | | |

#### Listing 14.2. Healthcare Resource Utilization During Hospitalization - Percutaneous procedures (2)


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

| _ | Subjid | Age/Sex | Percutaneous<br>procedures SOC | • | Was percutaneous procedure performed to control infection? | Procedure/Date of procedure/Other | Was other procedure performed to control infection? |
|---|---|---|---|---|---|---|---|
| _ | хх | xx/F | xx | xx | xx | xx | xx |

#### Listing 14.3. Healthcare Resource Utilization During Hospitalization - Surgical Interventions (3)

| Subjid | Age/Sex | Surgical | Surgical | Surgical Indication | Surgical Indication | Was surgical |
|---|---|---|---|---|---|---|
| | | intervention date | Type | SOC | Preferred term | procedure performed |
| | | | | | | to control infection? |
| xx | xx/F | xxx | xx | xxx | xxx | xx |

#### Listing 15. Hospital Readmissions

Document:

| Subjid | Age/Sex | Was the patient readmitted to hospital within 60 days post-initial discharge? | Patient readmitted within 30 days of initial discharge or 60 days? | Date of<br>readmission/<br>Date of<br>discharge | Reason for readmission | Specify infection |
|---|---|---|---|---|---|---|
| xx | xx/F | xx | xx | xxx | xxxx | xxxxx |


Path: \\quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications

Title: Annotated TLF Shells

Listing 16 Treatment Evaluation for Initial Hospitalization and at 60-Days Post-Discharge

| Subjid | Age/Sex | Period | Date of evaluation | Clinical<br>success | Reason<br>for<br>success | Clinical<br>failure | Reason<br>for<br>failure | Clinical<br>Indeterminate | Reason<br>for<br>indeterminate |
|---|---|---|---|---|---|---|---|---|---|
| хх | xx/M | Initial<br>hospitalization<br>60 days post-<br>discharge | хх | ххх | ххх | ххх | ххх | xxx | ххх |
| xx | xx/M | Initial<br>hospitalization<br>60 days post-<br>discharge | хх | xxx | xxx | ххх | xxx | xxx | xxx |
| хх | xx/M | Initial<br>hospitalization<br>60 days post-<br>discharge | хх | xxx | xxx | ххх | ххх | xxx | ххх |

#### Listing 17. Microbiology Sample Taken

Document:

| Subjid | Age/Sex | Sample taken? | Date of identification | Timing of sample collection | Number of<br>bacterial<br>pathogen(s)<br>identified in<br>specimens<br>sampled | Was a fungal pathogen identified? | Type of<br>specimen |
|---|---|---|---|---|---|---|---|
| | xx/F | | | | | | |


 $Path: $$ \Path: $$ \operatorname{Local} BioStat Pfizer \array* Documentation \array* Descriptions $$ Path: $$ \array* Descriptions $$ Path: $$ \array* Description \array* Descri$ 

Title: Annotated TLF Shells

#### Zavicefta

#### C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS

#### **PLAN**

| Listing 18. Microbiology Bacterial Pathogens Identified in Specimen Sampled | Listing 18. | Microbiology | Bacterial | Pathogens | Identified | in | Specimen | Sampled |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

| Subjid | Age/Sex | Ceftazidime- | Infection | Date of | Sample type | Pathogen | Does the | How many | Ambler's | Type |
|---|---|---|---|---|---|---|---|---|---|---|
| | | avibactam<br>start date | type | identification -<br>sample time | | Identified | bacteria<br>present<br>any beta-<br>lactamase? | were identified? | class | |
| | xx/F | | | | | | | | | |
| | xx/F | | | | | | | | | |
| | xx/F | | | | | | | | | |

#### Footnote

Document:

<sup>1</sup> ST1: Sample Time 1 - ST2: Sample Time 2 - ST3: Sample Time 3 - ST4: Sample Time 4 - ST5: Sample Time 5 Sample time 1: Before initial antibiotic therapy - Sample time 2: After initial antibiotic therapy but before ceftazidime - avibactam therapy - Sample time 3: After initiation or during ceftazidime-avibactam therapy - Sample time 4: After end of ceftazidime-avibactam therapy - Sample time 5: After end of any antibiotic therapy.

#### Listing 18.1. Pathogen Susceptibility

| Subjid | Age/Sex | Ceftazidime-<br>Avibactam<br>start and<br>stop dates | Pathogen/date | Date of identification | Class of<br>antibiotic<br>tested | Antibiotic<br>tested | Susceptibility |
|---|---|---|---|---|---|---|---|
| ж | xx/F | | | | | | |


 $Path: $$ \Path: $$ \Path: $$ \Path: $$ Path: $$ P$ 

Title: Annotated TLF Shells


# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

Listing 19. Mortality and Cumulative Mortality in-Hospital, 30-Days and 60-Days Post Discharge

| Subjid | Period | Age/Sex | Did the patient die during the hospitalization or within 60 days post discharge? | Date of last ceftazidime avibactam administration | Date of<br>hospital<br>discharge | Date of<br>death | Cause of<br>death SOC | Cause of<br>death<br>Preferred<br>term |
|---|---|---|---|---|---|---|---|---|
| хх | Initial hospitalization 30-days post- discharge 60 days post- discharge | xx/F | ххх | хх | ж | ж | ххх | жж |
| жx | Initial hospitalization 30-days post- discharge 60 days post- discharge | xx/F | xxx | xx | хx | хx | | xxx |
| хх | Initial<br>hospitalization<br>30-days post-<br>discharge | xx/F | ххх | xx | хх | хх | | xxx |
| хх | 60 days post-<br>discharge | xx/F | xxx | xx | хx | xx | | xxx |

<sup>[1]</sup> Cumulative mortality up to 30 days post-discharge, including in-hospital mortality


 $Path: \underline{\Quintiles.net\Enterprise\Sites\USCBG\Depts\BioStat\Pfizer\Zavicefta\Documentation\Specifications}$ 

Title: Annotated TLF Shells

Document:

<sup>[2]</sup> Cumulative mortality up to 60 days post-discharge, including in-hospital mortality

Listing 20. Adverse Events

| | Age/Sex | AE SOC | AE<br>preferred<br>term | Start<br>date /End<br>date /<br>days | If, After<br>treatment<br>initiation<br>but before<br>hospital<br>discharge | Date of<br>death | Relationship | AE Serious?<br>Criteria<br>for<br>seriousness | Outcome | Action<br>taken |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx | xx/F | xxxxxx | xxxxxx | | | | | | | |
| isting | 21. Seriou | s Adverse | Events | | | | | | | |
| Subjid | Age/Sex | AE SOC | AE term | Start<br>date /End<br>date /<br>days | If, After<br>treatment<br>initiation<br>but before<br>hospital<br>discharge | Date of<br>death | Relationship | Criteria<br>for<br>seriousness | Outcome | Action<br>taken |
| ххх | xx/F | xxxxxx | xxxxxx | | | | | | | |
| Listing Subjid | 22. Advers<br>Age/Sex | | eading to Di | Start<br>date /End<br>date /<br>days | If, After treatment initiation but before hospital discharge | dime-Avib Date of death | actam<br>Relationship | AE Serious?<br>Criteria<br>for<br>seriousness | Outcome | Action<br>taken |


11 January 2022

Title: Annotated TLF Shells


 $\label{thm:lem:path$ 

# Zavicefta C3591031 NON-INTERVENTIONAL FINAL STUDY REPORT – APPENDIX 4 STATISTICAL ANALYSIS PLAN

| Subjid | Age/Sex | AE SOC | AE term | Start<br>date /End<br>date /<br>days | If, After treatment initiation but before hospital discharge | death | Relationship | AE Serious?<br>Criteria<br>for<br>seriousness | Outcome | Action<br>taken |
|---|---|---|---|---|---|---|---|---|---|---|
| isting 2 | 3. Patient | Disposition | on | | | | | | | |
| | | Date of | first | | | | If no, | | | |
| Subjid | Age/Sex | dose<br>Ceftazio<br>ibactam<br>of enrol | dime/av<br>(Date | Date of<br>Data<br>extraction | Date of ICF signature | Met<br>eligibility<br>criteria | inclusion | FAS72+ | FAS72- | Reason fo<br>exclusion<br>from FAS |
| xxx | xx/F | | | | DD-MMM-YYYY | Y | I1 | Y | Y | |
| | | | | | NA as per | | | | | |
| | | | | | local regulation | N | 12 | N | N | |
| | | | | | • | | 13 | | | |
| | | | | | | | 14 | | | |
| | | | | | | | 15 | | | |
| | | | | | | | E1 | | | |
| | | | | | | | E2 | | | |
| | | | | | | | E3 | | | |
| isting 2<br>Subjid | 4. End of Age/S | | Was p | oatient<br>owed through<br>cal records up | If No, re | ason Oth | mer, specify | Date of end<br>chart revie | | e of death |
| | | | | days after | • | | | | | |
| | | | hospi | tal discharge | 1? | | | | | |
| xxx | xx/F | | | | | | | | | |


 $\label{thm:lem:path$ 

Title: Annotated TLF Shells

Document:
